

#### STATISTICAL ANALYSIS PLAN

**Study Title:** A Phase 3, Randomized, Double-Blind Study to Evaluate the

Safety and Efficacy of Tenofovir Alafenamide (TAF) 25 mg QD versus Tenofovir Disoproxil Fumarate (TDF) 300 mg QD for the

Treatment of HBeAg Negative, Chronic Hepatitis B

Name of Test Drug: Tenofovir Alafenamide (TAF)

Study Number: GS-US-320-0108

**Protocol Version:** Amendment 3.1

**Protocol Date:** 23 February 2016

**Analysis Type:** Week 48 China

**Analysis Plan Version:** Version 1.0

**Analysis Plan Date:** 24 February 2017

Analysis Plan Author: PPD

CONFIDENTIAL AND PROPRIETARY INFORMATION

# **TABLE OF CONTENTS**

| TA | BLE OI | F CONTENTS | 2 |
|---|---|---|---|
| LIS | T OF I | N-TEXT TABLES | 4 |
| LIS | T OF A | BBREVIATIONS | 5 |
| 1. | INTR | Study Objectives Study Design Sample Size and Power OF PLANNED ANALYSIS Data Monitoring Committee (DMC) Analysis Week 48 Analysis (Primary Analysis) | |
| | 1.1. | Study Objectives | 8 |
| | 1.2. | | |
| | 1.3. | | |
| 2. | TYPE | OF PLANNED ANALYSIS | 14 |
| | 2.1. | Data Monitoring Committee (DMC) Analysis | 14 |
| | 2.2. | | |
| 3. | GENI | ERAL CONSIDERATIONS FOR DATA ANALYSES | 15 |
| | 3.1. | Analysis Sets | 15 |
| | | 3.1.1. Randomized Analysis Set | |
| | | 3.1.2. Safety Analysis Set | |
| | | 3.1.3. Full Analysis Set (FAS) | 15 |
| | | 3.1.4. Per-protocol Analysis Set | 15 |
| | | 3.1.5. Serologically Evaluable Full Analysis Set for HBsAg | |
| | | Loss/Seroconversion | |
| | | 3.1.6. DXA Analysis Set | |
| | 3.2. | Subject Grouping | |
| | 3.3. | Strata and Covariates | |
| | 3.4. | Examination of Subject Subgroups | |
| | 3.5. | Missing Data and Outliers | |
| | | 3.5.1. Missing Data | |
| | 3.6. | Data Handling Conventions and Transformations | |
| | 3.7. | Analysis Windows | |
| | 3.7. | 3.7.1. Definition of Study Day 1 and Other Definitions | |
| | | 3.7.2. Analysis Windows | |
| | | 3.7.3. Selection of Data in the Event of Multiple Records in a Window | |
| 4. | SUBJ | ECT DISPOSITION | |
| | 4.1. | Subject Enrollment | |
| | 4.1. | Disposition of Subjects | |
| | 4.3. | Extent of Exposure | |
| | ч.5. | 4.3.1. Duration of Exposure to Blinded Study Drug | |
| | | 4.3.2. Adherence with Blinded Study Drug Regimen | |
| | 4.4. | Protocol Deviations | |
| 5. | BASI | ELINE CHARACTERISTICS | 31 |
| | 5.1. Demographics and Baseline Characteristics | | |
| | 5.2. | Medical History | |
| 6. | | CACY ANALYSES | |
| υ. | | | |
| | 6.1. | Primary Efficacy Endpoints | |
| | | 6.1.1. Definition of the Primary Efficacy Endpoint | 33 |
| | | O 1 Z ADAIVSIS OF THE FIRMALY EMICACY EMODORNI | 11 |

| | | 6.1.3. | Secondary Analysis for the Primary Efficacy Endpoint | 33 |
|---|---|---|---|---|
| | | 6.1.4. | Subgroup Analysis for the Primary Efficacy Endpoint | |
| | 6.2. | - | y Efficacy Endpoints | |
| | | 6.2.1. | Definition of Secondary Efficacy Endpoints | |
| | 6.2 | 6.2.2. | Analysis Methods for Secondary Efficacy Endpoints | |
| | 6.3. | Changes I | From Protocol-Specified Efficacy Analyses | |
| 7. | SAFE | TY ANALY | YSES | 30 |
| | 7.1. | Adverse E | Events | |
| | | 7.1.1. | Adverse Event Dictionary | |
| | | 7.1.2. | Adverse Event Severity | 36 |
| | | 7.1.3. | Relationship of AEs to Study Drug | |
| | | 7.1.4. | Relationship of AEs to Study Procedure | |
| | | 7.1.5. | Serious AEs | |
| | | 7.1.6. | Treatment-Emergent AEs | |
| | | 7.1.7. | Summaries of AEs and Deaths | |
| | | 7.1.8. | Potential Uveitis Events | |
| | | 7.1.9. | Potential Cardiovascular Events | 40 |
| | 7.2. | Laborator | y Evaluations | |
| | | 7.2.1. | Summaries of Numeric Laboratory Results | 40 |
| | | 7.2.2. | Graded Laboratory Values | 42 |
| | | 7.2.3. | ALT Elevation | |
| | 7.3. | Bone Safe | ety Analyses | |
| | | 7.3.1. | Bone Mineral Density (BMD) | |
| | | 7.3.2. | Bone Biomakers | |
| | | 7.3.3. | Fracture Events. | 45 |
| | | 7.3.4. | Assessment of Fracture Probability | 45 |
| | | 7.3.5. | Bone Events | 45 |
| | 7.4. | Renal Saf | ety Analyses | 40 |
| | | 7.4.1. | Confirmed Renal Abnormalities | 40 |
| | | 7.4.2. | Serum Creatinine | 40 |
| | | 7.4.3. | Estimated Glomerular Filtration Rate | 40 |
| | | 7.4.4. | Treatment-Emergent Proteinuria (Dipstick) | 47 |
| | | 7.4.5. | Urine Creatinine, Urine RBP to Creatinine Ratio and | |
| | | | Beta-2-microglobulin to Creatinine Ratio | 47 |
| | | 7.4.6. | Proteinuria by Quantitative Assessment | 48 |
| | | 7.4.7. | Other Renal Biomarkers | 48 |
| | 7.5. | Ophthalm | ologic Assessment | 49 |
| | 7.6. | Body Wei | ight | 49 |
| | 7.7. | | atitis B Medications | |
| | 7.8. | Concomit | ant Medications | 49 |
| | 7.9. | Electrocar | rdiogram (ECG) Results | 50 |
| | 7.10. | Other Safe | ety Measures | 50 |
| | 7.11. | Changes I | From Protocol-Specified Safety Analyses | 50 |
| 8. | REFE | RENCES | | 5 |
| 9. | | | | |
| 10. | | | | |
| 11. | | | | |
| | Apper | | Table of Contents for Statistical Tables, Figures, and Listings | 55<br>66 |
| | Apper | ICHX Z | Fracture Events | 66 |

| Appendix 3. | Bone Events | |
|---|---|---|
| Appendix 4. Appendix 5. | Potential Uveitis | |
| | LIST OF IN-TEXT TABLES | |
| Table 3-1. | Subjects Excluded from Week 48 PP Analysis Set Due to Premature Discontinuation and/or Missing HBV DNA Assessment in Week 48 Analysis Window | 16 |
| Table 3-2. | Analysis Windows for HBV DNA, Hematology, Serum Chemistry and Liver Function Tests, Urinalysis, Urine Pregnancy Test, eGFR (by CG and CKD-EPI), PTH, UACR, UPCR, TmP/GFR, FEPO4, FEUA, Weight, and Vital Sign Assessments | |
| Table 3-3. | Analysis Windows for Safety ECG and Fibrotest | |
| Table 3-4. | Analysis Windows for BMD Results from DXAand Fasting Lipid Panel | |
| Table 3-5. | Analysis Windows for Serum HBsAg (Quantitative) and HBV Serology | |
| Table 3-6. | Analysis Windows for Fasting Glucose, Fasting Total Cholesterol, Fasting | |
| | Triglycerides, Renal, and Bone Biomarkers | 24 |
| Table 3-7. | Analysis Windows for PTH | |
| Table 3-8. | Analysis Windows for Hepatic Ultrasound | |
| Table 3-9. | Analysis Windows for Post-Treatment Assessments except HBV Serology | 26 |
| Table 3-10. | Analysis Windows for Post-Treatment HBV Serology | |
| Table 7-1. | Normal, Osteopenia, and Osteoporosis as Defined by T-score | 44 |

#### LIST OF ABBREVIATIONS

AASLD American Association for the Study of Liver Diseases

AE adverse event

ALT alanine aminotransferase (SGPT)

ANCOVA analysis of covariance
ANOVA analysis of variance
Anti-HBe antibody to HBeAg
Anti-HBs antibody to HBsAg

AST aspartate aminotransferase (SGOT)
BLQ below the limit of quantitation

BMD bone mineral density
BMI body mass index

bsAP bone specific alkaline phosphatase

CDER Center for Drug Evaluation and Research

CG Cockcroft-Gault
CHB chronic hepatitis B
CI confidence interval

CKD-EPI Chronic Kidney Disease Epidemiology Collaboration formula for calculating

glomerular filtration rate

CL<sub>Cr</sub> creatinine clearance

CMH Cochran-Mantel-Haenszel

CRF case report form

CTX c-type collagen sequence
CV coefficient of variation
DMC data monitoring committee
DNA deoxyribonucleic acid

DXA dual-energy x-ray absorptiometry

ECG electrocardiogram

eCRF electronic case report form ED early discontinuation

eGFR estimated glomerular filtration rate
ESDD early study drug discontinuation

FAS Full Analysis Set

FDA Food and Drug Administration

FEPO<sub>4</sub> fractional excretion of filtered phosphate

FEUA fractional excretion of uric acid

GFR glomerular filtration rate
Gilead Gilead Sciences, Inc.
HBeAb hepatitis B e antibody

HBeAg hepatitis B e antigen

HBsAb hepatitis B surface antibody HBsAg hepatitis B surface antigen

HBV hepatitis B virus

HCC hepatocellular carcinoma

HCV hepatitis C virus

HDL high density lipoprotein

HDV hepatitis D virus

HIV human immunodeficiency virus

HLGT high-level group term HLT high-level term

IVRS interactive voice response system IWRS interactive web response system

LDL low density lipoprotein

LLN lower limit of the normal range

LLT lower-level term

LOCF last observation carried forward

M = E Missing = ExcludedM = F Missing = Failure

MDRD Modification of Diet in Renal Disease

MedDRA Medical Dictionary for Regulatory Activities

MH Mantel-Haenszel OC osteocalcin

P1NP procollagen type 1 N-terminal propeptide

PBMC peripheral blood mononuclear cell

PP per protocol
PT preferred term
Q quartile
Q1 first quartile
Q3 third quartile
QD once daily

RBP retinol binding protein
SAE serious adverse event
SAP statistical analysis plan
SD standard deviation
SOC system organ class

TAF tenofovir alafenamide (Vemlidy®)
TDF tenofovir disoproxil fumarate (Viread®)

TFLs tables, figures, and listings

TFV tenofovir

TFV-DP tenofovir-diphosphate

TmP tubular maximum reabsorption rate of phosphate

UACR urine albumin to creatinine ratio

ULN upper limit of normal

UPCR urine protein to creatinine ratio
WHO World Health Organization

### 1. INTRODUCTION

GS-US-320-0108 is a randomized, double-blind, noninferiority study to compare the antiviral activity of tenofovir alafenamide (TAF) 25 mg once daily versus tenofovir disoproxil fumarate (TDF) 300 mg once daily for the treatment of HBeAg-negative, chronic hepatitis B (CHB) in treatment-naive and treatment-experienced subjects. For non-China part, 426 subjects were randomized in a 2:1 ratio to the treatment groups, and were stratified by plasma hepatitis B virus (HBV) DNA level (<  $7 \log_{10} IU/mL$ ,  $\geq 7 \log_{10} IU/mL$  - <  $8 \log_{10} IU/mL$ ,  $\geq 8 \log_{10} IU/mL$ ) and oral antiviral treatment status (treatment-naive vs treatment-experienced).

Treatment-naive subjects are defined as subjects with < 12 weeks of previous oral antiviral treatment with any nucleoside or nucleotide analogue. Treatment-experienced subjects are defined as subjects with  $\ge 12$  weeks of previous treatment with any nucleoside or nucleotide analogue.

For China, approximately 150 additional subjects (100 in TAF group and 50 in TDF group) will be enrolled for local registration purposes.

The duration of double-blind treatment is 144 weeks (96 weeks under Amendment 1 and 2.1). All subjects who complete the double-blind period of treatment are eligible for participation in the open label TAF 25 mg extension period for an additional 240 weeks (through Week 384/ED). Subjects who already entered open label phase at Week 96 per Amendment 2.1 will continue on open label TAF 25 mg QD through Week 384/ED. For the entire duration of the study, subjects and investigators will remain blinded to the initial treatment regimen to which they were randomized.

This statistical analysis plan (SAP) describes the analysis plan for the Week 48 analysis of subjects enrolled in China only.

#### 1.1. Study Objectives

The primary objectives of this study are as follows:

- To compare the efficacy of TAF 25 mg versus TDF 300 mg once daily for the treatment of hepatitis B e antigen (HBeAg)-negative, CHB at Week 48 in treatment-naive and treatment-experienced subjects. The primary efficacy parameter is the proportion of subjects with plasma HBV DNA levels below 29 IU/mL
- To compare the safety and tolerability of TAF 25 mg once daily versus TDF 300 mg once daily for the treatment of HBeAg-negative, CHB at Week 48 in treatment-naive and treatment-experienced subjects

The key secondary safety objectives of this study are as follows:

- To compare the safety of TAF 25 mg once daily versus TDF 300 mg once daily as determined by the percent change from baseline in hip and spine bone mineral density (BMD) at Week 48
- To compare the safety of TAF 25 mg once daily versus TDF 300 mg once daily as determined by the change from baseline in serum creatinine at Week 48
- To compare the safety of TAF 25 mg once daily versus TDF 300 mg once daily as determined by treatment-emergent proteinuria through Week 48

Other secondary objectives of this study are as follows:

- To compare the efficacy of TAF 25 mg once daily versus TDF 300 mg once daily for the treatment of HBeAg-negative, CHB in regard to the proportion of subjects with plasma HBV DNA levels below 29 IU/mL at Week 96, and 144
- To compare the efficacy of TAF 25 mg once daily versus TDF 300 mg once daily for the treatment of HBeAg-negative, CHB in regard to the proportion of subjects with plasma HBV DNA levels below 29 IU/mL (target not detected) at Weeks 48, 96, and 144
- To compare the biochemical (alanine aminotransferase [ALT] normalization) response of TAF 25 mg once daily versus TDF 300 mg once daily for the treatment of HBeAg-negative, CHB at Weeks 48, 96, and 144
- To compare the serological response (loss of hepatitis B surface antigen [HBsAg] with seroconversion to antibody to HBsAg [anti-HBs]) of TAF 25 mg once daily versus TDF 300 mg once daily for the treatment of HBeAg-negative, CHB at Weeks 48, 96, and 144
- To compare the change in fibrosis as assessed by FibroTest® of TAF 25 mg once daily versus TDF 300 mg once daily for the treatment of HBeAg-negative, CHB at Weeks 48, 96, and 144
- To compare the incidence of drug resistant mutations of TAF 25 mg once daily versus TDF 300 mg once daily at Weeks 48, 96, and 144
- To compare the change from baseline in ophthalmologic findings by fundoscopic examination of TAF 25 mg once daily versus TDF 300 mg once daily at Weeks 24, 48, 72, 96, and 144 (or ED visit if prior to Week 144 and more than 24 weeks since prior exam) in a subset of subjects
- To characterize the pharmacokinetics of TAF and tenofovir (TFV) and determine intracellular concentrations of tenofovir diphosphate (TFV-DP) within peripheral blood mononuclear cells (PBMCs) in subjects receiving TAF or TDF

- To evaluate the comparative open-label efficacy, safety, and drug resistance mutations of TAF 25 mg QD from Week 96 (Amendments 1 and 2.1) or Week 144 (Amendment 3.1) through Week 384 in subjects initially randomized to TAF 25 mg QD and in subjects sequentially treated with TDF 300 mg QD for 96 weeks (Amendments 1 and 2.1) or for 144 weeks (Amendment 3.1) and then switched to open-label TAF 25 mg QD
- To compare the safety and tolerability of TAF 25 mg once daily versus TDF 300 mg once daily for the treatment of HBeAg-negative, CHB beyond Week 48 during the double-blind phase in treatment-naive and treatment-experienced subjects

### 1.2. Study Design

#### **Design Configuration and Subject Population**

GS-US-320-0108 is a randomized, double-blind, noninferiority study to compare the antiviral activity of TAF 25 mg versus TDF 300 mg for the treatment of HBeAg-negative, CHB in treatment-naive and treatment-experienced subjects.

## **Treatment Groups**

For non-China part, subjects were randomized in a 2:1 ratio to the following 2 treatment groups:

- TAF group: TAF 25 mg once daily + matched placebo of TDF 300 mg once daily (n = 285)
- **TDF group:** TDF 300 mg once daily + matched placebo of TAF 25 mg once daily (n = 141)

For China, approximately 150 subjects (100 in TAF group and 50 in TDF group) will be enrolled for local registration purposes.

#### **Key Eligibility Criteria**

Subjects were to have met the following key eligibility criteria:

- Documented evidence of chronic HBV infection (eg, HBsAg positive for more than 6 months)
- HBeAg-negative, CHB with the following: HBeAg-negative and HBeAb-positive at screening; screening HBV DNA  $\geq 2 \times 10^4$  IU/mL; screening serum ALT level > 60 U/L (males) or > 38 U/L (females) and  $< 10 \times$  ULN (by central laboratory range)
- Estimated creatinine clearance (CLcr) ≥ 50 mL/min (using the Cockcroft-Gault [CG] method) based on serum creatinine and actual body weight as measured at screening

### **Study Periods/Phases**

The duration of randomized, double-blind treatment is 144 weeks (96 weeks under Amendment 1 and 2.1). At Week 144, all subjects remaining on blinded treatment will be switched to the open-label TAF 25 mg QD extension period for an additional 240 weeks (Week 144 through Week 384/ED). Subjects who already assigned to open-label phase at Week 96 per Amendment 2.1 and consented to Amendment 3.1 later will continue on open-label TAF 25 mg QD through Week 384/ED. All subjects who complete the double-blind period of treatment are eligible for participation in the open-label TAF 25 mg QD extension period. Subjects who permanently discontinue study drug (either prematurely [early discontinuation, ED] or at the end of study [Week 384]) for reasons other than HBsAg loss with confirmed seroconversion to anti-HBs will be followed every 4 weeks for 24 weeks off treatment or until initiation of alternative, commercially available HBV therapy, whichever occurs first.

#### **Schedule of Assessments**

Laboratory analyses (serum chemistry, liver tests, hematology, urinalysis, plasma HBV DNA levels, pregnancy testing [for females of childbearing potential]), vital signs, adverse events (AEs), and concomitant medications will be performed at screening, baseline, and every 4 weeks thereafter through Week 48, every 8 weeks through Week 96, every 12 weeks through Week 144, and every 24 weeks through Week 384/ED visit.

HBV serology (HBeAg, hepatitis B e antibody [HBeAb], HBsAg, and reflex hepatitis B surface antibody [HBsAb]) will be performed at screening and baseline, and HBsAg and reflex HBsAb will be performed every 12 to 16 weeks through Week 144, and every 24 weeks through Week 384 /ED, and at Follow up Weeks 12 and 24. Quantitative serum HBsAg will be assessed at screening, baseline, every 12-16 weeks until Week 144, every 24 weeks until Week 384/ED, and at all Follow Up visits. Bone and renal biomarker testing will be performed at baseline and then at defined intervals throughout the study. IL28B polymorphism genotype, HBV genotyping and vitamin D assessments will be performed at baseline only. FibroTest® will be performed at baseline, and every 48 weeks thereafter through Week 384/ED. Fasting metabolic assessments (fasting glucose and lipid panel) will be conducted at baseline, every 24 weeks until Week 144, and every 48 weeks until Week 384/ED visit.

Complete physical examinations will be performed at screening, baseline, and Weeks 24, 48, 72, 96, 120,144, 240, and 384/ED. Symptom directed physical examinations including body weight assessment will be conducted at all other visits. Electrocardiogram (ECG) will be performed at screening and every 48 weeks thereafter. At sites in China with the capability only, dual energy x-ray absorptiometry (DXA) scans of the hip and spine will be conducted anytime during the screening period, and should be conducted at least 14 days prior to the first dose of study drug, and will be conducted every 24 weeks through Week 144, and every 48 weeks thereafter until Week 384/ED visit if not done within the last 24 weeks of ED visit. Hepatic ultrasound for surveillance of hepatocellular carcinoma will be performed starting at Week 96 and then every 24 weeks thereafter until Week 384/ED. Plasma, serum, and urine will be collected at baseline and at every visit thereafter for storage.

Follow-up assessments will occur every 4 weeks for 24 weeks and include the following: vital signs, hematology, serum chemistry, liver function tests, and plasma HBV DNA. Plasma, serum and urine will be collected for storage. HBsAg and reflex HBsAb will be evaluated at follow-up Weeks 12 and 24.

### **Ophthalmologic Substudy**

For subjects who provide a separate informed consent (n = 30), a substudy will be conducted to assess ophthalmologic findings, including a fundoscopic examination with slit lamp and retinal photographs (both eyes) prior to the first dose of study drug and at Weeks 24, 48, 72, 96, and 144/ED visits at select sites. An exam should be performed at the ED visit if it is prior to Week 144 and not done within the last 24 weeks of this visit.

#### Randomization

Subjects will be randomized in a 2:1 ratio to the 2 treatment groups (TAF vs TDF, respectively). Randomization will be stratified by plasma HBV DNA level (<  $7 \log_{10} IU/mL$ ,  $\geq 7 \log_{10} IU/mL - < 8 \log_{10} IU/mL$ ,  $\geq 8 \log_{10} IU/mL$ ) and oral antiviral treatment status (treatment-naive vs treatment-experienced).

### Site and/or Stratum Enrollment Limits

Twenty-nine centers participated in China. There is no enrollment limit for individual sites.

#### **Study Duration**

The duration of the double-blind treatment is 144 weeks (96 weeks under Amendment 1 and 2.1). All subjects who complete the double-blind period of treatment are eligible for participation in the open label TAF 25 mg extension period for an additional 240 weeks (through Week 384/ED). Subjects already assigned to open label TAF 25 mg QD at Week 96 per Amendment 2.1 will continue on open label TAF 25 mg QD through Week 384/ED. Subjects who permanently discontinue study drug (either prematurely [ED] or at the end of study [Week 384]) for reasons other than HBsAg loss with confirmed seroconversion to anti-HBs will be followed every 4 weeks for 24 weeks off treatment or until initiation of alternative, commercially available HBV therapy, whichever occurs first. All subjects in China are currently enrolled under Amendment 3.1 and will complete 3 years of double-blind treatment before rolling over to open-label TAF 25 mg once daily.

Subjects with HBsAg loss with confirmed seroconversion to anti-HBs should discontinue study drug within 3-6 months following confirmation of seroconversion to anti-HBs. Subjects with HBsAg loss with confirmed seroconversion to anti-HBs prior to Week 48 are not permitted to discontinue study drug prior to the Week 48 visit. Subjects who discontinue study drug for confirmed seroconversion to anti-HBs will be followed off treatment every 4 weeks for 12 weeks and then per the study visit schedule through Week 384/ED. Discontinuation of study drug for subjects experiencing HBsAg loss with confirmed seroconversion, who have known bridging fibrosis or cirrhosis, should be considered on a case by case basis.

# 1.3. Sample Size and Power

For China, approximately 150 subjects (100 in TAF group and 50 in TDF group) will be enrolled for local registration purposes.

The sample size and power calculation described below was for non-China subjects. With respect to the primary efficacy endpoint of proportion of subjects with plasma HBV DNA levels below 29 IU/mL at Week 48, a sample size of 130 for the TDF group and 260 for the TAF group will have 90% power to rule out the noninferiority margin of 10% at a 1-sided significance level of 0.025. This assumes the expected difference (TAF – TDF) in proportion of subjects with HBV DNA < 29 IU/mL is 0 and the proportion of subjects with HBV DNA < 29 IU/mL in the TDF group is 91%. A similar response rate in the TDF group was observed in Study GS-US-174-0102.

This sample size (n = 260 for the TAF 25 mg group, n = 130 for the TDF 300 mg group) also provides the following:

- At least 90% power to detect a 1% difference in the percentage change from baseline in hip BMD at Week 48 (assuming a –1.17% change from baseline in TDF 300 mg group and –0.17% change from baseline in the TAF 25 mg group, with a common standard deviation (SD) of 2.20% and a 2-sided α = 0.025)
- At least 77% power to detect a 1% difference in the percent change from baseline in spine BMD at Week 48 (assuming a -1.69% change from baseline in the TDF 300 mg group and -0.69% change in the TAF 25 mg group, with a common SD of 3.08% and a 2-sided  $\alpha = 0.025$ )
- At least 52% power to detect a 0.03 mg/dL difference in the change from baseline in serum creatinine at Week 48 (assuming a 0.04 mg/dL change from baseline in the TDF 300 mg group and 0.01 mg/dL change from baseline in the TAF 25 mg group, with a common SD of 0.12)

These assumptions above were derived from Studies GS-98-437, GS-98-438, GS-US-174-0102, GS-US-174-0103, and GS-US-174-0121.

### 2. TYPE OF PLANNED ANALYSIS

The Week 48 analysis for Non-China subjects was already conducted after the last subject completed the Week 48 visit or prematurely discontinued study drug. This statistical analysis plan (SAP) describes the analysis plan for the Week 48 analysis of subjects enrolled in China only.

# 2.1. Data Monitoring Committee (DMC) Analysis

An external multidisciplinary data monitoring committee (DMC) will review the progress of the study and perform interim reviews of safety data and provide recommendation to Gilead whether the nature, frequency, and severity of adverse effects associated with study treatment warrant early termination of the study in the best interests of the participants and whether the study should continue as planned or with modifications. The DMC may also provide recommendations as needed regarding study design.

The DMC will convene approximately every 24 weeks during the blinded portion of the study and approximately every 48 weeks during the open-label phase. More details are documented in the independent DMC charter.

# 2.2. Week 48 Analysis (Primary Analysis)

The Week 48 analysis will be conducted after the last subject completes the Week 48 visit or prematurely discontinues study drug.

Further analyses after Week 48 will be conducted if warranted.

### 3. GENERAL CONSIDERATIONS FOR DATA ANALYSES

# 3.1. Analysis Sets

Analysis sets define which subjects are included in an analysis. The assignment of subjects to analysis sets will be done before the study blind is broken for analysis. A summary of the number and percentage of subjects in each analysis set will be provided by treatment group and in total.

# 3.1.1. Randomized Analysis Set

The Randomized Analysis Set includes all subjects who were randomized into the study. This is the primary analysis set for by-subject listings.

# 3.1.2. Safety Analysis Set

The Safety Analysis Set includes all randomized subjects who have received at least 1 dose of study drug. Subjects will be analyzed according to the treatment they actually received during the double-blinded phase. This is the primary analysis set for safety analyses.

#### 3.1.3. Full Analysis Set (FAS)

The FAS includes all randomized subjects who have received at least 1 dose of study drug. Subjects will be analyzed according to the treatment to which they were randomized during the double-blinded phase. This is the primary analysis set for efficacy analyses.

### 3.1.4. Per-protocol Analysis Set

The Week 48 Per-Protocol (PP) Analysis Set includes all subjects who (1) were randomized into the study, (2) had received at least 1 dose of study drug, and (3) had not been excluded based on criteria below. Subjects will be analyzed according to the treatment they actually received during the double-blinded phase. The PP analysis set is the secondary analysis set for efficacy analysis.

Subjects meeting any of the following criteria will be excluded from the Week 48 PP analysis set:

• Subjects who do not have on-treatment HBV DNA in the Week 48 analysis window, except for subjects who discontinue study drug due to lack of efficacy. (Note: lack of efficacy is defined as having the check-box for "Lack of Efficacy" marked as the reason for premature study drug discontinuation on the study drug completion electronic case report form [eCRF] page). The details are summarized in Table 3-1.

Table 3-1. Subjects Excluded from Week 48 PP Analysis Set Due to Premature Discontinuation and/or Missing HBV DNA Assessment in Week 48 Analysis Window

| Discontinuation from Study Drug Prior to or on the Upper Bound of Week 48 Analysis Window | | HBV DNA Data on Randomized Treatment<br>Available in Week 48 Analysis Window | |
|---|---|---|---|
| | | Yes | No |
| Vac | Due to Lack of Efficacy | + | + |
| Yes | Due to Other Reasons | + | - |
| No | | + | - |

<sup>+=</sup> Inclusion of Subjects in Week 48 PP analysis set; -= Exclusion of Subjects in Week 48 PP analysis set

- Subjects who meet the exclusion criterion for receiving ongoing therapy with any of the prohibited medications listed in the clinical study protocol (Section 4.3, Table 5.1).
- Subjects with adherence rate for active study drug up to the Week 48 visit below the 2.5th percentile.

#### 3.1.5. Serologically Evaluable Full Analysis Set for HBsAg Loss/Seroconversion

The Serologically Evaluable Full Analysis Set for HBsAg loss/seroconversion includes all subjects who were randomized and had received at least 1 dose of study drug, and with HBsAg positive and HBsAb negative or missing at baseline. Subjects will be analyzed according to the treatment they were randomized to during the double-blinded phase.

#### 3.1.6. DXA Analysis Set

DXA scans will be performed only at sites in China with capability.

#### 3.1.6.1. Hip DXA Analysis Set

The Hip DXA Analysis Set includes all subjects who were randomized and had received at least 1 dose of study drug, and had nonmissing baseline hip BMD values. Subjects will be analyzed according to the treatment they actually received during the double-blinded phase.

#### 3.1.6.2. Spine DXA Analysis Set

The Spine DXA Analysis Set will include all subjects who were randomized and had received at least 1 dose of study drug, and had nonmissing baseline spine BMD values. Subjects will be analyzed according to the treatment they actually received during the double-blinded phase.

# 3.2. Subject Grouping

For efficacy analysis using FAS and Serologically Evaluable Full Analysis Set, subjects will be analyzed by randomized treatment during the double-blinded phase. For efficacy analysis based on the PP analysis set and safety analysis, subjects will be analyzed by actual treatment received during the double-blinded phase. The actual treatment received will differ from the randomized treatment only when their actual treatment differs from randomized treatment for the entire double-blinded treatment duration.

#### 3.3. Strata and Covariates

Randomization was stratified by plasma HBV DNA level ( $<7 \log_{10} IU/mL$ ,  $\ge 7 \log_{10} IU/mL$  -  $<8 \log_{10} IU/mL$ ,  $\ge 8 \log_{10} IU/mL$ ) and oral antiviral treatment status (treatment-naive vs treatment-experienced) at screening. HBV DNA strata will be reclassified using baseline HBV DNA level for stratified statistical analysis.

# 3.4. Examination of Subject Subgroups

The primary endpoint will be analyzed for the following subject subgroups:

- Age: (a)  $\leq$  50 years and (b)  $\geq$  50 years
- Sex: (a) male and (b) female
- Baseline HBV DNA: (a)  $< 7 \log_{10} IU/mL$  and (b)  $\ge 7 \log_{10} IU/mL$
- Oral antiviral treatment status: (a) treatment-naive and (b) treatment-experienced
- Study drug adherence: (a) < 95% and (b)  $\ge 95\%$  (based on adherence up to Week 48 Visit)
- Genotype: (a) B, (b) C, and (c) Other
- Baseline ALT by central laboratory normal range: (a)  $\leq$  ULN and (b) > ULN
- Baseline fibrotest score: (a) < 0.75 and (b)  $\ge 0.75$

#### 3.5. Missing Data and Outliers

#### 3.5.1. Missing Data

A missing datum for a given study analysis window may be due to any of the following reasons:

- A visit occurring in the window but data were not collected or were unusable
- A visit not occurring in the window
- A subject permanently discontinuing from the study before reaching the window

For the primary endpoint and the secondary efficacy endpoints involving proportions, missing data will be handled using M = F approach. Sensitivity analyses will also be performed including an analysis excluding all missing data.

For the 3 key secondary safety endpoints (percentage change from baseline in hip BMD at Week 48, percentage change from baseline in spine BMD at Week 48, change from baseline in serum creatinine at Week 48), an analysis will be performed using the last observation carried forward (LOCF) method to impute missing data.

For the remaining endpoints, values for missing data will not be imputed, unless specified otherwise.

#### **3.5.2. Outliers**

Outliers may be identified during data management and data analysis process, but no sensitivity analyses will be done to evaluate the impact of outliers on efficacy or safety outcomes, unless specified otherwise. All data will be included in the analysis.

## 3.6. Data Handling Conventions and Transformations

Logarithm (base 10) will be used to transform HBV DNA and quantitative HBsAg data.

Data that are continuous in nature but are below the lower limit of quantitation or above the upper limit of quantitation will be imputed as follows except for direct bilirubin, urine creatinine, and serum cystatin C:

- A value that is 1 unit less than the limit of quantitation will be used for calculation of descriptive statistics if the datum is reported in the form of "< x" (x is considered as the limit of quantitation). For example, if the values are reported as < 50 and < 5.0, then values of 49 and 4.9 will be used for calculation of summary statistics, respectively.
- A value that is 1 unit above the limit of quantitation will be used for calculation of descriptive statistics if the datum is reported in the form of "> x" (x is considered as the limit of quantitation). Values with decimal points will follow the same logic as stated above.
- The limit of quantitation will be used for calculation of descriptive statistics if the data is reported in the form of " $\leq$  x" or " $\geq$  x" (x is considered as the limit of quantitation).

For direct bilirubin, a value of "< 0.1" is imputed as 0.09. For urine creatinine, a value of "< 1" is handled as a missing value in its summary and the calculation of related ratios. For serum cystatin C, a value of "< 0.10" is handled as a missing value in the calculation of estimated glomerular filtration rate (eGFR).

For HBV DNA, if the value in IU/mL (TaqMan) is above the upper limit of quantification, the corresponding diluted value (TaqDil), if available, will be used.

# 3.7. Analysis Windows

### 3.7.1. Definition of Study Day 1 and Other Definitions

**Study Day 1** is defined as the day when the first dose of the blinded study drug was taken, as recorded on the Study Drug Administration eCRF form.

**Open-Label Study Day 1** is defined as the day when the first dose of the open-label study drug was taken, as recorded on the Study Drug Administration eCRF form.

**Study days** are calculated relative to Study Day 1. For events that occurred on or after Study Day 1 date, study days are calculated as (visit date – Study Day 1 + 1). For events that occurred prior to Study Day 1, study days are calculated as (visit date – Study Day 1).

**Open-Label Study days** are calculated relative to Open-Label Study Day 1. For events that occurred on or after Open-Label Study Day 1 date, study days are calculated as (visit date – Open-Label Study Day 1 + 1).

**Follow-up days** are for visits occurred during 24-week treatment-free follow-up period and calculated as (visit date – last dose date).

Last Dose Date of Blinded Study Drug is the latest non-missing end date of blinded study drug, recorded on the Study Drug Administration eCRF form with "Study Drug Permanently Discontinued" box checked for subjects who prematurely discontinued blinded study drug or who completed blinded study drug according to Blinded Study Drug Completion eCRF. If the last dose date of blinded study drug is missing (eg, due to lost to follow up) for subjects who prematurely discontinued blinded study drug, or for subjects who are still on blinded study drug, the latest of nonmissing blinded study drug start dates and end dates, the clinical visit dates and the laboratory visit dates excluding the dates of open-label and 24-week treatment-free follow-up visits will be used to impute the last dose date of blinded study drug.

For subjects who prematurely discontinued blinded study drug or who completed blinded study drug but did not enter open-label phase, the **Last Dose Date** is the same as Last Dose Date of Blinded Study Drug.

For subjects who completed blinded study drug and entered open-label phase, the **Last Dose Date** is the latest non-missing end date of open-label study drug, recorded on the Study Drug Administration eCRF form with "Study Drug Permanently Discontinued" box checked for subjects who prematurely discontinued open-label study drug or who completed open-label study drug according to Open-Label Study Drug Completion eCRF. If the last dose date is missing (eg, due to lost to follow up) for subjects who prematurely discontinued open-label study drug, or for subjects who are still on open-label study drug, the latest of nonmissing open-label study drug start dates and end dates, the clinical visit dates and the laboratory visit dates excluding the dates of 24-week treatment-free follow-up visits will be used to impute the last dose date.

**Last Study Date** is the latest of nonmissing study drug (blinded or open-label) start dates and end dates, the clinic visit and the laboratory visit dates including the 24-week treatment-free follow-up visit date for subjects who prematurely discontinued study or who completed study according to Study Completion eCRF.

**Baseline value** is defined as the last nonmissing value obtained on or prior to Study Day 1. For DXA BMD, it is defined as the last value on or prior to Study Day 14.

#### 3.7.2. Analysis Windows

Subject visits might not occur on protocol specified days. Therefore, for the purpose of analysis, observations will be assigned to analysis windows.

The following windows (Table 3-2 to Table 3-8) apply to baseline and on-treatment assessments only, ie, data collected up to the last dose date for those who discontinued study drug prematurely (except efficacy data [HBV DNA, quantitative HBsAg, HBV serology, ALT, fibrotest score] for subjects who discontinue study drug after Week 48 due to HBsAg loss with confirmed seroconversion to anti-HBs), or data collected up to database finalization date for those who have not discontinued study drug permanently.

For subjects who discontinue study drug early due to HBsAg loss with confirmed seroconversion, all efficacy data including data collected after the last dose date of the study drug will be reassigned analysis visits using the on-treatment assessment windows (Table 3-2, Table 3-3, and Table 3-5).

The analysis windows for HBV DNA, hematology, serum chemistry and liver function tests, urinalysis, urine pregnancy test, eGFR (by CG and Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI]), renal biomarkers urine albumin to creatinine ratio (UACR), urine protein to creatinine ratio (UPCR), renal tubular maximum reabsorption rate of phosphate to the glomerular filtration rate (TmP/GFR), urine fractional excretion of filtered phosphate (FEPO<sub>4</sub>), fractional excretion of uric acid (FEUA), weight, and vital sign assessments are presented in Table 3-2.

Table 3-2. Analysis Windows for HBV DNA, Hematology, Serum Chemistry and Liver Function Tests, Urinalysis, Urine Pregnancy Test, eGFR (by CG and CKD-EPI), PTH, UACR, UPCR, TmP/GFR, FEPO4, FEUA, Weight, and Vital Sign Assessments

| Visit ID | Nominal Day | Lower Limit | Upper Limit |
|----------|-------------|-------------|-------------|
| Baseline | | | 1 |
| Week 4 | 28 | 2 | 41 |
| Week 8 | 56 | 42 | 69 |
| Week 12 | 84 | 70 | 97 |
| Week 16 | 112 | 98 | 125 |
| Week 20 | 140 | 126 | 153 |
| Week 24 | 168 | 154 | 181 |
| Week 28 | 196 | 182 | 209 |
| Week 32 | 224 | 210 | 237 |
| Week 36 | 252 | 238 | 265 |
| Week 40 | 280 | 266 | 293 |
| Week 44 | 308 | 294 | 321 |
| Week 48 | 336 | 322 | 363 |
| Week 56 | 392 | 364 | 419 |
| Week 64 | 448 | 420 | 475 |
| Week 72 | 504 | 476 | 531 |
| Week 80 | 560 | 532 | 587 |
| Week 88 | 616 | 588 | 643 |
| Week 96 | 672 | 644 | 713 |
| Week 108 | 756 | 714 | 797 |
| Week 120 | 840 | 798 | 881 |
| Week 132 | 924 | 882 | 965 |
| Week 144 | 1008 | 966 | 1091 |
| Week 168 | 1176 | 1092 | 1259 |
| Week 192 | 1344 | 1260 | 1427 |
| Week 216 | 1512 | 1428 | 1595 |
| Week 240 | 1680 | 1596 | 1763 |
| Week 264 | 1848 | 1764 | 1931 |
| Week 288 | 2016 | 1932 | 2099 |
| Week 312 | 2184 | 2100 | 2267 |
| Week 336 | 2352 | 2268 | 2435 |
| Week 360 | 2520 | 2436 | 2603 |
| Week 384 | 2688 | 2604 | 2771 |

The analysis windows for safety ECG and fibrotest are presented in Table 3-3.

Table 3-3. Analysis Windows for Safety ECG and Fibrotest

| Visit ID | Nominal Day | Lower Limit | Upper Limit |
|----------|-------------|-------------|-------------|
| Baseline | | | 1 |
| Week 48 | 336 | 2 | 503 |
| Week 96 | 672 | 504 | 839 |
| Week 144 | 1008 | 840 | 1175 |
| Week 192 | 1344 | 1176 | 1511 |
| Week 240 | 1680 | 1512 | 1847 |
| Week 288 | 2016 | 1848 | 2183 |
| Week 336 | 2352 | 2184 | 2519 |
| Week 384 | 2688 | 2520 | 2855 |

The analysis windows for BMD results from DXA, and fasting lipid panel including direct low density lipoprotein (LDL), high density lipoprotein (HDL) and total cholesterol to HDL ratio, are presented in Table 3-4.

Table 3-4. Analysis Windows for BMD Results from DXAand Fasting Lipid Panel

| Visit ID | Nominal Day | Lower Limit | Upper Limit |
|---|---|---|---|
| Baseline | | | 1(14 <sup>a</sup> ) |
| Week 24 | 168 | 2(15a) | 251 |
| Week 48 | 336 | 252 | 419 |
| Week 72 | 504 | 420 | 587 |
| Week 96 | 672 | 588 | 839 (755 <sup>b</sup> ) |
| Week 120 <sup>b</sup> | 840 | 756b | 923b |
| Week 144 | 1008 | 840 (924 <sup>b</sup> ) | 1175 |
| Week 192 | 1344 | 1176 | 1511 |
| Week 240 | 1680 | 1512 | 1847 |
| Week 288 | 2016 | 1848 | 2183 |
| Week 336 | 2352 | 2184 | 2519 |
| Week 384 | 2688 | 2520 | 2855 |

a This applies to DXA only. Upper limit for baseline DXA BMD is Day 14 and lower limit for Week 24 DXA BMD is Day 15.

b This applies to the subjects who consented to Amendment 3.1.

The analysis windows for serum HBsAg (quantitative) and HBV serology are presented in Table 3-5.

Table 3-5. Analysis Windows for Serum HBsAg (Quantitative) and HBV Serology

| Visit ID | Nominal Day | Lower Limit | Upper Limit |
|----------|-------------|-------------|-------------|
| Baseline | | | 1 |
| Week 12 | 84 | 2 | 125 |
| Week 24 | 168 | 126 | 209 |
| Week 36 | 252 | 210 | 293 |
| Week 48 | 336 | 294 | 391 |
| Week 64 | 448 | 392 | 503 |
| Week 80 | 560 | 504 | 615 |
| Week 96 | 672 | 616 | 713 |
| Week 108 | 756 | 714 | 797 |
| Week 120 | 840 | 798 | 881 |
| Week 132 | 924 | 882 | 965 |
| Week 144 | 1008 | 966 | 1091 |
| Week 168 | 1176 | 1092 | 1259 |
| Week 192 | 1344 | 1260 | 1427 |
| Week 216 | 1512 | 1428 | 1595 |
| Week 240 | 1680 | 1596 | 1763 |
| Week 264 | 1848 | 1764 | 1931 |
| Week 288 | 2016 | 1932 | 2099 |
| Week 312 | 2184 | 2100 | 2267 |
| Week 336 | 2352 | 2268 | 2435 |
| Week 360 | 2520 | 2436 | 2603 |
| Week 384 | 2688 | 2604 | 2771 |

The analysis windows for fasting glucose, fasting total cholesterol, fasting triglycerides, renal biomarkers including urine retinol binding protein (RBP) to creatinine ratio, urine beta-2-microglobulin to creatinine ratio, and bone biomarkers including C-type collagen sequence (CTX), procollagen type 1 N-terminal propeptide (P1NP), osteocalcin (OC), and bone specific alkaline phosphatase (bsAP) are presented in Table 3-6.

Table 3-6. Analysis Windows for Fasting Glucose, Fasting Total Cholesterol, Fasting Triglycerides, Renal, and Bone Biomarkers

| Visit ID | Nominal Day | Lower Limit | Upper Limit |
|---|---|---|---|
| Baseline | | | 1 |
| Week 4 | 28 | 2 | 55 |
| Week 12 | 84 | 56 | 125 |
| Week 24 | 168 | 126 | 251 |
| Week 48 | 336 | 252 | 419 |
| Week 72 | 504 | 420 | 587 |
| Week 96 | 672 | 588 | 839 (755 <sup>a</sup> ) |
| Week 120 <sup>a</sup> | 840 | 756ª | 923ª |
| Week 144 | 1008 | 840 (924 <sup>a</sup> ) | 1175 |
| Week 192 | 1344 | 1176 | 1511 |
| Week 240 | 1680 | 1512 | 1847 |
| Week 288 | 2016 | 1848 | 2183 |
| Week 336 | 2352 | 2184 | 2519 |
| Week 384 | 2688 | 2520 | 2855 |

a This applies to the subjects who consented to Amendment 3.1

The analysis window for serum parathyroid hormone (PTH) is presented in Table 3-7.

Table 3-7. Analysis Windows for PTH

| Visit ID | Nominal Day | Lower Limit | Upper Limit |
|----------|-------------|-------------|-------------|
| Baseline | | | 1 |
| Week 4 | 28 | 2 | 41 |
| Week 8 | 56 | 42 | 69 |
| Week 12 | 84 | 70 | 97 |
| Week 16 | 112 | 98 | 125 |
| Week 20 | 140 | 126 | 153 |
| Week 24 | 168 | 154 | 181 |
| Week 28 | 196 | 182 | 209 |
| Week 32 | 224 | 210 | 237 |
| Week 36 | 252 | 238 | 265 |
| Week 40 | 280 | 266 | 293 |
| Week 44 | 308 | 294 | 321 |
| Week 48 | 336 | 322 | 363 |
| Week 56 | 392 | 364 | 419 |
| Week 64 | 448 | 420 | 475 |
| Week 72 | 504 | 476 | 531 |
| Week 80 | 560 | 532 | 587 |
| Week 88 | 616 | 588 | 643 |
| Week 96 | 672 | 644 | 713 |
| Week 108 | 756 | 714 | 797 |
| Week 120 | 840 | 798 | 881 |
| Week 132 | 924 | 882 | 965 |
| Week 144 | 1008 | 966 | 1175 |
| Week 192 | 1344 | 1176 | 1511 |
| Week 240 | 1680 | 1512 | 1847 |
| Week 288 | 2016 | 1848 | 2183 |
| Week 336 | 2352 | 2184 | 2519 |
| Week 384 | 2688 | 2520 | 2855 |

The analysis window for hepatic ultrasound for hepatocellular carcinoma (HCC) surveillance is presented in Table 3-8.

Table 3-8. Analysis Windows for Hepatic Ultrasound

| Visit ID | Nominal Day | Lower Limit | Upper Limit |
|----------|-------------|-------------|-------------|
| Baseline | | | 1 |
| Week 96 | 672 | 588 | 755 |
| Week 120 | 840 | 756 | 923 |
| Week 144 | 1008 | 924 | 1091 |
| Week 168 | 1176 | 1092 | 1259 |
| Week 192 | 1344 | 1260 | 1427 |
| Week 216 | 1512 | 1428 | 1595 |
| Week 240 | 1680 | 1596 | 1763 |
| Week 264 | 1848 | 1764 | 1931 |
| Week 288 | 2016 | 1932 | 2099 |
| Week 312 | 2184 | 2100 | 2267 |
| Week 336 | 2352 | 2268 | 2435 |
| Week 360 | 2520 | 2436 | 2603 |
| Week 384 | 2688 | 2604 | 2855 |

This applies to the subjects who consented to Amendment 3.1.

Data collected after the last dose date will be considered as post-treatment visits. The analysis windows for post-treatment assessments are presented in Table 3-9 and Table 3-10.

Table 3-9. Analysis Windows for Post-Treatment Assessments except HBV Serology

| Visit ID | Nominal Follow-Up Day | Lower Limit | Upper Limit |
|-------------------|-----------------------|-------------|-------------|
| Follow-Up Week 4 | 28 | 1 | 41 |
| Follow-Up Week 8 | 56 | 42 | 69 |
| Follow-Up Week 12 | 84 | 70 | 97 |
| Follow-Up Week 16 | 112 | 98 | 125 |
| Follow-Up Week 20 | 140 | 126 | 153 |
| Follow-Up Week 24 | 168 | 154 | 181 |

Table 3-10. Analysis Windows for Post-Treatment HBV Serology

| Visit ID | Nominal Follow-Up Day | Lower Limit | Upper Limit |
|-------------------|-----------------------|-------------|-------------|
| Follow-Up Week 12 | 84 | 1 | 125 |
| Follow-Up Week 24 | 168 | 126 | 209 |

# 3.7.3. Selection of Data in the Event of Multiple Records in a Window

Depending on the statistical analysis method, single values are required for each analysis window. For example, change from baseline by visit usually requires a single value, whereas a time-to-event analysis would not require 1 value per analysis window. When a single value is needed, the following rule(s) will be used.

For baseline, the last available record on or prior to the first dose of study drug will be selected. For DXA BMD, it is defined as the last value on or prior to Study Day 14. If there are multiple records with the same time or no time recorded on the same day for numeric observations, average will be computed for that day, except that for HBV DNA and Quantitative HBsAg, geometric mean will be taken. If there are multiple records with the same time or no time recorded on the same day for categorical observations, the most conservative value will be taken, eg, negative will be selected over positive for HBeAg and HBsAg, and positive will be selected over negative for HBeAb and HBsAb.

The following specified rules will be used for postbaseline visits:

- **ALT:** The largest value will be included in the analysis when 2 or more ALT values occur within the same visit window.
- **BMD:** The latest record in the window will be selected.
- HBV DNA (IU/mL) and Quantitative HBsAg (IU/mL): The record closest to the nominal day for that visit will be selected. If there are 2 records equidistant from the nominal day, the latest will be selected. If there is more than 1 record on the selected day, the geometric mean will be taken.
- **Serology:** For HBeAg, HBeAb, HBsAg, and HBsAb, the record closest to the nominal day for that visit will be selected. If there are 2 records equidistant from the nominal day, the latest will be selected. If there is more than 1 record on the selected day, the most conservative value will be taken, ie, positive will be selected over negative for HBeAg and HBsAg, and negative will be selected over positive for HBeAb and HBsAb.

For all other laboratory parameters:

- If multiple valid non-missing **numeric** observations exist in a window, then records will be chosen as follows:
  - The record closest to the nominal day for that visit will be selected. If there are 2 records equidistant from the nominal day, the latest will be selected. If there is more than 1 record on the selected day, the average will be taken.
- If multiple valid non-missing **categorical** observations (eg, safety ECG results) exist in a window, then records will be chosen as follows:
  - The most conservative value (eg, abnormal will be selected over normal for safety ECG) within the window will be selected. In the event that 2 values within a window are of equal abnormality, the value collected nearest to the nominal date will be used.

#### 4. SUBJECT DISPOSITION

# 4.1. Subject Enrollment

The number and percentage of subjects randomized each investigator will be summarized by treatment group and overall using the Safety Analysis Set. Similarly, the number and percentage of subjects enrolled in each randomization stratum will be summarized based on interactive voice response system/web response system (IVRS/IWRS) data.

If there are discrepancies between IVRS/IWRS and laboratory data with regard to stratum assignment, a listing of the discrepancies will be provided. If there are differences between randomization stratum for HBV DNA using screening and baseline HBV DNA value, a listing of the differences will be provided.

### 4.2. Disposition of Subjects

The summary of subject disposition will be provided by treatment group and overall. This summary will include the number of subjects screened, screen failure subjects who were not randomized, subjects who met all eligibility criteria and were not randomized, subjects in the Randomized Analysis Set, subjects randomized but not treated, subjects in the Safety Analysis Set, and subjects in FAS.

In addition, the number and percentage of the subjects in the following categories will be summarized using the Safety Analysis Set:

### **Study Drug Completion**

- Remaining on double-blind study treatment up to the data-cut date
- Prematurely discontinued double-blind study treatment prior to the data-cut date (with summary of reasons for discontinuing treatment)
- Completed double-blind study treatment up to the data-cut date
- Entered open-label phase up to the data-cut date

#### **Study Completion**

- Entered 24-week treatment-free follow-up period up to the data-cut date
- Remaining on study up to the data-cut date
- Prematurely discontinued study prior to the data-cut date (with summary of reasons for discontinuing study)

- Started another HBV therapy up to the data-cut date
- Completed protocol-planned duration of the study up to the data-cut date

A data listing of reasons for premature study drug/study discontinuation will be provided.

#### 4.3. Extent of Exposure

Exposure data described below will be summarized for the double-blind phase only.

## 4.3.1. Duration of Exposure to Blinded Study Drug

Duration of exposure to blinded study drug will be defined as (last dose date of blinded study drug – first dose date of blinded study drug + 1), regardless of temporary interruptions in study drug administration, and will be expressed in weeks (recorded to 1 decimal place, eg, 4.5 weeks). If subjects are still on blinded study drug, the latest of blinded study drug start and end dates, and the clinic and laboratory visit dates (excluding the open-label and 24-week treatment-free follow-up visit dates) will be used to impute the last dose date of blinded study drug for calculating the duration of blinded study drug exposure.

Duration of exposure to blinded study drug will be summarized using descriptive statistics (sample size, mean, standard deviation [SD], median, Q1, Q3, minimum, and maximum) and as the number and percentage of subjects exposed for specified periods, eg,  $\geq$  4 weeks (28 days),  $\geq$  8 weeks (56 days), etc.

Summaries will be provided by treatment group for subjects in the Safety Analysis Set.

Time to premature discontinuation of blinded study drug will be analyzed by the Kaplan-Meier method using the Safety Analysis Set. Subjects who completed the blinded study drug will be censored on the last dose date of blinded study drug. Subjects who remain on blinded study drug will be censored on the imputed last dose date of blinded study drug as defined in this section.

#### 4.3.2. Adherence with Blinded Study Drug Regimen

Study drug regimen adherence will be computed based on tablet counts for the active drug only (eg, adherence in TAF group only includes TAF and not placebo for TDF). The numbers of tablets of study drug dispensed and returned are captured on study drug accountability forms.

Adherence (%) of study drug regimen will be calculated as follows:

Adherence (%) = 
$$100 \times \frac{\text{Number of tablets taken}}{\text{Number of tablets prescribed}}$$

= 
$$100 \times \frac{\sum \text{No. of tablets taken at each dispensing period [1]}}{\sum \text{No. of tablets prescribed at each dispensing period [2]}}$$

- [1] Number of tablets taken at a distinct dispensing period for a study drug is calculated as the minimum of (a) the daily number of tablets prescribed for the study drug multiplied by **the duration of treatment** at the dispensing period of the same dispensing date, and (b) the number of tablets taken for the study drug (number of tablets dispensed minus the number of tablets returned). Total number of tablets taken is determined by summing the number of tablets taken from all evaluable dispensing periods.
- [2] Number of tablets prescribed at a distinct dispensing period for a study drug is calculated as the daily number of tablets prescribed for the study drug multiplied by **the duration of treatment** at the dispensing period of the same dispensing date. Total number of tablets prescribed is determined by summing the number of tablets prescribed from all evaluable dispensing periods.

The duration of treatment at a dispensing period for a study drug is calculated as the minimum of (a) the last returned date of the same dispensing period for the study drug, (b) date of premature discontinuation of the study drug, and (c) next dispensing date of the study drug, minus dispensing date of the study drug.

The next dispensing date is the following dispensing date of the study drug regardless of the bottle return date.

For a record where the number of tablets returned was missing (with "Yes" answered for "Was bottle returned?" question), it is assumed the number of tablets returned was 0. If the number of tablets dispensed was missing or any study drug bottle was not returned or the bottle return status was unknown for the same dispensing date, then all records for the same dispensing date for that study drug will be excluded from both denominator and numerator calculation.

Adherence up to Week 48 visit will be calculated for each subject.

The number and percentage of subjects who return at least 1 bottle and have calculable adherence during the study, descriptive statistics for adherence up to Week 48 visit for a study drug regimen (sample size, mean, SD, median, Q1, Q3, minimum, and maximum) along with the number and percentage of subjects belonging to adherence categories (eg, < 80%,  $\ge 80\%$  to < 90%,  $\ge 90\%$  to < 95%,  $\ge 95\%$ ) will be provided by treatment group for the Safety Analysis Set.

#### 4.4. Protocol Deviations

A listing will be provided for subjects in the Randomized Analysis Set who violated at least 1 inclusion or exclusion criterion. The listing will include the unmet criteria. A listing of subjects who received the wrong study treatment will also be provided.

#### 5. BASELINE CHARACTERISTICS

# 5.1. Demographics and Baseline Characteristics

Subject demographic data (eg, age, sex) and baseline characteristics (eg, body weight, height, body mass index [BMI], and Vitamin D) will be summarized by treatment group and overall using descriptive statistics (sample size, mean, SD, median, Q1, Q3, minimum, and maximum) for continuous data and by the number and percentage of subjects for categorical data. Age is calculated as age in years at the first dose of study drug. The summaries of demographic data and baseline subject characteristics will be provided for the Safety Analysis Set.

In addition, the following baseline characteristics and medical history will be summarized:

- BMI categories ( $< 18.5 \text{ kg/m}^2 \text{ [underweight]}, \ge 18.5 25.0 \text{ kg/m}^2 \text{ [normal]},$  $\ge 25.0 - 30.0 \text{ kg/m}^2 \text{ [overweight]}, \text{ and } \ge 30.0 \text{ kg/m}^2 \text{ [obese]})$
- HBV DNA (log<sub>10</sub> IU/mL)
- HBV DNA categories (<  $7 \log_{10} IU/mL$ ,  $\geq 7 \log_{10} IU/mL$  <  $8 \log_{10} IU/mL$ ,  $\geq 8 \log_{10} IU/mL$ )
- ALT (U/L)
- ALT level based on central laboratory normal range ( $\leq$  ULN, > ULN 5  $\times$  ULN, > 5  $\times$  ULN 10  $\times$  ULN, > 10 ULN)
- ALT level based on American Association for the Study of Liver Diseases (AASLD) normal range with the ULN as 19 U/L for female and 30 U/L for male (≤ ULN, > ULN 5 × ULN, > 5 × ULN 10 × ULN, > 10 ULN)
- Estimated GFR by CG, CKD-EPI creatinine, and CKD-EPI Cystatin C methods
- HBeAg status (positive, negative)
- HBeAb status (positive, negative)
- Previous oral nucleoside/nucleotide treatment experience (yes, no)
- Previous interferon experience (yes, no)
- Years positive for HBV
- HBV Genotype (A, B, C, D, E, F, etc)
- Fibrotest score

- Fibrosis stage by fibrotest score (0 0.48, 0.49 0.74, 0.75 1)
- Cirrhosis history (yes, no, indeterminate/unknown)
- Proteinuria by urinalysis (dipstick) (Grade 0, Grade 1, Grade 2, Grade 3)
- Medical history: diabetes mellitus (yes, no), hypertension (yes, no), cardiovascular disease (yes, no), and hyperlipidemia (yes, no)
- Clinical BMD status (normal, osteopenia, osteoporosis)
- Hip fracture and major osteoporotic fracture probabilities estimated using FRAX<sup>®</sup> (see Section 7.3.4)
- IL28B Genotype

Diabetes mellitus, hypertension, cardiovascular disease, and hyperlipidemia above are determined by medical history and/or concomitant medication data, which will be reviewed by the Gilead medical monitor before unblinding.

# **5.2.** Medical History

A listing of medical history data will be provided for the Randomized Analysis Set.

### 6. EFFICACY ANALYSES

For the Week 48 analyses, efficacy data will be summarized for the double-blind phase up to Week 96), with the exception that summaries using M = F approach will be presented up to Week 48 only. All efficacy data up to the Week 48 data-cut including data collected during open-label phase and 24-week treatment-free follow-up period will be listed.

# 6.1. Primary Efficacy Endpoints

# 6.1.1. Definition of the Primary Efficacy Endpoint

The primary efficacy endpoint is the proportion of subjects with HBV DNA < 29 IU/mL at Week 48.

### 6.1.2. Analysis of the Primary Efficacy Endpoint

The primary efficacy analysis will be conducted after the last randomized subject reaches Week 48 or discontinues study drug prematurely. An M = F approach will be employed. In this approach, all missing data will be treated as not achieving the primary endpoint (ie, having HBV DNA  $\geq$  29 IU/mL). The primary analysis will use the FAS.

The number and percentage of subjects who achieved and did not achieve HBV DNA < 29 IU/mL, and reasons for no HBV DNA data at Week 48 will be summarized.

# 6.1.3. Secondary Analysis for the Primary Efficacy Endpoint

A Missing = Excluded (M = E) approach will be used to summarize proportion of subjects with HBV DNA < 29 IU/mL by visit. In this approach, all missing data will be excluded in the computation (ie, missing data points will be excluded from both the numerator and denominator in proportion computation).

A secondary analysis based on the Week 48 PP analysis set will also be performed to evaluate the robustness of the primary analysis of the primary endpoint.

#### 6.1.4. Subgroup Analysis for the Primary Efficacy Endpoint

The analysis of proportion of subjects who achieved HBV DNA < 29 IU/mL at Week 48 will be repeated within each subgroup specified in Section 3.4 using FAS.

For each level of subgroup factors, the number and percentage of subjects who achieved HBV DNA < 29 IU/mL at Week 48 will be summarized.

# 6.2. Secondary Efficacy Endpoints

# 6.2.1. Definition of Secondary Efficacy Endpoints

The secondary efficacy endpoints are as follows:

- The proportion of subjects with plasma HBV DNA < 29 IU/mL at Weeks 96, 144, 240, and 384
- The proportion of subjects with plasma HBV DNA < 29 IU/mL (target not detected) at Weeks 48, 96, 144, 240, and 384
- The proportion of subjects with ALT normalization (by central laboratory and AASLD criteria) at Weeks 48, 96, 144, 240, and 384
- The proportion of subjects with HBsAg loss at Weeks 48, 96, 144, 240, and 384
- The proportion of subjects with HBsAg seroconversion to anti-HBs at Weeks 48, 96, 144, 240, and 384
- The change from baseline in fibrosis as assessed by FibroTest<sup>®</sup> at Weeks 48, 96, 144, 240, and 384
- The incidence of drug resistant mutations at Weeks 48, 96, 144, 240, and 384
- The change from baseline in log<sub>10</sub> (HBV DNA) (IU/mL) at Weeks 48, 96, 144, 240, and 384
- The change from baseline in log<sub>10</sub> (HBsAg) (IU/mL) at Weeks 48, 96, 144, 240, and 384
- The change from baseline in ALT at Weeks 48, 96, 144, 240, and 384

The secondary endpoints beyond Week 96 (Weeks 144, 240, and 384) will not be summarized for the Week 48 analysis. Incidence of drug resistant mutations will be reported in a separate virology report.

For the Week 48 analysis, the following definitions will be used:

- HBsAg loss is defined as HBsAg test result changes from HBsAg positive at baseline to HBsAg negative at a postbaseline visit with baseline HBsAb negative or missing
- HBsAg seroconversion is defined as HBsAg loss and HBsAb test result changes from HBsAb negative or missing at baseline to HBsAb positive at a postbaseline visit
- ALT normalization is defined as ALT > ULN (by central laboratory normal range or AASLD normal range) at baseline but within normal range at a postbaseline visit

Both baseline and postbaseline borderline serology results will be imputed using the following rules:

- HBsAg and HBeAg borderline will be considered as HBsAg positive and HBeAg positive
- HBsAb and HBeAb borderline will be considered as HBsAb negative and HBeAb negative

#### 6.2.2. Analysis Methods for Secondary Efficacy Endpoints

The analyses for the secondary efficacy endpoints will be conducted using the FAS.

All the secondary efficacy endpoints involving proportions will be analyzed using the same statistical method (M = F) applied to the analysis of the primary efficacy endpoint. Sensitivity analyses will be performed using the M = E approach as well.

The change from baseline in  $\log_{10}$  (HBV DNA) (IU/mL),  $\log_{10}$  (HBsAg) (IU/mL), and ALT will be summarized by visit using observed data (ie, missing will be excluded). In addition, the proportion of subjects with HBV DNA < 29 IU/mL, mean change from baseline in  $\log_{10}$  (HBV DNA) (IU/mL),  $\log_{10}$  (HBsAg) (IU/mL), and ALT (U/L) will be plotted with 95% CI over time using observed data for FAS.

Fibrosis assessed by FibroTest<sup>®</sup> at each visit and the change from baseline in fibrotest score will be summarized using descriptive statistics (sample size, mean, SD, median, Q1, Q3, minimum, and maximum) by treatment group. A shift table of fibrosis stage based on fibrotest score by visit will also be provided. Mean change from baseline in fibrotest score will be plotted with 95% CI over time using observed data for FAS. A listing of fibrosis assessment by FibroTest<sup>®</sup> will also be provided.

#### 6.3. Changes From Protocol-Specified Efficacy Analyses

Change from baseline in log<sub>10</sub> (HBV DNA) (IU/mL), log<sub>10</sub> (HBsAg) (IU/mL), and ALT were added in the SAP as secondary efficacy endpoints to fully explore the treatment effect of TAF versus TDF.

Randomized Analysis Set was not defined in the protocol but is added in the SAP.

#### 7. SAFETY ANALYSES

For Week 48 analysis, safety data will be summarized for the double-blind phase only up to Week 96. The upper limit of the least frequent schedule analysis window of Week 96 (Study Day 839) will be used as Week 96 data cut for cumulative summaries of safety events (eg, treatment-emergent AEs, treatment-emergent laboratory abnormalities). All safety data up to the Week 48 data-cut including data collected during the open-label phase and the 24-week treatment-free follow-up period will be included in data listings.

#### 7.1. Adverse Events

# 7.1.1. Adverse Event Dictionary

AEs will be coded using the Medical Dictionary for Regulatory Activities (MedDRA). System Organ Class (SOC), high-level group term (HLGT), high-level term (HLT), preferred term (PT), and lower-level term (LLT) will be attached to the clinical database.

#### 7.1.2. Adverse Event Severity

AEs are graded by the investigator as Grade 1 (mild), Grade 2 (moderate), Grade 3 (severe) or Grade 4 (life threatening) according to toxicity criteria specified in Appendix 5 of the clinical study protocol. The severity grade of events for which the investigator did not record severity will be categorized as "missing" for tabular summaries and data listings, and will be considered the least severe for the purposes of sorting for data presentation.

### 7.1.3. Relationship of AEs to Study Drug

Related AEs are those for which the investigator answers "Yes" to the question "Related to Study Treatment?" in the eCRF. Events for which the investigator did not record relationship to study drug will be considered related to study drug for summary purpose. Data listings will show relationship as missing.

# 7.1.4. Relationship of AEs to Study Procedure

AEs for which 'Yes' is marked for question 'Related to Study Procedures?' in the eCRF will be identified and included in AE listing.

#### 7.1.5. Serious AEs

Serious AEs are those identified as serious in the eCRF, where 'Yes' was marked for 'AE serious'. The clinical database will be reconciled with the serious AE database (from the Drug Safety and Public Health Department) before database finalization.
# 7.1.6. Treatment-Emergent AEs

# 7.1.6.1. Definition of Treatment-Emergent

Treatment-emergent AEs occurring during the double-blind phase are defined as:

- Any AE with an onset date on or after the blinded study drug start date and no later than the study drug stop date for those who discontinued blinded study drug permanently, or
- Any AE with an onset date on or after the blinded study drug start date for those who remain on the blinded study drug, or
- Any AE leading to blinded study drug discontinuation.

Treatment-emergent AEs occurring during the open-label phase are defined as:

- Any AE with an onset date on or after the open-label study drug start date and no later than
  the open-label study drug stop date for those who discontinued open-label study drug
  permanently, or
- Any AE with an onset date on or after the open-label study drug start date for those who remain on the open-label study drug, or
- Any AE leading to open-label study drug discontinuation.

#### 7.1.6.2. Incomplete Dates

If an AE onset date is incomplete or completely missing, the following rules will be used to define treatment-emergent AE during the double-blind and open-label phases:

#### Events with Missing Onset Day and/or Month

The event is treatment-emergent during the double-blind phase if the following criteria are met:

- The month and year (or year) of onset date is the same as or after the month and year (or year) of the first dose of the blinded study drug, and
- For those who discontinued the blinded study drug permanently only: the month and year (or year) of onset date is the same as or before the month and year (or year) of the date of the last dose of the blinded study drug, and
- End date is as follows:
  - The (complete) end date is on or after the first dose date of the blinded study drug, or
  - The month and year (or year) of end date is the same or after the month and year (or year) of the first dose of the blinded study drug, or
  - End date is completely missing

The event is treatment-emergent during the open-label phase if the following criteria are met:

- The month and year (or year) of onset date is the same as or after the month and year (or year) of the first dose of the open-label study drug, and
- For those who discontinued the open-label study drug permanently only: the month and year (or year) of onset date is the same as or before the month and year (or year) of the date of the last dose of the open-label study drug, and
- End date is as follows:
  - The (complete) end date is on or after the first dose date of the open-label study drug, or
  - The month and year (or year) of end date is the same or after the month and year (or year) of the first dose of the open-label study drug, or
  - End date is completely missing

# **Events with Completely Missing Onset Date**

An AE with a completely missing onset date is defined as treatment-emergent AE during the double-blind phase if end date is as follows:

- The (complete) end date is on or after the first dose date of the blinded study drug, or
- The month and year (or year) of end date is the same or after the month and year (or year) of the first dose of the blinded study drug, or
- End date is completely missing

An AE with a completely missing onset date is defined as treatment-emergent AE during the open-label phase if end date is as follows:

- The (complete) end date is on or after the first dose date of the open-label study drug, or
- The month and year (or year) of end date is the same or after the month and year (or year) of the first dose of the open-label study drug, or
- End date is completely missing

#### 7.1.7. Summaries of AEs and Deaths

A brief summary of AEs (ie, the number and percentage of subjects) will be presented by treatment group for the following: (1) any treatment-emergent AE, (2) any Grade 3 or 4 treatment-emergent AE, (3) any Grade 2, 3 or 4 treatment-emergent AE, (4) any treatment-emergent study drug-related AE, (5) any Grade 3 or 4 treatment-emergent study drug-related AE, (6) any Grade 2, 3 or 4 treatment-emergent study drug-related AE, (7) any treatment-emergent serious adverse event (SAE), (8) any treatment-emergent study drug-related SAE,

- (9) any treatment-emergent AE leading to premature study drug discontinuation,(10) any treatment-emergent AE leading to dose modification or study drug interruption, and
- (11) any treatment-emergent death.

Treatment-emergent death refers to death that occurs between the first dose date and the last dose date (inclusive).

Summaries (number and percentage of subjects) of AEs (by SOC, HLT [if specified below], and PT) will be provided by treatment group and overall using the Safety Analysis Set as follows:

- All treatment-emergent AEs summarized by SOC, HLT, and PT
- Any Grade 3 or 4 treatment-emergent AEs
- Any Grade 2, 3, or 4 treatment-emergent AEs
- All treatment-emergent nonserious AEs occurring in at least 5% of subjects in any treatment group (this summary is generated per requirement for reporting in ClinicalTrials.gov)
- All treatment-emergent study drug-related AE summarized by SOC, HLT, and PT
- Any Grade 3 or 4 treatment-emergent study drug-related AEs
- Any Grade 2, 3, or 4 treatment-emergent study drug-related AEs
- All treatment-emergent SAEs
- All treatment-emergent study drug-related SAEs
- All treatment-emergent AEs leading to premature discontinuation from study drug
- All treatment-emergent AEs leading to dose modification or study drug interruption

Multiple events will be counted once only per subject in each summary. For data presentation, SOC (and HLT) will be ordered alphabetically, with PT sorted by decreasing total frequency. For summaries by severity grade, the most severe event will be selected.

In addition to the by-treatment summaries, data listings will be provided for the following:

- All AEs
- Grade 3 and 4 AEs
- SAEs

- Study drug-related SAEs
- Deaths
- AEs leading to premature discontinuation of study drug
- AEs leading to dose modification or study drug interruption

#### 7.1.8. Potential Uveitis Events

Analysis will be performed to detect AEs where the symptoms reported may potentially represent uveitis. The list of PTs for potential uveitis events were defined by selecting eye disorder PTs based on MedDRA 19.1, which will be reviewed and edited by an external ophthalmologist for comprehensiveness.

A summary (number and percentage of subjects) of treatment-emergent potential uveitis events by PT will be provided by treatment group based on the Safety Analysis Set. A data listing of potential uveitis events will be provided.

#### 7.1.9. Potential Cardiovascular Events

Potential cardiovascular events are defined as events with predefined list of MedDRA PTs based on 3 MedDRA SMQs: Ischemic central nervous system vascular conditions, Other ischemic heart disease, and Myocardial infarction, which was provided by Gilead Drug Safety and Public Health representative and reviewed by Gilead medical monitors.

A summary (number and percentage of subjects) of potential treatment-emergent cardiovascular events and serious cardiovascular events by PT will be provided by treatment group based on the Safety Analysis Set. A data listing of potential cardiovascular events will be provided.

#### 7.2. Laboratory Evaluations

Summaries of laboratory data will be provided for the Safety Analysis Set. Analysis will be based on values reported in conventional units.

#### 7.2.1. Summaries of Numeric Laboratory Results

Descriptive statistics (sample size, mean, SD, median, Q1, Q3, minimum, and maximum) will be provided by treatment group for each laboratory test specified in the study protocol as follows:

- Baseline values
- Values at each postbaseline analysis window
- Change from baseline to each postbaseline analysis window
- Percentage change from baseline to each postbaseline analysis window (if specified)

In the case of multiple values in an analysis window, data will be selected for analysis as described in Section 3.7.3.

Median (Q1, Q3) change from baseline in selected safety endpoints including the fasting lipid panel parameters, and fasting glucose over time will be plotted.

#### **Metabolic Assessments**

For the lipid panel and glucose measurements, only those under fasting status will be summarized

Fasting lipid data (including total cholesterol, LDL, HDL and triglycerides) will also be analyzed using the following National Cholesterol Education Program (NCEP) Adult Treatment Panel (ATP) III categories {National Cholesterol Education Program (NCEP) 2001}:

- For total cholesterol (mg/dL): < 200 (desirable), 200-239 (borderline high), and  $\ge 240$  (high)
- For LDL (mg/dL): < 100 (optimal), 100-129 (near optimal/above optimal), 130-159 (borderline high), 160-189 (high), and  $\ge 190$  (very high)
- For HDL (mg/dL): < 40 (low), 40-59 (normal), and  $\ge 60$  (high)
- For triglycerides (mg/dL): < 150 (normal), 150-199 (borderline high), 200-499 (high), and ≥ 500 (very high)

The number and proportion of subjects for the above categories of each lipid parameter will be summarized by its baseline category for each treatment group at each visit.

In addition, the number and proportion of subjects who took lipid modifying medications at the study entry and initiated the medications will be provided, respectively.

A lipid modifying medication is defined as a medication with drug class = "LIPID MODIFYING AGENTS" and CMDECOD containing the wording of "STATIN".

A sensitivity analysis of fasting lipid tests (including total cholesterol, LDL, HDL, triglycerides, and total cholesterol to HDL ratio) will be performed by excluding subjects who took lipid modifying medications at study entry or initiated the medications: baseline, postbaseline, and changes from baseline at Weeks 48 and 96 will be summarized. Only subjects with both baseline and postbaseline values (at Weeks 48 and 96 respectively) will be included in the analysis.

#### **Calcium Corrected for Albumin**

Calcium corrected for albumin will be calculated and summarized. The following formula will be used when both serum calcium and albumin results for a given blood draw are available and serum albumin value is < 4.0 g/dL.

Calcium corrected for albumin (mg/dL) = serum calcium (mg/dL) +  $0.8 \times (4.0 - \text{albumin (g/dL)})$ .

When albumin value is  $\geq$  4.0 g/dL, the actual calcium results will be used. Toxicity grading for calcium will be applied based on the corrected values.

# 7.2.2. Graded Laboratory Values

The criteria specified in the protocol will be used to grade laboratory results as Grade 0, Grade 1 (mild), Grade 2 (moderate), Grade 3 (severe) or Grade 4 (life-threatening). Grade 0 includes all values that do not meet criteria for an abnormality of at least Grade 1. Some laboratory tests have criteria for both increased and decreased levels; analysis for each direction (ie, increased, decreased) will be presented separately.

For triglycerides, LDL, and total cholesterol, the protocol-specified toxicity grade scale is for fasting test values; non-fasting lipid results (or lipid results without known fasting status) will not be graded or summarized by toxicity grades.

If any laboratory toxicity grading scale overlaps with normal reference ranges (eg, Grade 1 scale overlaps with normal reference ranges), laboratory values within normal range will not be graded except for lipid tests.

# 7.2.2.1. Treatment-Emergent Laboratory Abnormalities

Treatment-emergent laboratory abnormalities occuring in the double-blind phase are defined as values that increase by at least 1 toxicity grade from baseline at any postbaseline visit up to and including the last does date of the blinded study drug (or 'last dose date of the blinded study drug + 1' for those who enter the open-label phase) for those who discontinued blinded study drug prematurely, or values that increase by at least 1 toxicity grade from baseline at any postbaseline visit for those who are still on the blinded study drug. If the relevant baseline laboratory data are missing, any laboratory abnormality of at least Grade 1 will be considered treatment-emergent.

Treatment-emergent laboratory abnormalities occurring in the open-label phase are defined as values that increase by at least 1 toxicity grade from the open-label baseline at any open-label postbaseline visit up to and including the last dose date of open-label study drug for those who discontinued open-label study drug prematurely, or values that increase by at least 1 toxicity grade from the open-label baseline at any open-label postbaseline visit for those who are still on the open-label study drug. For the analyses of abnormalities occurring during open-label treatment, baseline will be considered to be the last available record on or prior to Open-Label Study Day 1.

Fasting glucose and nonfasting glucose are graded based on different grading scales. Treatment-emergent laboratory abnormalities will be summarized for fasting glucose. Since nonfasting glucose was not assessed at baseline, the maximum postbaseline grade will be summarized.

#### 7.2.2.2. Treatment-Emergent Marked Laboratory Abnormalities

Treatment-emergent marked laboratory abnormalities occurring in the double-blind phase are defined as values that worsen by at least 3 grades from baseline at any postbaseline visit up to and including the last dose date of the blinded study drug (or 'last dose date of the blinded study drug + 1' for those who enter the open-label phase) for those who discontinued study drug

prematurely, or values that worsen by at least 3 grades from baseline at any postbaseline visit for those who are still on blinded study drug. If relevant baseline laboratory data are missing, any laboratory abnormalities of at least Grade 3 or 4 will be considered as treatment-emergent marked laboratory abnormalities.

Treatment-emergent marked laboratory abnormalities occurring in the open-label phase are defined as values that worsen by at least 3 grades from the open-label baseline at any open-label postbaseline visit up to and including the last dose date of open-label study drug for those who discontinued open-label study drug prematurely, or values that worsen by at least 3 grades from the open-label baseline at any open-label postbaseline visit for those who are still on open-label study drug.

### 7.2.2.3. Summaries of Laboratory Abnormalities

The following summaries (number and percentage of subjects) of laboratory abnormalities will be provided by treatment group (subjects categorized according to most severe abnormality grade):

- Treatment-emergent laboratory abnormalities
- Treatment-emergent Grade 3 and 4 laboratory abnormalities
- Treatment-emergent marked laboratory abnormalities

For all summaries of laboratory abnormalities, the denominator is the number of subjects with any nonmissing postbaseline value in the given study period. A listing of treatment-emergent Grade 3 or 4 laboratory abnormalities will be provided.

#### 7.2.3. ALT Elevation

An ALT elevation is defined as serum ALT  $> 2 \times$  baseline value and  $> 10 \times$  ULN, with or without associated symptoms. Confirmed ALT elevation (ALT flare) is defined as ALT elevations at 2 consecutive postbaseline visits. All treatment-emergent ALT elevations including confirmed ALT elevations will be summarized for the double-blind phase. All treatment-emergent and nontreatment-emergent ALT elevations will be included in a listing.

# 7.3. Bone Safety Analyses

#### 7.3.1. Bone Mineral Density (BMD)

For BMD analysis during the double-blind phase, any available on-treatment record on or prior to Open-label Study Day 14 will be included into the double-blind phase summary for those who enter the open-label phase after completion of the double-blind phase.

Percentage change from baseline in hip BMD and spine BMD a will be summarized by treatment group and visit using descriptive statistics for subjects in the Hip and Spine DXA Analysis Sets, respectively.

Missing values for hip and spine BMD will be imputed using LOCF up to Week 96 for the analyses of percentage change from baseline. The last on-treatment postbaseline observation will be carried forward to impute the missing value. Baseline observation will not be carried forward.

Percentage change from baseline in observed hip and spine BMD will be analyzed similarly provided up to Week 96.

Observed BMD values will be used for all the analyses described below:

For each subject and each visit, the clinical BMD status will be defined for hip and spine BMD based on the corrected t-score in Table 7-1.

Table 7-1. Normal, Osteopenia, and Osteoporosis as Defined by T-score

| Clinical Status | BMD T-score |
|-----------------|------------------------|
| Normal | $t$ -score $\geq -1.0$ |
| Osteopenia | -2.5 ≤ t-score < -1.0 |
| Osteoporosis | t-score < -2.5 |

The number and percentage of subjects in each clinical BMD status (normal, osteopenia, and osteoporosis) will be summarized by visit and by baseline clinical status for both hip and spine.

For each subject and each visit, percentage change from baseline in hip BMD and spine BMD will be classified into 10 categories: > 7% decrease, > 5% to  $\leq$  7% decrease, > 3% to  $\leq$  5% decrease, > 1% to  $\leq$  3% decrease, > 0 to  $\leq$  1% decrease, 0 to  $\leq$  1% increase, > 1% to  $\leq$  3% increase, > 5% to  $\leq$  7% increase, and > 7% increase. The number and percentage of subjects in each category will be summarized by visit.

Median (Q1, Q3) and mean (95% CI) of percentage change from baseline in observed hip and spine BMD over time will be plotted by treatment group. Listings of hip and spine DXA results will be provided.

#### 7.3.2. Bone Biomakers

Bone biomarkers include serum CTX, P1NP, PTH, OC, and bsAP.

Baseline, postbaseline, change from baseline, and percentage change from baseline in bone biomarkers will be summarized by treatment group and visit using descriptive statistics.

Median (Q1, Q3) percentage change from baseline in bone biomarkers over time will be plotted by treatment group. A listing of bone biomarker data will be provided.

#### 7.3.3. Fracture Events

The PTs for fracture events were defined based on both Standardised MedDRA Query (SMQ) of Osteoporosis/Osteopenia and HLGT of Fractures from MedDRA 19.1. These PTs were reviewed by the Gilead medical monitor before unblinding to identify appropriate fracture event PTs from the SMQ of Osteoporosis/Osteopenia and HLGT of Fractures. Treatment-emergent fracture events will be summarized based on the identified PTs from SMQ alone and both SMQ and HLGT combined. The number and percentage of subjects who experienced fracture events will be summarized by treatment group. A data listing of fracture events will be provided.

### 7.3.4. Assessment of Fracture Probability

Fracture probabilities will be assessed using FRAX®, a computer based algorithm developed by the World Health Organization (WHO; http://www.shef.ac.uk/FRAX).

The FRAX algorithm is based on individual patient models that integrate the risks associated with clinical risk factors as well as BMD at the femoral neck. The algorithm provides both the 10-year probability of hip fracture and the 10-year probability of a major osteoporotic fracture (clinical spine, forearm, hip, or shoulder fracture).

The FRAX model is constructed from real data in population-based cohorts around the world that have a limited age range. For an age below 40 or above 90 years, the tool will calculate the probability of fracture at the age of 40 or 90 years, respectively. Due to the age limitation, 2 sets of analyses of fracture probabilities will be performed.

In the first set of analysis, summaries of baseline and change from baseline in the 10-year probabilities of hip fracture, as well as major osteoporotic fracture will be presented by treatment group and visit for subjects aged between 40 and 90 years.

In the second set of analysis, the above-specified analysis will be performed to include all subjects, where subjects with an age below 40 or above 90 years will be treated as having an age of 40 or 90 years, respectively, in computing their fracture probabilities.

Data listings of fracture risk assessment questionnaire and FRAX fracture probabilities will be provided.

#### 7.3.5. Bone Events

The PTs for bone events were defined by selecting relevant bone PTs based on MedDRA 19.1. The predefined list of PTs, included Osteoporosis/Osteopenia and Osteonecrosis SMQ, HLGT of Fractures, and HLTs relevant to bone disorders, bone metabolism, and bone procedures. These PTs were reviewed by the Gilead medical monitor before unblinding to identify appropriate bone event PTs. The number and percentage of subjects who experienced treatment-emergent bone events will be summarized by treatment group. A data listing of bone events will be provided.

# 7.4. Renal Safety Analyses

#### 7.4.1. Confirmed Renal Abnormalities

Confirmed renal abnormalities are defined as follows:

- Confirmed increase from baseline in creatinine of at least 0.5 mg/dL or
- Confirmed CLcr by CG below 50 mL/min or
- Confirmed phosphorous < 2 mg/dL

Treatment-emergent confirmed renal abnormalities will be summarized for double-blind phase. All confirmed renal abnormalities including those occurred during open-label phase and 24-week treatment-free follow-up period will be listed.

#### 7.4.2. Serum Creatinine

The baseline and change from baseline in serum creatinine at Week 48 will be summarized using descriptive statistics.

Missing values for serum creatinine will be imputed using LOCF up to Week 96 for the analyses of change from baseline in serum creatinine. The last on-treatment postbaseline observation will be carried forward to impute the missing value. Baseline observation will not be carried forward.

Change from baseline in observed serum creatinine will be analyzed similarly.

For all of the other renal safety analyses, observed creatinine values will be used.

Median (Q1, Q3) and mean (95% CI) of change from baseline in observed serum creatinine overtime will be plotted by treatment group.

#### 7.4.3. Estimated Glomerular Filtration Rate

The following formulae will be used to calculate eGFR:

• CG:

```
eGFRcg (mL/min) = [(140 - age (yrs)) \times weight (kg) \times (0.85 \text{ if female})] / (SCr (mg/dL) \times 72), where weight is actual total body mass in kilograms, and SCr is serum creatinine.
```

CKD-EPI Creatinine Based:

```
eGFRCKD-EPI, creatinine (mL/min/1.73 m<sup>2</sup>) = 141 \times \min(SCr/\kappa, 1)^{\alpha} \times \max(SCr/\kappa, 1)^{-1.209} \times 0.993^{Age} \times 1.018 (if female) \times 1.159 (if black),
```

where  $\kappa$  is 0.7 for females and 0.9 for males,  $\alpha$  is –0.329 for females and –0.411 for males, min indicates the minimum of SCr/ $\kappa$  or 1, and max indicates the maximum of SCr/ $\kappa$  or 1 {Levey 2009}.

CKD-EPI Cystatin C based:

```
eGFR<sub>CKD-EPI, cys</sub>C (mL/min/1.73 m<sup>2</sup>) = 133 \times min(SCys/0.8, 1)^{-0.499} \times max(SCys/0.8, 1)^{-1.328} \times 0.996^{age} [× 0.932 if female],
```

where SCys is serum cystatin C.

Change from baseline in eGFRcg and eGFRckd-EPI, creatinine at each postbaseline visit will also be provided.

The number and proportion of subjects with decrease from baseline of  $\geq$  25% and  $\geq$  50% in eGFRcg and eGFR<sub>CKD-EPI, creatinine</sub> will be summarized by treatment groups.

The number and proportion of subjects in each stage of CKD will be summarized by baseline stages of CKD for the double-blind phase up to Week 96.

The stages of CKD are defined as follows:

- Stage 1: eGFR<sub>CG</sub>  $\geq$  90 mL/min
- Stage 2: eGFR<sub>CG</sub>  $\geq$  60 and  $\leq$  90 mL/min
- Stage 3: eGFR<sub>CG</sub>  $\geq$  30 and  $\leq$  60 mL/min
- Stage 4:  $eGFR_{CG} < 30 \text{ mL/min}$

Cystatin C will be collected for each subject at baseline visit (protocol amendment 2.1 and after) and whenever their postbaseline eGFR by CG < 50 mL/min. Therefore, eGFR<sub>CKD-EPI, cysC</sub> will be summarized as the baseline disease characteristics only. All postbaseline eGFR<sub>CKD-EPI, cysC</sub> with percentage change from baseline will be listed.

Median (Q1, Q3) change from baseline in  $eGFR_{CG}$  and  $eGFR_{CKD-EPI, creatinine}$  over time will be plotted.

#### 7.4.4. Treatment-Emergent Proteinuria (Dipstick)

Treatment-emergent proteinuria by urinalysis (dipstick) through Week 48 will be summarized by treatment group. A listing of subjects with treatment-emergent proteinuria will be provided.

# 7.4.5. Urine Creatinine, Urine RBP to Creatinine Ratio and Beta-2-microglobulin to Creatinine Ratio

Baseline, postbaseline, change from baseline and percentage change from baseline in urine creatinine, urine RBP to creatinine ratio and beta-2-microglobulin to creatinine ratio will be summarized by treatment group and visit using descriptive statistics. Median (Q1, Q3) percentage change from baseline over time will be plotted by treatment group.

### 7.4.6. Proteinuria by Quantitative Assessment

Baseline, postbaseline, changes from baseline, and percentage change from baseline in UPCR and UACR will be summarized by treatment group and visit using descriptive statistics.

The number and proportion of subjects with UPCR  $\leq$  200 mg/g versus > 200 mg/g will be summarized by baseline category for each postbaseline visit {KDIGO Guideline Development Staff 2013}.

Median (Q1, Q3) percentage change from baseline over time will be plotted by treatment group.

#### 7.4.7. Other Renal Biomarkers

Other renal biomarkers include TmP/GFR, FEPO<sub>4</sub>, and FEUA.

TmP/GFR based on serum creatinine {Barth 2000} will be calculated as follows:

$$TmP/GFR = TRP \times SPO_4$$
 if  $TRP \le 0.86$   
 $TmP/GFR = 0.3 \times TRP/[1 - (0.8 \times TRP)] \times SPO_4$  if  $TRP > 0.86$ 

where TRP (tubular reabsoprtion of phosphate) is calculated by:

$$TRP = 1 - \frac{UPO_4}{SPO_4} \times \frac{SCr}{UCr}$$

where SCr is serum creatinine concentration (mg/dL), UPO<sub>4</sub> is urine phosphate concentration (mg/dL), SPO<sub>4</sub> is serum phosphate concentration, and UCr is urine creatinine concentration (mg/dL).

Urine FEPO4 will be calculated as follows:

$$FEPO_4$$
 (%) = (SCr × UPO<sub>4</sub>) / (SPO<sub>4</sub> × UCr) × 100 (%)

**Urine FEUA** will be calculated as follows:

FEUA (%) = 
$$(SCr \times UUa) / (SUa \times UCr) \times 100$$
 (%)

where UUa and SUa are urine and serum uric acid (mg/dL), respectively.

The baseline, postbaseline, and change from baseline in TmP/GFR, FEPO<sub>4</sub>, and FEUA will be summarized by treatment group and visit using descriptive statistics.

Median (Q1, Q3) change from baseline in TmP/GFR, FEPO<sub>4</sub>, and FEUA over time will be plotted by treatment group. A listing of renal biomarker data will be provided.

# 7.5. Ophthalmologic Assessment

As no Ophthalmologic assessment was performed in China, no analysis will be conducted.

# 7.6. Body Weight

Body weight at each visit and change from baseline in body weight will be summarized using descriptive statistics (sample size, mean, SD, median, Q1, Q3, minimum, and maximum) by treatment group for each postbaseline analysis window. In the case of multiple values in an analysis window, data will be selected for analysis as described in Section 3.7.3.

### 7.7. Prior Hepatitis B Medications

Prior HBV medications will be summarized by treatment group. A listing of prior HBV medications will also be provided.

#### 7.8. Concomitant Medications

Concomitant medications (ie, medications other than study drug that are taken while receiving study drug) will be coded using the WHO Drug Dictionary. The WHO preferred name and drug code will be attached to the clinical database. Use of concomitant medications from study Day 1 up to the date of last dose of blinded study drug will be summarized (number and percentage of subjects) for the double-blind phase by treatment group and WHO drug class and preferred name. Multiple drug use (by preferred name) will be counted only once per subject. The summary will be sorted alphabetically by drug class and then by decreasing total frequency within a class.

If the start or stop date of concomitant medications is incomplete, the month and year (or year alone if month is not recorded) of start or stop date will be used to determine if the medications are concomitant as follows. The medication is concomitant for the double-blind phase if the month and year of start or stop (or year of the start or stop) of the medication do not meet any of following criteria:

- The month and year of start of the medication is after the date of the last dose of blinded study drug
- The month and year of stop of the medication is before the date of the first dose of blinded study drug

If the start and stop date of the medications are not missing, and the start date is not after the last dose date of double-blind phase and the stop date is not before the first dose date of double-blind phase, or the medications are marked as ongoing and start date is on or before the last dose date of double-blind phase, the medications are considered concomitant of double-blind phase.

Summaries of concomitant medications will be provided for the Safety Analysis Set. Subjects with any concomitant medication use will also be listed.

# 7.9. Electrocardiogram (ECG) Results

The number and percentage of subjects in the Safety Analysis Set with an investigator's ECG assessment of normal, abnormal but not clinically significant, or abnormal and clinically significant will be summarized by treatment group and by baseline result for each visit.

A by-subject listing of safety ECG results will be provided including treatment, assessment date and time, and ECG results.

# 7.10. Other Safety Measures

A data listing will be provided for subjects experiencing pregnancy during the study.

Listings of cirrhosis and hepatocellular carcinoma assessment results will be provided.

Alcohol use data will also be listed.

# 7.11. Changes From Protocol-Specified Safety Analyses

Treatment-emergent proteinuria was not included as a key secondary safety endpoint in protocol amendment 3.1 and is added in the SAP.

As no Ophthalmologic assessment was performed in China, no analysis will be conducted.

Comparison of the safety and tolerability of TAF versus TDF for the treatment of HBeAg-negative, CHB beyond Week 48 during the double-blind phase in treatment-naive and treatment-experienced subjects was not included as a secondary objective of this study and is added in the SAP.

# 8. REFERENCES

- Barth JH, Jones RG, Payne RB. Calculation of renal tubular reabsorption of phosphate: the algorithm performs better than the nomogram. Ann Clin Biochem 2000;37 ( Pt 1):79-81.
- KDIGO Guideline Development Staff. KDIGO 2012 Clinical Practice Guideline for the Evaluation and Management of Chronic Kidney Disease. Kidney international. Supplement 2013;3 (1):v-150.
- Levey AS, Stevens LA, Schmid CH, Zhang YL, Castro AF, 3rd, Feldman HI, et al. A new equation to estimate glomerular filtration rate. Ann Intern Med 2009;150 (9):604-12.
- National Cholesterol Education Program (NCEP). Detection, Evaluation, and Treatment of High Blood Cholesterol in Adults (Adult Treatment Panel III) Executive Summary. National Institute of Health May, 2001.

# 9. SOFTWARE

SAS® (SAS Institute Inc., Version 9.4, Cary, NC) is to be used for all programming of tables, listings, and figures.

nQuery Advisor® (Statistical Solutions Ltd., Version 6.0, Cork, Ireland) was used for the sample size and power calculation.

FRAX® (WHO Collaborating Center for Metabolic Bone Disease, University of Sheffield, UK) is to be used for the 10-year probabilities of hip fracture or a major osteoporotic fracture.

# 10. SAP REVISION

| Revision Date<br>(dd month yyyy) | Section | Summary of Revision | Reason for Revision |
|---|---|---|---|

# 11. APPENDICES

Appendix 1. Table of Contents for Statistical Tables, Figures, and Listings

Appendix 1. Table of Contents
Appendix 2. Fracture Events
Appendix 3. Bone Events
Appendix 4. Potential Uveitis

Appendix 5. Potential Cardiovascular or Cerebrovascular Events

# Appendix 1. Table of Contents for Statistical Tables, Figures, and Listings

Table of contents of TFLs for Week 48 analysis is as follows:

| Table Number | Title | Analysis Set |
|---|---|---|
| 1 | Enrollment by Region, Country, and Investigator | Safety Analysis Set |
| 2 | Enrollment by Randomization Stratum | Safety Analysis Set |
| 3 | Subject Disposition | All Screened Subjects |
| 4 | Analysis Set | Randomized Analysis Set |
| 5 | Demographics and Baseline Characteristics | Safety Analysis Set |
| 6 | Baseline Disease Characteristics | Safety Analysis Set |
| 7 | Risk Factors for HBV Infections | Safety Analysis Set |
| 8 | Prior HBV Medications | Safety Analysis Set |
| 9 | Duration of Exposure to Blinded Study Drug | Safety Analysis Set |
| 10.1 | Time to Premature Discontinuation of Blinded Study Drug (Kaplan-Meier Estimate) | Safety Analysis Set |
| 10.2 | Supporting Table for Table 11.1: Percentiles of Time to Premature Discontinuation of Blinded Study Drug | Safety Analysis Set |
| 10.3 | Supporting Table for Table 11.1: Listing of Time and Censoring Status of Premature Discontinuation of Blinded Study Drug | Safety Analysis Set |
| 11 | Adherence to Blinded Study Drug | Safety Analysis Set |
| 12 | HBV DNA Outcome at Week 48 (HBV DNA Cutoff at 29 IU/mL, Missing = Failure) | Full Analysis Set |
| 13 | HBV DNA Outcome at Week 48 (HBV DNA Cutoff at 29 IU/mL, Missing = Failure) | Week 48 PP Analysis Set |
| 14.1 | Proportion of Subjects with HBV DNA < 29 IU/mL by Visit (Missing = Failure) | Full Analysis Set |
| 14.2 | Proportion of Subjects with HBV DNA < 29 IU/mL by Visit (Missing = Excluded) | Full Analysis Set |
| 15 | Proportion of Subjects with HBV DNA < 29 IU/mL by Visit (Missing = Failure) | Week 48 PP Analysis Set |
| 16 | Proportion of Subjects with HBV DNA < 29 IU/mL at Week 48 by Subgroup (Missing = Failure) | Full Analysis Set |
| 17 | HBV DNA (log <sub>10</sub> IU /mL) and Change from Baseline in HBV DNA (log <sub>10</sub> IU /mL) by Visit | Full Analysis Set |
| 18.1 | Proportion of Subjects with HBeAg Loss/Seroconversion by Visit (Missing = Failure) | Serologically Evaluable<br>Full Analysis Set |
| 18.2 | Proportion of Subjects with HBeAg Loss/Seroconversion by Visit (Missing = Excluded) | Serologically Evaluable<br>Full Analysis Set |
| 19.1 | Proportion of Subjects with HBsAg Loss/Seroconversion by Visit (Missing = Failure) | Serologically Evaluable<br>Full Analysis Set |
| 19.2 | Proportion of Subjects with HBsAg Loss/Seroconversion by Visit (Missing = Excluded) | Serologically Evaluable<br>Full Analysis Set |

| 20 HBsAg (log <sub>10</sub> IU /mL) and Change from Baseline in HBsAg (log <sub>10</sub> IU /mL) by Visit | Table Number | Title | Analysis Set |
|---|---|---|---|
| Normal Range (Missing = Failure) | 20 | | Full Analysis Set |
| Normal Range (Missing = Excluded) Full Analysis Set | 21.1.1 | | Full Analysis Set |
| Normal Range (Missing = Failure) | 21.1.2 | | Full Analysis Set |
| Normal Range (Missing = Excluded) Full Analysis Set | 21.2.1 | | Full Analysis Set |
| Central Lab Normal Range (Missing = Failure) Baseline ALT > ULN | 21.2.2 | | Full Analysis Set |
| Central LabNormal Range (Missing = Excluded) Baseline ALT > ULN | 22.1.1 | | Full Analysis Set with Baseline ALT > ULN |
| AASLD Normal Range (Missing = Failure) Proportion of Subjects with ALT Normalization by Visit by AASLD Normal Range (Missing = Excluded) ALT (U/L) and Change from Baseline in ALT (U/L) by Visit Full Analysis Set with Baseline ALT > ULN ALT (U/L) and Change from Baseline in Fibrotest Score by Visit Full Analysis Set Fibrotest Score and Change from Baseline in Fibrotest Score by Visit Full Analysis Set Shift Table of Fibrosis Stage by FibroTest* by Visit Full Analysis Set Treatment-Emergent Adverse Events: Overall Summary Safety Analysis Set Treatment-Emergent Adverse Events Occurring in >= 5% of Subjects in Any Treatment Group Grade 2, 3, or 4 Treatment-Emergent Adverse Events Grade 3 or 4 Treatment-Emergent Adverse Events Treatment-Emergent Study Drug-Related Adverse Events Grade 2, 3, or 4 Treatment-Emergent Study Drug-Related Adverse Events Grade 2, 3, or 4 Treatment-Emergent Study Drug-Related Adverse Events Grade 3 or 4 Treatment-Emergent Study Drug-Related Adverse Events Grade 3 or 4 Treatment-Emergent Study Drug-Related Adverse Events Grade 3 or 4 Treatment-Emergent Study Drug-Related Adverse Events Grade 3 or 4 Treatment-Emergent Study Drug-Related Adverse Events Treatment-Emergent Serious Adverse Events Safety Analysis Set Treatment-Emergent Serious Adverse Events Safety Analysis Set Treatment-Emergent Study Drug-Related Serious Adverse Events Treatment-Emergent Study Drug-Related Serious Adverse Events Treatment-Emergent Adverse Events Leading to Premature Study Drug Discontinuation Treatment-Emergent Adverse Events Leading to Dose Modification or Study Drug Interruption Treatment-Emergent Potential Uveitis Events Safety Analysis Set | 22.1.2 | | |
| AASLD Normal Range (Missing = Excluded) ALT (U/L) and Change from Baseline in ALT (U/L) by Visit Full Analysis Set Fibrotest Score and Change from Baseline in Fibrotest Score by Visit Full Analysis Set Shift Table of Fibrosis Stage by FibroTest® by Visit Full Analysis Set Shift Table of Fibrosis Stage by FibroTest® by Visit Full Analysis Set Treatment-Emergent Adverse Events: Overall Summary Safety Analysis Set Treatment-Emergent Nonserious Adverse Events Occurring in >= 5% of Subjects in Any Treatment Group Grade 2, 3, or 4 Treatment-Emergent Adverse Events Grade 3 or 4 Treatment-Emergent Adverse Events Full Analysis Set Safety Analysis Set Treatment-Emergent Nonserious Adverse Events Occurring in >= 5% of Subjects in Any Treatment Group Grade 2, 3, or 4 Treatment-Emergent Adverse Events Grade 3 or 4 Treatment-Emergent Adverse Events Grade 3 or 4 Treatment-Emergent Study Drug-Related Adverse Events Grade 2, 3, or 4 Treatment-Emergent Study Drug-Related Safety Analysis Set Grade 3 or 4 Treatment-Emergent Study Drug-Related Adverse Events Grade 3 or 4 Treatment-Emergent Study Drug-Related Safety Analysis Set Treatment-Emergent Serious Adverse Events Treatment-Emergent Study Drug-Related Serious Adverse Full Analysis Set Safety Analysis Set Safety Analysis Set Safety Analysis Set Treatment-Emergent Study Drug-Related Serious Adverse Events Treatment-Emergent Adverse Events Leading to Premature Safety Analysis Set Treatment-Emergent Adverse Events Leading to Dose Modification or Study Drug Interruption Treatment-Emergent Potential Uveitis Events Safety Analysis Set | 22.2.1 | | |
| Fibrotest Score and Change from Baseline in Fibrotest Score by Visit Shift Table of Fibrosis Stage by FibroTest® by Visit Full Analysis Set Treatment-Emergent Adverse Events: Overall Summary Safety Analysis Set Treatment-Emergent Nonserious Adverse Events Occurring in Safety Analysis Set Treatment-Emergent Nonserious Adverse Events Occurring in Safety Analysis Set Full Analysis Set Treatment-Emergent Nonserious Adverse Events Occurring in Safety Analysis Set Full Analysis Set Treatment-Emergent Nonserious Adverse Events Occurring in Safety Analysis Set Full Analysis Set Safety Analysis Set Treatment-Emergent Nonserious Adverse Events Occurring in Safety Analysis Set Full Analysis Set Safety Analysis Set Safety Analysis Set Safety Analysis Set Treatment-Emergent Study Drug-Related Adverse Events Safety Analysis Set Safety Analysis Set Grade 2, 3, or 4 Treatment-Emergent Study Drug-Related Adverse Events Grade 3 or 4 Treatment-Emergent Study Drug-Related Safety Analysis Set Adverse Events Treatment-Emergent Serious Adverse Events Safety Analysis Set Treatment-Emergent Study Drug-Related Serious Adverse Events Treatment-Emergent Study Drug-Related Serious Adverse Events Treatment-Emergent Adverse Events Leading to Premature Study Drug Discontinuation Treatment-Emergent Adverse Events Leading to Dose Modification or Study Drug Interruption Treatment-Emergent Potential Uveitis Events Safety Analysis Set | 22.2.2 | | |
| by Visit Shift Table of Fibrosis Stage by FibroTest® by Visit Full Analysis Set Treatment-Emergent Adverse Events: Overall Summary Safety Analysis Set Treatment-Emergent Adverse Events Treatment-Emergent Nonserious Adverse Events Occurring in >= 5% of Subjects in Any Treatment Group Grade 2, 3, or 4 Treatment-Emergent Adverse Events Grade 3 or 4 Treatment-Emergent Adverse Events Treatment-Emergent Study Drug-Related Adverse Events Grade 2, 3, or 4 Treatment-Emergent Study Drug-Related Adverse Events Grade 2, 3, or 4 Treatment-Emergent Study Drug-Related Adverse Events Grade 2, 3, or 4 Treatment-Emergent Study Drug-Related Adverse Events Grade 3 or 4 Treatment-Emergent Study Drug-Related Adverse Events Grade 3 or 4 Treatment-Emergent Study Drug-Related Adverse Events Treatment-Emergent Serious Adverse Events Treatment-Emergent Serious Adverse Events Treatment-Emergent Study Drug-Related Serious Adverse Events Treatment-Emergent Study Drug-Related Serious Adverse Events Treatment-Emergent Adverse Events Events Treatment-Emergent Adverse Events Leading to Premature Safety Analysis Set Treatment-Emergent Adverse Events Leading to Dose Modification or Study Drug Interruption Treatment-Emergent Potential Uveitis Events Safety Analysis Set | 23 | ALT (U/L) and Change from Baseline in ALT (U/L) by Visit | Full Analysis Set |
| Treatment-Emergent Adverse Events: Overall Summary Treatment-Emergent Adverse Events Treatment-Emergent Nonserious Adverse Events Occurring in >= 5% of Subjects in Any Treatment Group Grade 2, 3, or 4 Treatment-Emergent Adverse Events Grade 3 or 4 Treatment-Emergent Adverse Events Treatment-Emergent Study Drug-Related Adverse Events Grade 2, 3, or 4 Treatment-Emergent Study Drug-Related Adverse Events Grade 2, 3, or 4 Treatment-Emergent Study Drug-Related Adverse Events Grade 3 or 4 Treatment-Emergent Study Drug-Related Adverse Events Grade 3 or 4 Treatment-Emergent Study Drug-Related Safety Analysis Set Grade 3 or 4 Treatment-Emergent Study Drug-Related Adverse Events Treatment-Emergent Serious Adverse Events Treatment-Emergent Serious Adverse Events Treatment-Emergent Study Drug-Related Serious Adverse Events Treatment-Emergent Adverse Events Leading to Premature Study Drug Discontinuation Treatment-Emergent Adverse Events Leading to Dose Modification or Study Drug Interruption Treatment-Emergent Potential Uveitis Events Safety Analysis Set Treatment-Emergent Potential Uveitis Events Safety Analysis Set | 24 | | Full Analysis Set |
| 27Treatment-Emergent Adverse EventsSafety Analysis Set28Treatment-Emergent Nonserious Adverse Events Occurring in >= 5% of Subjects in Any Treatment GroupSafety Analysis Set29Grade 2, 3, or 4 Treatment-Emergent Adverse EventsSafety Analysis Set30Grade 3 or 4 Treatment-Emergent Adverse EventsSafety Analysis Set31Treatment-Emergent Study Drug-Related Adverse EventsSafety Analysis Set32Grade 2, 3, or 4 Treatment-Emergent Study Drug-Related Adverse EventsSafety Analysis Set33Grade 3 or 4 Treatment-Emergent Study Drug-Related Adverse EventsSafety Analysis Set34Treatment-Emergent Serious Adverse EventsSafety Analysis Set35Treatment-Emergent Study Drug-Related Serious Adverse EventsSafety Analysis Set36Treatment-Emergent Adverse Events Leading to Premature Study Drug DiscontinuationSafety Analysis Set37Treatment-Emergent Adverse Events Leading to Dose Modification or Study Drug InterruptionSafety Analysis Set38Treatment-Emergent Potential Uveitis EventsSafety Analysis Set | 25 | Shift Table of Fibrosis Stage by FibroTest® by Visit | Full Analysis Set |
| Treatment-Emergent Nonserious Adverse Events Occurring in >= 5% of Subjects in Any Treatment Group Grade 2, 3, or 4 Treatment-Emergent Adverse Events Grade 3 or 4 Treatment-Emergent Adverse Events Treatment-Emergent Study Drug-Related Adverse Events Grade 2, 3, or 4 Treatment-Emergent Study Drug-Related Adverse Events Grade 2, 3, or 4 Treatment-Emergent Study Drug-Related Adverse Events Grade 2, 3, or 4 Treatment-Emergent Study Drug-Related Safety Analysis Set Grade 3 or 4 Treatment-Emergent Study Drug-Related Safety Analysis Set Grade 3 or 4 Treatment-Emergent Study Drug-Related Safety Analysis Set Treatment-Emergent Serious Adverse Events Treatment-Emergent Study Drug-Related Serious Adverse Events Treatment-Emergent Adverse Events Leading to Premature Safety Analysis Set Treatment-Emergent Adverse Events Leading to Dose Modification or Study Drug Interruption Treatment-Emergent Potential Uveitis Events Safety Analysis Set Safety Analysis Set | 26 | Treatment-Emergent Adverse Events: Overall Summary | Safety Analysis Set |
| Safety Analysis Set | 27 | Treatment-Emergent Adverse Events | Safety Analysis Set |
| 30Grade 3 or 4 Treatment-Emergent Adverse EventsSafety Analysis Set31Treatment-Emergent Study Drug-Related Adverse EventsSafety Analysis Set32Grade 2, 3, or 4 Treatment-Emergent Study Drug-Related Adverse EventsSafety Analysis Set33Grade 3 or 4 Treatment-Emergent Study Drug-Related Adverse EventsSafety Analysis Set34Treatment-Emergent Serious Adverse EventsSafety Analysis Set35Treatment-Emergent Study Drug-Related Serious Adverse EventsSafety Analysis Set36Treatment-Emergent Adverse Events Leading to Premature Study Drug DiscontinuationSafety Analysis Set37Treatment-Emergent Adverse Events Leading to Dose Modification or Study Drug InterruptionSafety Analysis Set38Treatment-Emergent Potential Uveitis EventsSafety Analysis Set | 28 | | Safety Analysis Set |
| Treatment-Emergent Study Drug-Related Adverse Events Grade 2, 3, or 4 Treatment-Emergent Study Drug-Related Adverse Events Grade 3 or 4 Treatment-Emergent Study Drug-Related Adverse Events Treatment-Emergent Serious Adverse Events Treatment-Emergent Study Drug-Related Serious Adverse Events Treatment-Emergent Study Drug-Related Serious Adverse Events Treatment-Emergent Study Drug-Related Serious Adverse Events Treatment-Emergent Adverse Events Leading to Premature Safety Analysis Set Treatment-Emergent Adverse Events Leading to Dose Modification or Study Drug Interruption Treatment-Emergent Adverse Events Leading to Dose Modification or Study Drug Interruption Treatment-Emergent Potential Uveitis Events Safety Analysis Set | 29 | Grade 2, 3, or 4 Treatment-Emergent Adverse Events | Safety Analysis Set |
| Grade 2, 3, or 4 Treatment-Emergent Study Drug-Related Adverse Events Grade 3 or 4 Treatment-Emergent Study Drug-Related Adverse Events Treatment-Emergent Serious Adverse Events Treatment-Emergent Study Drug-Related Serious Adverse Events Treatment-Emergent Study Drug-Related Serious Adverse Events Treatment-Emergent Adverse Events Leading to Premature Study Drug Discontinuation Treatment-Emergent Adverse Events Leading to Dose Modification or Study Drug Interruption Treatment-Emergent Adverse Events Leading to Dose Modification or Study Drug Interruption Treatment-Emergent Potential Uveitis Events Safety Analysis Set Safety Analysis Set | 30 | Grade 3 or 4 Treatment-Emergent Adverse Events | Safety Analysis Set |
| Adverse Events Grade 3 or 4 Treatment-Emergent Study Drug-Related Adverse Events Treatment-Emergent Serious Adverse Events Safety Analysis Set Treatment-Emergent Study Drug-Related Serious Adverse Events Treatment-Emergent Study Drug-Related Serious Adverse Events Treatment-Emergent Adverse Events Leading to Premature Study Drug Discontinuation Treatment-Emergent Adverse Events Leading to Dose Modification or Study Drug Interruption Treatment-Emergent Potential Uveitis Events Safety Analysis Set Safety Analysis Set Safety Analysis Set | 31 | Treatment-Emergent Study Drug-Related Adverse Events | Safety Analysis Set |
| Adverse Events Adverse Events Treatment-Emergent Serious Adverse Events Safety Analysis Set Treatment-Emergent Study Drug-Related Serious Adverse Events Treatment-Emergent Adverse Events Leading to Premature Study Drug Discontinuation Treatment-Emergent Adverse Events Leading to Dose Modification or Study Drug Interruption Treatment-Emergent Adverse Events Leading to Dose Modification or Study Drug Interruption Treatment-Emergent Potential Uveitis Events Safety Analysis Set Safety Analysis Set | 32 | | Safety Analysis Set |
| Treatment-Emergent Study Drug-Related Serious Adverse Events Safety Analysis Set Treatment-Emergent Adverse Events Leading to Premature Study Drug Discontinuation Treatment-Emergent Adverse Events Leading to Dose Modification or Study Drug Interruption Treatment-Emergent Potential Uveitis Events Safety Analysis Set Safety Analysis Set | 33 | | Safety Analysis Set |
| Events Treatment-Emergent Adverse Events Leading to Premature Safety Analysis Set Treatment-Emergent Adverse Events Leading to Dose Safety Analysis Set Treatment-Emergent Adverse Events Leading to Dose Modification or Study Drug Interruption Treatment-Emergent Potential Uveitis Events Safety Analysis Set Safety Analysis Set | 34 | Treatment-Emergent Serious Adverse Events | Safety Analysis Set |
| Study Drug Discontinuation Treatment-Emergent Adverse Events Leading to Dose Modification or Study Drug Interruption Safety Analysis Set Safety Analysis Set Safety Analysis Set Safety Analysis Set | 35 | , , | Safety Analysis Set |
| Modification or Study Drug Interruption Safety Analysis Set Treatment-Emergent Potential Uveitis Events Safety Analysis Set | 36 | | Safety Analysis Set |
| | 37 | | Safety Analysis Set |
| 39 Treatment-Emergent Potential Cardiovascular Events Safety Analysis Set | 38 | Treatment-Emergent Potential Uveitis Events | Safety Analysis Set |
| | 39 | Treatment-Emergent Potential Cardiovascular Events | Safety Analysis Set |

| Table Number | Title | Analysis Set |
|---|---|---|
| 40 | Treatment-Emergent Potential Serious Cardiovascular Events | Safety Analysis Set |
| 41 | Treatment-Emergent Laboratory Abnormalities | Safety Analysis Set |
| 42 | Treatment-Emergent Grade 3 or 4 Laboratory Abnormalities | Safety Analysis Set |
| 43 | Treatment-Emergent Marked Laboratory Abnormalities | Safety Analysis Set |
| 44 | Treatment-Emergent ALT Elevation | Safety Analysis Set |
| 45.1 | Hematology: Summary of Hemoglobin (g/dL) by Visit | Safety Analysis Set |
| 45.2 | Hematology: Summary of Hematocrit (%) by Visit | Safety Analysis Set |
| 45.3 | Hematology: Summary of MCH (pg) by Visit | Safety Analysis Set |
| 45.4 | Hematology: Summary of MCHC (g/dL) by Visit | Safety Analysis Set |
| 45.5 | Hematology: Summary of MCV (fL) by Visit | Safety Analysis Set |
| 45.6 | Hematology: Summary of RBC (10^6/uL) by Visit | Safety Analysis Set |
| 45.7 | Hematology: Summary of Absolute Basophils (10^3/uL) by Visit | Safety Analysis Set |
| 45.8 | Hematology: Summary of Absolute Eosinophils (10^3/uL) by Visit | Safety Analysis Set |
| 45.9 | Hematology: Summary of Absolute Lymphocytes (10^3/uL) by Visit | Safety Analysis Set |
| 45.10 | Hematology: Summary of Absolute Monocytes (10^3/uL) by Visit | Safety Analysis Set |
| 45.11 | Hematology: Summary of Absolute Neutrophils (10^3/uL) by Visit | Safety Analysis Set |
| 45.12 | Hematology: Summary of Platelet Count (10^3/uL) by Visit | Safety Analysis Set |
| 45.13 | Hematology: Summary of WBC (10^3/uL) by Visit | Safety Analysis Set |
| 46.1 | Chemistry: Summary of Bicarbonate (mEq/L) by Visit | Safety Analysis Set |
| 46.2 | Chemistry: Summary of Calcium (Albumin Corrected, mg/dL) by Visit | Safety Analysis Set |
| 46.3 | Chemistry: Summary of Chloride (mEq/L) by Visit | Safety Analysis Set |
| 46.4 | Chemistry: Summary of Magnesium (mg/dL) by Visit | Safety Analysis Set |
| 46.5 | Chemistry: Summary of Phosphorus (mg/dL) by Visit | Safety Analysis Set |
| 46.6 | Chemistry: Summary of Potassium (mEq/L) by Visit | Safety Analysis Set |
| 46.7 | Chemistry: Summary of Sodium (mEq/L) by Visit | Safety Analysis Set |
| 46.8 | Chemistry: Summary of Alkaline Phosphatase (U/L) by Visit | Safety Analysis Set |
| 46.9 | Chemistry: Summary of AST (U/L) by Visit | Safety Analysis Set |
| 46.10 | Chemistry: Summary of Amylase (U/L) by Visit | Safety Analysis Set |
| 46.11 | Chemistry: Summary of Lipase (U/L) by Visit | Safety Analysis Set |
| 46.12 | Chemistry: Summary of Total Bilirubin (mg/dL) by Visit | Safety Analysis Set |
| 46.13 | Chemistry: Summary of Direct Bilirubin (mg/dL) by Visit | Safety Analysis Set |
| 46.14 | Chemistry: Summary of Indirect Bilirubin (mg/dL) by Visit | Safety Analysis Set |
| 46.15 | Chemistry: Summary of GGT (U/L) by Visit | Safety Analysis Set |

| Table Number | Title | Analysis Set |
|---|---|---|
| 46.16 | Chemistry: Summary of LDH (U/L) by Visit | Safety Analysis Set |
| 46.17 | Chemistry: Summary of Blood Urea Nitrogen (BUN, mg/dL) by Visit | Safety Analysis Set |
| 46.18 | Chemistry: Summary of Uric Acid (mg/dL) by Visit | Safety Analysis Set |
| 46.19 | Chemistry: Summary of Albumin (g/dL) by Visit | Safety Analysis Set |
| 46.20 | Chemistry: Summary of Creatine Kinase (U/L) by Visit | Safety Analysis Set |
| 46.21 | Chemistry: Summary of Total Protein (g/dL) by Visit | Safety Analysis Set |
| 47.1.1 | Metabolic Assessments: Summary of Fasting Total Cholesterol (mg/dL) by Visit | Safety Analysis Set |
| 47.1.2 | Metabolic Assessments: Shift Table of Fasting Total Cholesterol (mg/dL) by Visit | Safety Analysis Set |
| 47.2.1 | Metabolic Assessments: Summary of Fasting Direct LDL (mg/dL) by Visit | Safety Analysis Set |
| 47.2.2 | Metabolic Assessments: Shift Table of Fasting Direct LDL (mg/dL) by Visit | Safety Analysis Set |
| 47.3.1 | Metabolic Assessments: Summary of Fasting HDL (mg/dL) by Visit | Safety Analysis Set |
| 47.3.2 | Metabolic Assessments: Shift Table of Fasting HDL (mg/dL) by Visit | Safety Analysis Set |
| 47.4 | Metabolic Assessments: Summary of Fasting Total Cholesterol to HDL Ratio by Visit | Safety Analysis Set |
| 47.5.1 | Metabolic Assessments: Summary of Fasting Triglycerides (mg/dL) by Visit | Safety Analysis Set |
| 47.5.2 | Metabolic Assessments: Shift Table of Fasting Triglycerides (mg/dL) by Visit | Safety Analysis Set |
| 47.6 | Metabolic Assessments: Summary of Fasting Glucose (mg/dL) by Visit | Safety Analysis Set |
| 47.7.1 | Summary of Subjects Taking Lipid Modifying Medications at Study Entry | Safety Analysis Set |
| 47.7.2 | Summary of Subjects Initiating Lipid Modifying Medications during Double-Blind Phase | Safety Analysis Set |
| 47.8.1 | Summary of Fasting Total Cholesterol (mg/dL) at Baseline and Week 48 (Excluding Subjects Taking any Lipid Modifying Medication) | Safety Analysis Set |
| 47.8.2 | Summary of Fasting Direct LDL (mg/dL) at Baseline and Week 48 (Excluding Subjects Taking any Lipid Modifying Medication) | Safety Analysis Set |
| 47.8.3 | Summary of Fasting HDL (mg/dL) at Baseline and Week 48 (Excluding Subjects Taking any Lipid Modifying Medication) | Safety Analysis Set |
| 47.8.4 | Summary of Fasting Triglycerides (mg/dL) at Baseline and<br>Week 48 (Excluding Subjects Taking any Lipid Modifying<br>Medication) | Safety Analysis Set |

| Table Number | Title | Analysis Set |
|---|---|---|
| 47.8.5 | Summary of Fasting Total Cholesterol to HDL Ratio at Baseline and Week 48 (Excluding Subjects Taking any Lipid Modifying Medication) | Safety Analysis Set |
| 48.1.1 | Percentage Change from Baseline in Hip Bone Mineral Density by Visit (LOCF Imputation) | Hip DXA Analysis Set |
| 48.1.2 | Percentage Change from Baseline in Hip Bone Mineral Density by Visit (Observed Data) | Hip DXA Analysis Set |
| 48.2.1 | Percentage Change from Baseline in Spine Bone Mineral Density<br>by Visit (LOCF Imputation) | Spine DXA Analysis Set |
| 48.2.2 | Percentage Change from Baseline in Spine Bone Mineral Density<br>by Visit (Observed Data) | Spine DXA Analysis Set |
| 49.1 | Clinical Hip Bone Mineral Density Status by Baseline Status and Visit | Hip DXA Analysis Set |
| 49.2 | Clinical Spine Bone Mineral Density Status by Baseline Status and Visit | Spine DXA Analysis Set |
| 50.1 | Gradation of the Percentage Change in Hip Bone Mineral<br>Density by Visit | Hip DXA Analysis Set |
| 50.2 | Gradation of the Percentage Change in Spine Bone Mineral<br>Density by Visit | Spine DXA Analysis Set |
| 51.1 | Bone Biomarkers: Summary of Serum C-type Collagen<br>Sequence (CTX, ng/mL) by Visit | Safety Analysis Set |
| 51.2 | Bone Biomarkers: Summary of Serum Bone Procollagen Type 1<br>N-terminal Propeptide (P1NP, ng/mL) by Visit | Safety Analysis Set |
| 51.3 | Bone Biomarkers: Summary of Serum Parathyroid Hormone (PTH, pg/mL) by Visit | Safety Analysis Set |
| 51.4 | Bone Biomarkers: Summary of Osteocalcin (OC, ng/mL) by Visit | Safety Analysis Set |
| 51.5 | Bone Biomarkers: Summary of Bone Specific Alkaline<br>Phosphatase (bsAP, ug/L) by Visit | Safety Analysis Set |
| 52 | Treatment-Emergent Fracture Events | Safety Analysis Set |
| 53.1.1 | Summary of 10 Year Probability of Hip Fracture (%) by Visit (Age ≥ 40 Years) | Hip DXA Analysis Set |
| 53.1.2 | Summary of 10 Year Probability of Hip Fracture (%) by Visit (All Subjects) | Hip DXA Analysis Set |
| 53.2.1 | Summary of 10 Year Probability of Major Osteoporotic Fracture (%) by Visit (Age ≥ 40 Years) | Hip DXA Analysis Set |
| 53.2.2 | Summary of 10 Year Probability of Major Osteoporotic Fracture (%) by Visit (All Subjects) | Hip DXA Analysis Set |
| 54 | Treatment-Emergent Bone Events | Safety Analysis Set |
| 55 | Treatment-Emergent Confirmed Renal Laboratory Abnormality | Safety Analysis Set |
| 56.1 | Summary of Serum Creatinine (mg/dL) by Visit (LOCF Imputation) | Safety Analysis Set |
| 56.2 | Summary of Serum Creatinine (mg/dL) by Visit (Observed Data) | Safety Analysis Set |

| Table Number | Title | Analysis Set |
|---|---|---|
| 57.1 | Summary of Estimated Glomerular Filtration Rate (eGFR) by Cockeroft-Gault (mL/min) by Visit | Safety Analysis Set |
| 57.2 | Summary of Estimated Glomerular Filtration Rate (eGFR) by CKD-EPI Creatinine (mL/min/1.73 m^2) by Visit | Safety Analysis Set |
| 57.3 | Summary of Subjects with Percentage Decrease from Baseline >= 25% and >= 50% in eGFR | Safety Analysis Set |
| 57.4 | Shift Table of Chronic Kidney Disease (CKD) Stage by Baseline CKD Stage | Safety Analysis Set |
| 58 | Treatment-Emergent Proteinuria by Urinalysis (Dipstick) | Safety Analysis Set |
| 59.1 | Renal Biomarkers: Summary of Urine Creatinine (mg/dL) by<br>Visit | Safety Analysis Set |
| 59.2 | Renal Biomarkers: Summary of Urine RBP to Creatinine Ratio (ug/g) by Visit | Safety Analysis Set |
| 59.3 | Renal Biomarkers: Summary of Urine Beta-2-Microglobulin to Creatinine Ratio (ug/g) by Visit | Safety Analysis Set |
| 59.4 | Renal Biomarkers: Summary of Urine Protein to Creatinine Ratio (UPCR, mg/g) by Visit | Safety Analysis Set |
| 59.5 | Renal Biomarkers: Summary of Urine Albumin to Creatinine<br>Ratio (UACR, mg/g) by Visit | Safety Analysis Set |
| 60.1 | Shift Table of Urine Protein to Creatinine Ratio (UPCR) Category (≤ 200 vs > 200 mg/g) by Baseline Category | Safety Analysis Set |
| 60.2 | Shift Table of Urine Albumin to Creatinine Ratio (UACR) Category (< 30 vs ≥ 30 mg/g) by Baseline Category | Safety Analysis Set |
| 61 | Summary of TmP/GFR Ratio (mg/dL) by Visit | Safety Analysis Set |
| 62 | Summary of Urine Fractional Excretion of Phosphate (FEPO <sub>4</sub> , %) by Visit | Safety Analysis Set |
| 63 | Summary of Urine Fractional Excretion of Uric Acid (FEUA, %) by Visit | Safety Analysis Set |
| 64 | Summary of Body Weight (kg) by Visit | Safety Analysis Set |
| 65 | Concomitant Medications During Study by Drug Class and<br>Generic Name | Safety Analysis Set |
| 66 | Safety ECG Results by Baseline ECG Category and Visit | Safety Analysis Set |

| Figure Number | Title | Analysis Set |
|---|---|---|
| 1 | Subject Disposition | All Screened Subjects |
| 2 | Time to Premature Discontinuation of Blinded Study Drug (Kaplan-Meier Estimate) | Safety Analysis Set |
| 3.1 | Proportion of Subjects with HBV DNA < 29 IU/mL by Visit:<br>Missing = Failure | Full Analysis Set |
| 3.2 | Proportion of Subjects with HBV DNA < 29 IU/mL by Visit:<br>Missing = Excluded | Full Analysis Set |
| 4 | Proportion of Subjects with HBV DNA < 29 IU/mL by Visit:<br>Missing = Failure | Week 48 PP Analysis Set |
| 5 | Mean and 95% CIs of Change from Baseline in HBV DNA (log <sub>10</sub> IU/mL) by Visit (Observed Data) | Full Analysis Set |
| 6 | Mean and 95% CIs of Change from Baseline in HBsAg (log <sub>10</sub> IU/mL) by Visit (Observed Data) | Full Analysis Set |
| 7.1 | Proportion of Subjects with ALT Normalization by Visit by<br>Central Laboratory Normal Range: Missing = Failure | Full Analysis Set |
| 7.2 | Proportion of Subjects with ALT Normalization by Visit by AASLD Normal Range: Missing = Failure | Full Analysis Set |
| 8 | Mean and 95% CIs of Change from Baseline in ALT (U/L) (Observed Data) | Full Analysis Set |
| 9 | Mean and 95% CIs of Change from Baseline in Fibrotest Score (Observed Data) | Full Analysis Set |
| 10.1 | Median (Q1, Q3) of Change from Baseline in Fasting Total<br>Cholesterol (mg/dL) by Visit | Safety Analysis Set |
| 10.2 | Median (Q1, Q3) of Change from Baseline in Fasting Direct LDL (mg/dL) by Visit | Safety Analysis Set |
| 10.3 | Median (Q1, Q3) of Change from Baseline in Fasting HDL (mg/dL) by Visit | Safety Analysis Set |
| 10.4 | Median (Q1, Q3) of Change from Baseline in Fasting Total<br>Cholesterol to HDL Ratio by Visit | Safety Analysis Set |
| 10.5 | Median (Q1, Q3) of Change from Baseline in Fasting<br>Triglycerides (mg/dL) by Visit | Safety Analysis Set |
| 10.6 | Median (Q1, Q3) of Change from Baseline in Fasting Glucose (mg/dL) by Visit | Safety Analysis Set |
| 11.1.1 | Median (Q1, Q3) of Percentage Change from Baseline in Hip<br>Bone Mineral Density by Visit (Observed Data) | Hip DXA Analysis Set |
| 11.1.2 | Median (Q1, Q3) of Percentage Change from Baseline in Spine<br>Bone Mineral Density by Visit (Observed Data) | Spine DXA Analysis Set |
| 11.2.1 | Mean and 95% CIs of Percentage Change from Baseline in Hip<br>Bone Mineral Density by Visit (Observed Data) | Hip DXA Analysis Set |

| Figure Number | Title | Analysis Set |
|---|---|---|
| 11.2.2 | Mean and 95% CIs of Percentage Change from Baseline in Spine<br>Bone Mineral Density by Visit (Observed Data) | Spine DXA Analysis Set |
| 12.1 | Median (Q1, Q3) of Percentage Change from Baseline in Serum C-type Collagen Sequence (CTX) by Visit | Safety Analysis Set |
| 12.2 | Median (Q1, Q3) of Percentage Change from Baseline in Serum<br>Bone Procollagen Type 1 N-terminal Propeptide (P1NP) by Visit | Safety Analysis Set |
| 12.3 | Median (Q1, Q3) of Percentage Change from Baseline in Serum<br>Parathyroid Hormone (PTH) by Visit | Safety Analysis Set |
| 12.4 | Median (Q1, Q3) of Percentage Change from Baseline in Osteocalcin (OC) by Visit | Safety Analysis Set |
| 12.5 | Median (Q1, Q3) of Percentage Change from Baseline in Bone<br>Specific Alkaline Phosphatase (bsAP) by Visit | Safety Analysis Set |
| 13.1 | Median (Q1, Q3) of Change from Baseline in Serum Creatinine (mg/dL) by Visit (Observed Data) | Safety Analysis Set |
| 13.2 | Mean and 95% CIs of Change from Baseline in Serum Creatinine (mg/dL) by Visit (Observed Data) | Safety Analysis Set |
| 14.1 | Median (Q1, Q3) of Change from Baseline in Estimated GFR by Cockcroft-Gault (mL/min) by Visit | Safety Analysis Set |
| 14.2 | Median (Q1, Q3) of Change from Baseline in Estimated GFR by CKD-EPI Creatinine (mL/min/1.73 m^2) by Visit | Safety Analysis Set |
| 15.1 | Median (Q1, Q3) of Percentage Change from Baseline in Urine RBP to Creatinine Ratio by Visit | Safety Analysis Set |
| 15.2 | Median (Q1, Q3) of Percentage Change from Baseline in Urine<br>Beta-2-Microglobulin to Creatinine Ratio by Visit | Safety Analysis Set |
| 16.1 | Median (Q1, Q3) of Percentage Change from Baseline in Urine<br>Protein to Creatinine Ratio (UPCR) by Visit | Safety Analysis Set |
| 16.2 | Median (Q1, Q3) of Percentage Change from Baseline in Urine<br>Albumin to Creatinine Ratio (UACR) by Visit | Safety Analysis Set |
| 17 | Median (Q1, Q3) of Change from Baseline in TmP/GFR Ratio (mg/dL) by Visit | Safety Analysis Set |
| 18 | Median (Q1, Q3) of Change from Baseline in Urine Fractional Excretion of Phosphate (FEPO <sub>4</sub> , %) by Visit | Safety Analysis Set |
| 19 | Median (Q1, Q3) of Change from Baseline in Urine Fractional Excretion of Uric Acid (FEUA, %) by Visit | Safety Analysis Set |

| Listing Number | Title | Analysis Set |
|---|---|---|
| 1 | Subject Profiles | Randomized Analysis Set |
| 2 | Subject Disposition | Randomized Analysis Set |
| 3.1 | Subjects Who Were Excluded from Analysis Sets | Randomized Analysis Set |
| 3.2 | Subjects Who Were in the Full Analysis Set but Not in the PP Analysis Set | Full Analysis Set |
| 4.1 | Enrollment | Randomized Analysis Set |
| 4.2 | Eligibility Criteria Not Met | Randomized Analysis Set |
| 4.3 | Enrollment Summary | Subjects Not Enrolled |
| 5.1 | HBV DNA Stratification Discrepancies Between HBV DNA<br>Stratum Entered into IWRS and Actual Screening HBV DNA<br>Stratum | Randomized Analysis Set |
| 5.2 | HBV DNA Level Classification Difference Between<br>Randomization Stratum by Screening and Baseline HBV DNA<br>Level | Randomized Analysis Set |
| 6 | Subjects Who Received the Wrong Study Drug Treatment (Other Than That They Were Randomized to) | Randomized Analysis Set |
| 7 | Demographics and Baseline Characteristics | Randomized Analysis Set |
| 8.1 | Baseline Disease Characteristics (Part I) | Randomized Analysis Set |
| 8.2 | Baseline Disease Characteristics (Part II) | Randomized Analysis Set |
| 9 | Medical History | Randomized Analysis Set |
| 10 | Risk Factors for HBV Infection | Randomized Analysis Set |
| 11 | Prior HBV Medications | Randomized Analysis Set |
| 12 | Study Drug Administration | Randomized Analysis Set |
| 13 | Study Drug Accountability and Adherence | Randomized Analysis Set |
| 14 | HBV DNA | Randomized Analysis Set |
| 15 | Subjects with HBV DNA value above or at 29 IU/mL at Week 48 (or Last Visit if Prior to Week 48) | Randomized Analysis Set |
| 16 | HBV Serology | Randomized Analysis Set |
| 17 | Subjects with HBeAg Loss and/or HBeAg Seroconversion | Randomized Analysis Set:<br>Subjects with Serologically<br>Evaluable Data |
| 18 | Subjects with HBsAg Loss and/or HBsAg Seroconversion | Randomized Analysis Set:<br>Subjects with Serologically<br>Evaluable Data |
| 19 | Fibrosis Assessment by FibroTest® | Randomized Analysis Set |
| 20 | All Adverse Events | Randomized Analysis Set |
| 21 | Grade 3 and 4 Adverse Events | Randomized Analysis Set |

| <b>Listing Number</b> | Title | Analysis Set |
|---|---|---|
| 22 | Serious Adverse Events | Randomized Analysis Set |
| 23 | Study Drug-Related Serious Adverse Events | Randomized Analysis Set |
| 24 | Adverse Events Leading to Premature Study Drug Discontinuation | Randomized Analysis Set |
| 25 | Adverse Events Leading to Dose Modification or Study Drug<br>Interruption | Randomized Analysis Set |
| 26 | Death Report | Randomized Analysis Set |
| 27 | Potential Uveitis Events | Randomized Analysis Set |
| 28 | Potential Cardiovascular Events | Randomized Analysis Set |
| 29 | Graded Laboratory Abnormalities | Randomized Analysis Set |
| 30 | Grade 3 or 4 Laboratory Abnormalities | Randomized Analysis Set |
| 31 | Laboratory Tests Related to Hepatic Function | Randomized Analysis Set |
| 32 | Hepatic Ultrasound for Hepatocellular Carcinoma (HCC)<br>Surveillance | Randomized Analysis Set |
| 33 | ALT Elevation | Randomized Analysis Set |
| 34.1 | Clinical Laboratory Data: Hematology (Part I) | Randomized Analysis Set |
| 34.2 | Clinical Laboratory Data: Hematology (Part II) | Randomized Analysis Set |
| 34.3 | Clinical Laboratory Data: Hematology (Part III) | Randomized Analysis Set |
| 34.4 | Clinical Laboratory Data: Hematology (Part IV) | Randomized Analysis Set |
| 35.1 | Clinical Laboratory Data: Chemistry (Part I) | Randomized Analysis Set |
| 35.2 | Clinical Laboratory Data: Chemistry (Part II) | Randomized Analysis Set |
| 35.3 | Clinical Laboratory Data: Chemistry (Part III) | Randomized Analysis Set |
| 35.4 | Clinical Laboratory Data: Chemistry (Part IV) | Randomized Analysis Set |
| 36 | Metabolic Assessment: Glucose and Lipid Panel | Randomized Analysis Set |
| 37.1 | Clinical Laboratory Data: Urinalysis (Part I) | Randomized Analysis Set |
| 37.2 | Clinical Laboratory Data: Urinalysis (Part II) | Randomized Analysis Set |
| 37.3 | Clinical Laboratory Data: Urinalysis (Part III) | Randomized Analysis Set |
| 38.1 | Clinical Laboratory Data: Urine Chemistry (Part I) | Randomized Analysis Set |
| 38.2 | Clinical Laboratory Data: Urine Chemistry (Part II) | Randomized Analysis Set |
| 39 | Clinical Laboratory Data: HAV/HCV/HDV/HEV/HIV Serology | Randomized Analysis Set |
| 40 | Clinical Laboratory Data: Pregnancy Test | Randomized Analysis Set |
| 41 | Reference Ranges for Laboratory Tests | |
| 42.1 | Hip Bone Mineral Density Results | Randomized Analysis Set:<br>Subjects with Any<br>Hip DXA Data |

| Listing Number | Title | Analysis Set |
|---|---|---|
| 42.2 | Spine Bone Mineral Density Results | Randomized Analysis Set:<br>Subjects with Any Spine<br>DXA Data |
| 43.1 | Subjects with > 5% Decline in Hip Bone Mineral Density | Randomized Analysis Set:<br>Subjects with Any Hip<br>DXA Data |
| 43.2 | Subjects with > 5% Decline in Spine Bone Mineral Density | Randomized Analysis Set:<br>Subjects with Any Spine<br>DXA Data |
| 44.1 | Bone Biomarkers Results (Part I) | Randomized Analysis Set |
| 44.2 | Bone Biomarkers Results (Part II) | Randomized Analysis Set |
| 45 | Fracture Events | Randomized Analysis Set |
| 46.1 | FRAX 10 Year Fracture Probabilities | Randomized Analysis Set:<br>Subjects with Any<br>Hip DXA Data |
| 46.2 | FRAX Risk Assessment Questionnaire | Randomized Analysis Set |
| 47 | Bone Events | Randomized Analysis Set |
| 48 | Confirmed Renal Abnormalities | Randomized Analysis Set |
| 49 | Serum Creatinine and Estimated Glomerular Filtration Rate (eGFR) | Randomized Analysis Set |
| 50 | Subjects with eGFR < 50 (by CG, CKD-EPI Creatinine, or CKD-EPI Cystatin C) | Randomized Analysis Set |
| 51 | Treatment-Emergent Proteinuria | Randomized Analysis Set |
| 52.1 | Renal Biomarkers Results (Part I) | Randomized Analysis Set |
| 52.2 | Renal Biomarkers Results (Part II) | Randomized Analysis Set |
| 53.1 | Subjects with UPCR > 200 mg/g | Randomized Analysis Set |
| 53.2 | Subjects with UACR ≥ 30 mg/g | Randomized Analysis Set |
| 54 | Vital Signs | Randomized Analysis Set |
| 55 | Concomitant Medications | Randomized Analysis Set |
| 56 | 12-Lead Electrocardiogram Results | Randomized Analysis Set |
| 57 | Pregnancy Report | Randomized Analysis Set |
| 58 | Cirrhosis Assessment | Randomized Analysis Set |
| 59 | Hepatocellular Carcinoma Assessment | Randomized Analysis Set |
| 60 | Alcohol Use | Randomized Analysis Set |

# **Appendix 2.** Fracture Events

The selected PTs of fracture events from SMQ of Osteoporosis/Osteopenia and HLGT of Fractures are listed as follows:

| | Selected Preferred Terms | Selection Type |
|----|------------------------------------------|----------------|
| 1 | Acetabulum fracture | cSMQ+cHLGT |
| 2 | Ankle fracture | cHLGT |
| 3 | Atypical femur fracture | cSMQ+cHLGT |
| 4 | Atypical fracture | cHLGT |
| 5 | Avulsion fracture | cHLGT |
| 6 | Bone fissure | cHLGT |
| 7 | Bone fragmentation | cHLGT |
| 8 | Cervical vertebral fracture | cSMQ+cHLGT |
| 9 | Chance fracture | cHLGT |
| 10 | Clavicle fracture | cHLGT |
| 11 | Closed fracture manipulation | cSMQ |
| 12 | Comminuted fracture | cHLGT |
| 13 | Complicated fracture | cHLGT |
| 14 | Compression fracture | cHLGT |
| 15 | Craniofacial fracture | cHLGT |
| 16 | Epiphyseal fracture | cHLGT |
| 17 | External fixation of fracture | cSMQ |
| 18 | Facial bones fracture | cHLGT |
| 19 | Femoral neck fracture | cSMQ+cHLGT |
| 20 | Femur fracture | cSMQ+cHLGT |
| 21 | Fibula fracture | cHLGT |
| 22 | Flail chest | cHLGT |
| 23 | Foot fracture | cHLGT |
| 24 | Forearm fracture | cSMQ+cHLGT |
| 25 | Fracture | cSMQ+cHLGT |
| 26 | Fracture displacement | cHLGT |
| 27 | Fracture of clavicle due to birth trauma | cHLGT |
| 28 | Fracture treatment | cSMQ |
| 29 | Fractured coccyx | cHLGT |
| 30 | Fractured ischium | cSMQ+cHLGT |
| 31 | Fractured sacrum | cSMQ+cHLGT |
| 32 | Fractured skull depressed | cHLGT |
| 33 | Greenstick fracture | cHLGT |
| 34 | Hand fracture | cHLGT |
| 35 | Hip fracture | cSMQ+cHLGT |
| 36 | Humerus fracture | cHLGT |

| | Selected Preferred Terms | Selection Type |
|----|-----------------------------------------------|----------------|
| 37 | Ilium fracture | cSMQ+cHLGT |
| 38 | Impacted fracture | cHLGT |
| 39 | Internal fixation of fracture | cSMQ |
| 40 | Jaw fracture | cHLGT |
| 41 | Limb fracture | cHLGT |
| 42 | Lower limb fracture | cHLGT |
| 43 | Lumbar vertebral fracture | cSMQ+cHLGT |
| 44 | Multiple fractures | cSMQ+cHLGT |
| 45 | Open fracture | cHLGT |
| 46 | Open reduction of fracture | cSMQ |
| 47 | Open reduction of spinal fracture | cSMQ |
| 48 | Osteochondral fracture | cHLGT |
| 49 | Osteoporotic fracture | cSMQ+cHLGT |
| 50 | Patella fracture | cHLGT |
| 51 | Pathological fracture | cSMQ+cHLGT |
| 52 | Pelvic fracture | cSMQ+cHLGT |
| 53 | Periprosthetic fracture | cHLGT |
| 54 | Pubis fracture | cSMQ+cHLGT |
| 55 | Radius fracture | cSMQ+cHLGT |
| 56 | Rib fracture | cSMQ+cHLGT |
| 57 | Sacroiliac fracture | cSMQ+cHLGT |
| 58 | Scapula fracture | cHLGT |
| 59 | Scapulothoracic dissociation | cHLGT |
| 60 | Skull fracture | cHLGT |
| 61 | Skull fractured base | cHLGT |
| 62 | Spinal compression fracture | cSMQ+cHLGT |
| 63 | Spinal fracture | cSMQ+cHLGT |
| 64 | Sternal fracture | cHLGT |
| 65 | Stress fracture | cHLGT |
| 66 | Tartrate-resistant acid phosphatase decreased | cSMQ |
| 67 | Thoracic vertebral fracture | cSMQ+cHLGT |
| 68 | Tibia fracture | cHLGT |
| 69 | Torus fracture | cHLGT |
| 70 | Traumatic fracture | cHLGT |
| 71 | Ulna fracture | cHLGT |
| 72 | Upper limb fracture | cHLGT |
| 73 | Vertebroplasty | cSMQ |
| 74 | Wrist fracture | cSMQ+cHLGT |
| 75 | Vertebral body replacement | cSMQ |

# **Appendix 3.** Bone Events

The selected PTs of bone events based on MedDRA 19.1 are listed as follows:

| | Selected Preferred Terms |
|----|--------------------------------------------------|
| 1 | Costal cartilage fracture |
| 2 | Chronic kidney disease-mineral and bone disorder |
| 3 | Astragalectomy |
| 4 | Gluteoplasty |
| 5 | Rotationplasty |
| 6 | Orthoroentgenogram |
| 7 | Atypical femur fracture |
| 8 | Carpal collapse |
| 9 | Osteonecrosis |
| 10 | Osteonecrosis of external auditory canal |
| 11 | Osteonecrosis of jaw |
| 12 | Osteoradionecrosis |
| 13 | Abscess jaw |
| 14 | Abscess oral |
| 15 | Alveolar osteitis |
| 16 | Arthrodesis |
| 17 | Biopsy bone abnormal |
| 18 | Bone abscess |
| 19 | Bone debridement |
| 20 | Bone graft |
| 21 | Bone infarction |
| 22 | Bone loss |
| 23 | Bone pain |
| 24 | Bone scan abnormal |
| 25 | Candida osteomyelitis |
| 26 | Chronic recurrent multifocal osteomyelitis |
| 27 | Dental necrosis |
| 28 | Exposed bone in jaw |
| 29 | Face and mouth X-ray abnormal |
| 30 | Groin pain |

| | Selected Preferred Terms |
|----|------------------------------|
| 31 | Hip arthroplasty |
| 32 | Hip surgery |
| 33 | Jaw lesion excision |
| 34 | Jaw operation |
| 35 | Joint arthroplasty |
| 36 | Joint prosthesis user |
| 37 | Joint resurfacing surgery |
| 38 | Maxillofacial operation |
| 39 | Oral surgery |
| 40 | Osteitis |
| 41 | Osteoarthropathy |
| 42 | Osteomyelitis |
| 43 | Osteomyelitis acute |
| 44 | Osteomyelitis bacterial |
| 45 | Osteomyelitis blastomyces |
| 46 | Osteomyelitis chronic |
| 47 | Osteomyelitis drainage |
| 48 | Osteomyelitis fungal |
| 49 | Osteomyelitis salmonella |
| 50 | Osteomyelitis viral |
| 51 | Osteotomy |
| 52 | Pain in jaw |
| 53 | Periodontal destruction |
| 54 | Primary sequestrum |
| 55 | Resorption bone increased |
| 56 | Secondary sequestrum |
| 57 | Sequestrectomy |
| 58 | Staphylococcal osteomyelitis |
| 59 | Subperiosteal abscess |
| 60 | Tertiary sequestrum |
| 61 | Tooth abscess |
| 62 | Tooth infection |
| 63 | X-ray limb abnormal |

| 64 X-ray of pelvis and hip abnormal 65 Bone density decreased 66 Bone formation decreased 67 Bone marrow oedema syndrome 68 Osteoporosis 69 Osteoporosis 70 Osteoporosis postmenopausal 71 Osteoporosis 72 Senile osteoporosis 73 Acetabulum fracture 74 Body height abnormal 75 Body height below normal 76 Body height decreased 77 Bone density abnormal 78 Bone formation test abnormal 79 Bone metabolism disorder 80 Bone resorption test abnormal 81 Cervical vertebral fracture 82 Closed fracture manipulation 83 C-telopeptide increased 84 Deoxypyridinoline urine increased 85 External fixation of fracture 86 Femur fracture 87 Femur fracture 88 Forearm fracture 89 Fracture testimen <th></th> <th>Selected Preferred Terms</th> | | Selected Preferred Terms |
|---|---|---|
| 66 Bone formation decreased 67 Bone marrow oedema syndrome 68 Osteopenia 69 Osteoporosis 70 Osteoporosis postmenopausal 71 Osteoporosis facture 72 Senile osteoporosis 73 Acetabulum fracture 74 Body height abnormal 75 Body height below normal 76 Body height decreased 77 Bone density abnormal 78 Bone formation test abnormal 79 Bone metabolism disorder 80 Bone resorption test abnormal 81 Cervical vertebral fracture 82 Closed fracture manipulation 83 C-telopeptide increased 84 Deoxypyridinoline urine increased 85 External fixation of fracture 86 Femoral neck fracture 87 Femoral neck fracture 88 Forearm fracture 89 Fracture treatment 91 Fractured ischium 92 Fractured sacrum <td>64</td> <td>X-ray of pelvis and hip abnormal</td> | 64 | X-ray of pelvis and hip abnormal |
| 67 Bone marrow oedema syndrome 68 Osteopenia 69 Osteoporosis 70 Osteoporosis postmenopausal 71 Osteoporosis 72 Senile osteoporosis 73 Acetabulum fracture 74 Body height abnormal 75 Body height below normal 76 Body height decreased 77 Bone density abnormal 78 Bone formation test abnormal 79 Bone metabolism disorder 80 Bone resorption test abnormal 81 Cervical vertebral fracture 82 Closed fracture manipulation 83 C-telopeptide increased 84 Deoxypyridinoline urine increased 85 External fixation of fracture 86 Femur fracture 87 Femur fracture 88 Forearm fracture 90 Fracture 90 Fracture treatment 91 Fracture dischium 91 Fracture 92 Fracture 94 Ilium fracture 95 Internal fixation of fracture | 65 | Bone density decreased |
| 68 Osteopenia 69 Osteoporosis 70 Osteoporosis postmenopausal 71 Osteoporosis postmenopausal 71 Osteoporosis 73 Acetabulum fracture 74 Body height abnormal 75 Body height below normal 76 Body height decreased 77 Bone density abnormal 78 Bone formation test abnormal 79 Bone metabolism disorder 80 Bone resorption test abnormal 81 Cervical vertebral fracture 82 Closed fracture manipulation 83 C-telopeptide increased 84 Deoxypyridinoline urine increased 85 External fixation of fracture 86 Femoral neck fracture 87 Femur fracture 88 Forearm fracture 89 Fracture 90 Fracture treatment 91 Fracture dischium 92 Fracture 93 Hip fracture 94 Ilium fracture 95 Internal fixation of fracture | 66 | Bone formation decreased |
| 69 Osteoporosis 70 Osteoporosis postmenopausal 71 Osteoporotic fracture 72 Senile osteoporosis 73 Acetabulum fracture 74 Body height abnormal 75 Body height below normal 76 Body height decreased 77 Bone density abnormal 78 Bone formation test abnormal 79 Bone metabolism disorder 80 Bone resorption test abnormal 81 Cervical vertebral fracture 82 Closed fracture manipulation 83 C-telopeptide increased 84 Deoxypyridinoline urine increased 85 External fixation of fracture 86 Femoral neck fracture 87 Femur fracture 88 Forearm fracture 89 Fracture treatment 90 Fracture treatment 91 Fractured ischium 92 Fractured sacrum 93 Hip fracture 94 Ilium fracture 95 Internal fixation of fracture | 67 | Bone marrow oedema syndrome |
| Osteoporosis postmenopausal Osteoporotic fracture Senile osteoporosis Accetabulum fracture Body height abnormal Body height below normal Body height decreased Body height decreased Bone density abnormal Bone density abnormal Bone metabolism disorder Bone metabolism disorder Bone metabolism disorder Bone presorption test abnormal Cervical vertebral fracture Closed fracture manipulation C-telopeptide increased Bone prospridinoline urine increased External fixation of fracture Femoral neck fracture Femoral neck fracture Ferneur fracture Fracture treatment Fracture treatment Fracture dischium Fracture Fracture dischium Fracture Firacture firacture Firacture Firacture F | 68 | Osteopenia |
| 71 Osteoporotic fracture 72 Senile osteoporosis 73 Acetabulum fracture 74 Body height abnormal 75 Body height below normal 76 Body height decreased 77 Bone density abnormal 78 Bone formation test abnormal 79 Bone metabolism disorder 80 Bone resorption test abnormal 81 Cervical vertebral fracture 82 Closed fracture manipulation 83 C-telopeptide increased 84 Deoxypyridinoline urine increased 85 External fixation of fracture 86 Femoral neck fracture 87 Femur fracture 88 Forearm fracture 89 Fracture 90 Fracture treatment 91 Fracture dischium 92 Fractured sacrum 93 Hip fracture 94 Ilium fracture 95 Internal fixation of fracture | 69 | Osteoporosis |
| Senile osteoporosis Acetabulum fracture Body height abnormal Body height abnormal Body height below normal Body height decreased Body height decreased Bone density abnormal Bone formation test abnormal Bone metabolism disorder Bone metabolism disorder Bone resorption test abnormal Cervical vertebral fracture Closed fracture manipulation C-telopeptide increased Bone peoxypyridinoline urine increased External fixation of fracture Femoral neck fracture Femoral neck fracture Fracture dischium Fracture Hip fracture | 70 | Osteoporosis postmenopausal |
| Acctabulum fracture Body height abnormal Body height below normal Body height below normal Body height decreased Bone density abnormal Bone density abnormal Bone formation test abnormal Bone metabolism disorder Bone metabolism disorder Bone resorption test abnormal Cervical vertebral fracture Closed fracture manipulation C-telopeptide increased Bone resorption in creased External fixation of fracture Femoral neck fracture Femoral neck fracture Fracture treatment Fracture dischium Fracture Fracture dischium Fracture Hip fracture Hip fracture Ilium fracture Internal fixation of fracture | 71 | Osteoporotic fracture |
| Body height abnormal Body height below normal Body height below normal Body height decreased Body height decreased Bone density abnormal Bone density abnormal Bone formation test abnormal Bone metabolism disorder Bone metabolism disorder Bone resorption test abnormal Cervical vertebral fracture Closed fracture manipulation C-telopeptide increased Bone resorption test abnormal External fixation of fracture Femoral neck fracture Femoral neck fracture Femoral neck fracture Fracture Firacture Fracture Fracture Firacture Fracture treatment Fracture dischium Fracture Firacture firacture Firacture firacture | 72 | Senile osteoporosis |
| Body height below normal Body height decreased Body height decreased Bone density abnormal Bone density abnormal Bone formation test abnormal Bone metabolism disorder Bone resorption test abnormal Cervical vertebral fracture Closed fracture manipulation C-telopeptide increased Bone resorption test abnormal Cervical vertebral fracture Example Colosed fracture manipulation Bone resorption test abnormal Cervical vertebral fracture Example Colosed fracture manipulation Bone resorption test abnormal Cervical vertebral fracture Example Colosed fracture manipulation External fixation of fracture Femoral neck fracture Femoral neck fracture Femoral neck fracture Femoral recture Forearm fracture Forearm fracture Fracture Fracture Fracture Fracture Fracture treatment Fracture dischium Fractured sacrum Hip fracture Hip fracture Ilium fracture Ilium fracture | 73 | Acetabulum fracture |
| Body height decreased Bone density abnormal Bone density abnormal Bone formation test abnormal Bone metabolism disorder Bone metabolism disorder Bone resorption test abnormal Cervical vertebral fracture Closed fracture manipulation C-telopeptide increased Bone resorption test abnormal Cervical vertebral fracture Closed fracture manipulation Bone resorption test abnormal Cervical vertebral fracture Closed fracture manipulation Bone resorption test abnormal Cervical vertebral fracture Bone resorption test abnormal Cervical vertebral fracture Fermanipulation Fermani fracture Fermani fracture Fermani fracture Fermani fracture Forearm fracture Forearm fracture Forearm fracture Fracture Fracture Fracture Fracture Fracture sacrum Firacture Jilium fracture Finternal fixation of fracture | 74 | Body height abnormal |
| Bone density abnormal Bone formation test abnormal Bone metabolism disorder Bone metabolism disorder Bone resorption test abnormal Cervical vertebral fracture Closed fracture manipulation C-telopeptide increased Bone resorption test abnormal Cervical vertebral fracture Closed fracture manipulation C-telopeptide increased External fixation of fracture Femoral neck fracture Femoral neck fracture Forearm fracture Forearm fracture Forearm fracture Fracture Fracture Fracture Fracture Fracture Fracture Ilium fracture Ilium fracture Internal fixation of fracture | 75 | Body height below normal |
| Bone formation test abnormal Bone metabolism disorder Bone resorption test abnormal Cervical vertebral fracture Closed fracture manipulation C-telopeptide increased Deoxypyridinoline urine increased External fixation of fracture Femur fracture Femur fracture Forearm fracture Fracture Fracture Fracture Fracture Fracture Fracture treatment Fracture dischium Fracture Fracture dischium Firacture dischium Firacture Firacture Firacture Firacture firacture | 76 | Body height decreased |
| Bone metabolism disorder Bone resorption test abnormal Cervical vertebral fracture Closed fracture manipulation C-telopeptide increased Deoxypyridinoline urine increased External fixation of fracture Femoral neck fracture Femoral neck fracture Forearm fracture Fracture Firacture Fracture Firacture dischium Firacture fixation Firacture Firactu | 77 | Bone density abnormal |
| Bone resorption test abnormal Cervical vertebral fracture Closed fracture manipulation C-telopeptide increased External fixation of fracture External fixation of fracture External fracture Ext | 78 | Bone formation test abnormal |
| Cervical vertebral fracture Closed fracture manipulation C-telopeptide increased C-telopeptide increased External fixation of fracture External fixation of fracture Femoral neck fracture Femur fracture Forearm fracture Fracture Fracture Fracture Fracture treatment Fracture dischium Fractured sacrum Hip fracture Ilium fracture Internal fixation of fracture | 79 | Bone metabolism disorder |
| Closed fracture manipulation C-telopeptide increased Deoxypyridinoline urine increased External fixation of fracture External fixation of fracture Femoral neck fracture Femur fracture Femur fracture Fracture Fracture Fracture Fracture Fracture treatment Fractured ischium Fractured sacrum Hip fracture Ilium fracture Internal fixation of fracture | 80 | Bone resorption test abnormal |
| C-telopeptide increased B4 Deoxypyridinoline urine increased B5 External fixation of fracture B6 Femoral neck fracture B7 Femur fracture B8 Forearm fracture B9 Fracture 90 Fracture treatment 91 Fractured ischium 92 Fractured sacrum 93 Hip fracture 94 Ilium fracture 95 Internal fixation of fracture | 81 | Cervical vertebral fracture |
| B4 Deoxypyridinoline urine increased B5 External fixation of fracture B6 Femoral neck fracture B7 Femur fracture B8 Forearm fracture B9 Fracture 90 Fracture treatment 91 Fractured ischium 92 Fractured sacrum 93 Hip fracture 94 Illium fracture 95 Internal fixation of fracture | 82 | Closed fracture manipulation |
| External fixation of fracture Femoral neck fracture Femur fracture Femur fracture Forearm fracture Fracture Fracture Fracture treatment Fractured ischium Fractured sacrum Hip fracture Ilium fracture Internal fixation of fracture | 83 | C-telopeptide increased |
| Femoral neck fracture Femur fracture Femur fracture Forearm fracture Fracture Fracture Fracture treatment Fractured ischium Fractured sacrum Hip fracture Ilium fracture Internal fixation of fracture | 84 | Deoxypyridinoline urine increased |
| Femur fracture Forearm fracture Fracture Fracture Fracture treatment Fracture dischium Fractured sacrum Hip fracture Ilium fracture Internal fixation of fracture | 85 | External fixation of fracture |
| Forearm fracture Fracture Fracture Fracture treatment Fractured ischium Fractured sacrum Hip fracture Ilium fracture Internal fixation of fracture | 86 | Femoral neck fracture |
| Fracture Fracture treatment Fracture dischium Fractured sacrum Fractured sacrum Hip fracture Ilium fracture Internal fixation of fracture | 87 | Femur fracture |
| Fracture treatment Fractured ischium Fractured sacrum Hip fracture Ilium fracture Internal fixation of fracture | 88 | Forearm fracture |
| 91 Fractured ischium 92 Fractured sacrum 93 Hip fracture 94 Ilium fracture 95 Internal fixation of fracture | 89 | Fracture |
| 92 Fractured sacrum 93 Hip fracture 94 Ilium fracture 95 Internal fixation of fracture | 90 | Fracture treatment |
| 93 Hip fracture 94 Ilium fracture 95 Internal fixation of fracture | 91 | Fractured ischium |
| 94 Ilium fracture 95 Internal fixation of fracture | 92 | Fractured sacrum |
| 95 Internal fixation of fracture | 93 | Hip fracture |
| | 94 | Ilium fracture |
| 96 Kyphoscoliosis | 95 | Internal fixation of fracture |
| | 96 | Kyphoscoliosis |

| | Selected Preferred Terms |
|-----|-----------------------------------------------|
| 97 | Kyphosis |
| 98 | Lumbar vertebral fracture |
| 99 | Multiple fractures |
| 100 | N-telopeptide urine increased |
| 101 | Open reduction of fracture |
| 102 | Open reduction of spinal fracture |
| 103 | Osteocalcin increased |
| 104 | Osteoporosis prophylaxis |
| 105 | Pathological fracture |
| 106 | Pelvic fracture |
| 107 | Post-traumatic osteoporosis |
| 108 | Pubis fracture |
| 109 | Pyridinoline urine increased |
| 110 | Radius fracture |
| 111 | Rib fracture |
| 112 | Sacroiliac fracture |
| 113 | Spinal compression fracture |
| 114 | Spinal deformity |
| 115 | Spinal fracture |
| 116 | Tartrate-resistant acid phosphatase decreased |
| 117 | Thoracic vertebral fracture |
| 118 | Vertebral body replacement |
| 119 | Vertebroplasty |
| 120 | Wrist fracture |
| 121 | Wrist surgery |
| 122 | Ankle fracture |
| 123 | Atypical fracture |
| 124 | Avulsion fracture |
| 125 | Bone fissure |
| 126 | Bone fragmentation |
| 127 | Chance fracture |
| 128 | Clavicle fracture |
| 129 | Comminuted fracture |
| J | |

| | Selected Preferred Terms |
|----------|------------------------------------------|
| 130 | Complicated fracture |
| 131 | Compression fracture |
| 132 | Craniofacial fracture |
| 133 | Epiphyseal fracture |
| 134 | Facial bones fracture |
| 135 | Fibula fracture |
| 136 | Flail chest |
| 137 | Foot fracture |
| 138 | Fracture delayed union |
| 139 | Fracture displacement |
| 140 | Fracture malunion |
| 141 | Fracture nonunion |
| 142 | Fracture of clavicle due to birth trauma |
| 143 | Fractured coccyx |
| 144 | Fractured skull depressed |
| 145 | Greenstick fracture |
| 146 | Hand fracture |
| 147 | Humerus fracture |
| 148 | Impacted fracture |
| 149 | Jaw fracture |
| 150 | Limb fracture |
| 151 | Lower limb fracture |
| 152 | Open fracture |
| 153 | Osteochondral fracture |
| 154 | Patella fracture |
| 155 | Periprosthetic fracture |
| 156 | Pseudarthrosis |
| 157 | Scapula fracture |
| 158 | Scapulothoracic dissociation |
| 159 | Skull fracture |
| 160 | Skull fractured base |
| 161 | Spinal fusion fracture |
| 162 | Sternal fracture |
| <u> </u> | |
| | Selected Preferred Terms |
|-----|-------------------------------------|
| 163 | Stress fracture |
| 164 | Tibia fracture |
| 165 | Torus fracture |
| 166 | Traumatic fracture |
| 167 | Ulna fracture |
| 168 | Upper limb fracture |
| 169 | Bone formation test |
| 170 | Bone resorption test |
| 171 | C-telopeptide |
| 172 | Deoxypyridinoline urine |
| 173 | N-telopeptide |
| 174 | N-telopeptide urine |
| 175 | N-telopeptide urine abnormal |
| 176 | N-telopeptide urine decreased |
| 177 | N-telopeptide urine normal |
| 178 | Osteocalcin |
| 179 | Osteocalcin decreased |
| 180 | Osteoprotegerin |
| 181 | Osteoprotegerin decreased |
| 182 | Osteoprotegerin increased |
| 183 | Osteoprotegerin ligand |
| 184 | Osteoprotegerin ligand decreased |
| 185 | Pyridinoline urine |
| 186 | Pyridinoline urine decreased |
| 187 | Tartrate-resistant acid phosphatase |
| 188 | Aneurysmal bone cyst |
| 189 | Bone callus excessive |
| 190 | Bone contusion |
| 191 | Bone cyst |
| 192 | Bone development abnormal |
| 193 | Bone disorder |
| 194 | Bone erosion |
| 195 | Bone fistula |

| | Selected Preferred Terms |
|-----|--------------------------------------|
| 196 | Bone formation increased |
| 197 | Bone hyperpigmentation |
| 198 | Bone lesion |
| 199 | Callus formation delayed |
| 200 | Cemento osseous dysplasia |
| 201 | Dental alveolar anomaly |
| 202 | Dental cyst |
| 203 | Enostosis |
| 204 | Erdheim-Chester disease |
| 205 | Exostosis |
| 206 | Exostosis of external ear canal |
| 207 | Exostosis of jaw |
| 208 | Extraskeletal ossification |
| 209 | Hyperphosphatasaemia |
| 210 | Hypertrophic osteoarthropathy |
| 211 | Inadequate osteointegration |
| 212 | Jaw cyst |
| 213 | Jaw disorder |
| 214 | Medial tibial stress syndrome |
| 215 | Melorheostosis |
| 216 | Osteitis condensans |
| 217 | Osteitis deformans |
| 218 | Osteorrhagia |
| 219 | Osteosclerosis |
| 220 | Osteosis |
| 221 | Periosteal haematoma |
| 222 | Periostitis |
| 223 | Periostitis hypertrophic |
| 224 | Periostosis |
| 225 | Periprosthetic osteolysis |
| 226 | Post transplant distal limb syndrome |
| 227 | Radiation osteitis |
| 228 | Skeletal injury |

| | Selected Preferred Terms |
|-----|--------------------------------------|
| 229 | Spinal column injury |
| 230 | Spinal disorder |
| 231 | Sternal injury |
| 232 | Vertebral column mass |
| 233 | Vertebral lesion |
| 234 | Vertebral wedging |
| 235 | Bone atrophy |
| 236 | Bone decalcification |
| 237 | Brown tumour |
| 238 | Craniotabes |
| 239 | Gorham's disease |
| 240 | Hereditary hypophosphataemic rickets |
| 241 | High turnover osteopathy |
| 242 | Hungry bone syndrome |
| 243 | Hypochondroplasia |
| 244 | Hypophosphataemic rickets |
| 245 | Low turnover osteopathy |
| 246 | Oncogenic osteomalacia |
| 247 | Osteolysis |
| 248 | Osteomalacia |
| 249 | Osteoporosis circumscripta cranii |
| 250 | Rachitic rosary |
| 251 | Resorption bone decreased |
| 252 | Rickets |
| 253 | Bone marrow oedema |
| 254 | Bone swelling |
| 255 | Coccydynia |
| 256 | Eagle's syndrome |
| 257 | Metatarsalgia |
| 258 | Os trigonum syndrome |
| 259 | Pubic pain |
| 260 | Spinal pain |
| 261 | Bone cyst excision |

| | Selected Preferred Terms |
|-----|---------------------------------------|
| 262 | Bone electrostimulation therapy |
| 263 | Bone graft removal |
| 264 | Bone lesion excision |
| 265 | Bone operation |
| 266 | Bone prosthesis insertion |
| 267 | Bone trimming |
| 268 | Cementoplasty |
| 269 | Epiphyseal surgery |
| 270 | Epiphysiodesis |
| 271 | Orthopaedic procedure |
| 272 | Ostectomy |
| 273 | Osteopathic treatment |
| 274 | Osteosynthesis |
| 275 | Removal of epiphyseal fixation |
| 276 | Removal of internal fixation |
| 277 | Calcification metastatic |
| 278 | Calciphylaxis |
| 279 | Calcium deficiency |
| 280 | Calcium intoxication |
| 281 | Calcium metabolism disorder |
| 282 | Chondrocalcinosis pyrophosphate |
| 283 | Chvostek's sign |
| 284 | Dent's disease |
| 285 | Familial hypocalciuric hypercalcaemia |
| 286 | Hypercalcaemia |
| 287 | Hypercalcaemia of malignancy |
| 288 | Hypercalcaemic nephropathy |
| 289 | Hypercalcitoninaemia |
| 290 | Hypercalciuria |
| 291 | Hypocalcaemia |
| 292 | Hypocalcaemic seizure |
| 293 | Hypocalciuria |
| 294 | Hypoparathyroidism |

| | Selected Preferred Terms |
|-----|---------------------------------------|
| 295 | Hypoparathyroidism secondary |
| 296 | Latent tetany |
| 297 | Periarthritis calcarea |
| 298 | Primary hypoparathyroidism |
| 299 | Pseudohypercalcaemia |
| 300 | Pseudohypoparathyroidism |
| 301 | Tetany |
| 302 | Tooth demineralisation |
| 303 | Trousseau's sign |
| 304 | Williams syndrome |
| 305 | Congenital syphilitic osteochondritis |
| 306 | Epiphyseal disorder |
| 307 | Epiphyseal injury |
| 308 | Epiphyses delayed fusion |
| 309 | Epiphyses premature fusion |
| 310 | Epiphysiolysis |
| 311 | Epiphysitis |
| 312 | Fracture debridement |
| 313 | Fracture reduction |
| 314 | Fractured maxilla elevation |
| 315 | Fractured zygomatic arch elevation |
| 316 | Intramedullary rod insertion |
| 317 | Skeletal traction |
| 318 | Surgical fixation of rib fracture |
| 319 | Radial head dislocation |
| 320 | Amputation |
| 321 | Arm amputation |
| 322 | Calcanectomy |
| 323 | Finger amputation |
| 324 | Finger repair operation |
| 325 | Foot amputation |
| 326 | Foot operation |
| 327 | Hand amputation |

| 328 | Hand repair operation |
|-----|---------------------------------|
| 329 | Hip disarticulation |
| 330 | Interscapulothoracic amputation |
| 331 | Leg amputation |
| 332 | Limb amputation |
| 333 | Limb immobilisation |
| 334 | Limb operation |
| 335 | Limb reattachment surgery |
| 336 | Limb reconstructive surgery |
| 337 | Metacarpal excision |
| 338 | Metatarsal excision |
| 339 | Microsurgery to hand |
| 340 | Talipes correction |
| 341 | Toe amputation |
| 342 | Toe operation |
| 343 | Trapezectomy |
| 344 | Alveolar bone resorption |
| 345 | Dwarfism |
| 346 | Osteodystrophy |
| 347 | Renal rickets |
| 348 | Aspiration bursa |
| 349 | Aspiration bursa abnormal |
| 350 | Aspiration bursa normal |
| 351 | Aspiration joint |
| 352 | Aspiration joint abnormal |
| 353 | Aspiration joint normal |
| 354 | Biopsy abdominal wall |
| 355 | Biopsy abdominal wall abnormal |
| 356 | Biopsy abdominal wall normal |
| 357 | Biopsy bone |
| 358 | Biopsy bone normal |
| 359 | Biopsy cartilage |
| 360 | Biopsy cartilage abnormal |

| 361 Biopsy chest wall 362 Biopsy chest wall abnormal 363 Biopsy chest wall abnormal 364 Biopsy ligament 365 Biopsy ligament abnormal 366 Biopsy ligament normal 367 Biopsy ligament normal 368 Biopsy muscle 369 Biopsy muscle abnormal 370 Biopsy muscle normal 371 Biopsy tendon 372 Biopsy tendon 373 Biopsy tendon abnormal 374 Biopsy tendon normal 375 Intervertebral disc biopsy 376 Synovial biopsy abnormal 378 Synovial biopsy abnormal 379 Synovial fluid crystal 380 Synovial fluid crystal 381 Synovial fluid red blood cells 382 Synovial fluid red blood cells 383 Synovial fluid white blood cells 384 Synovial fluid white blood cells positive 385 Arthrogram normal 386 Arthrogram normal 387 | | Selected Preferred Terms |
|---|---|---|
| 363 Biopsy chest wall normal 364 Biopsy ligament 365 Biopsy ligament abnormal 366 Biopsy ligament normal 367 Biopsy ligament normal 368 Biopsy muscle 369 Biopsy muscle abnormal 370 Biopsy muscle normal 371 Biopsy soft tissue 372 Biopsy tendon 373 Biopsy tendon abnormal 374 Biopsy tendon normal 375 Intervertebral disc biopsy 376 Synovial biopsy abnormal 377 Synovial fluid cell count 378 Synovial fluid crystal 380 Synovial fluid crystal present 381 Synovial fluid red blood cells 382 Synovial fluid white blood cells 383 Synovial fluid white blood cells 384 Synovial fluid white blood cells 385 Arthrogram 386 Arthrogram normal 387 Arthogram abnormal 388 Arthrogram normal 389 Ar | 361 | Biopsy cartilage normal |
| 364 Biopsy ligament 365 Biopsy ligament 366 Biopsy ligament abnormal 367 Biopsy ligament normal 368 Biopsy muscle 369 Biopsy muscle abnormal 370 Biopsy muscle normal 371 Biopsy tendon 372 Biopsy tendon 373 Biopsy tendon normal 374 Biopsy tendon normal 375 Intervertebral disc biopsy 376 Synovial biopsy 377 Synovial biopsy abnormal 378 Synovial fluid cell count 379 Synovial fluid crystal 380 Synovial fluid crystal present 381 Synovial fluid red blood cells 382 Synovial fluid dred blood cells positive 383 Synovial fluid white blood cells positive 384 Synovial fluid white blood cells positive 385 Arthrogram 386 Arthrogram abnormal 387 Arthrogram normal 388 Arthroscopy 389 Arth | 362 | Biopsy chest wall |
| 365 Biopsy ligament 366 Biopsy ligament abnormal 367 Biopsy ligament normal 368 Biopsy muscle 369 Biopsy muscle abnormal 370 Biopsy muscle normal 371 Biopsy soft tissue 372 Biopsy tendon 373 Biopsy tendon abnormal 374 Biopsy tendon normal 375 Intervertebral disc biopsy 376 Synovial biopsy 377 Synovial biopsy abnormal 378 Synovial fluid cell count 379 Synovial fluid crystal 380 Synovial fluid crystal present 381 Synovial fluid red blood cells 382 Synovial fluid red blood cells positive 383 Synovial fluid white blood cells positive 384 Synovial fluid white blood cells positive 385 Arthrogram 386 Arthrogram abnormal 387 Arthrogram abnormal 388 Arthrogram pormal 389 Arthroscopy abnormal 390 <td>363</td> <td>Biopsy chest wall abnormal</td> | 363 | Biopsy chest wall abnormal |
| 366 Biopsy ligament abnormal 367 Biopsy ligament normal 368 Biopsy muscle 369 Biopsy muscle abnormal 370 Biopsy soft tissue 371 Biopsy tendon 372 Biopsy tendon 373 Biopsy tendon abnormal 374 Biopsy tendon normal 375 Intervertebral disc biopsy 376 Synovial biopsy 377 Synovial biopsy abnormal 378 Synovial fluid cell count 379 Synovial fluid crystal 380 Synovial fluid red blood cells 381 Synovial fluid red blood cells 382 Synovial fluid white blood cells positive 383 Synovial fluid white blood cells positive 384 Synovial fluid white blood cells positive 385 Arthrogram 386 Arthrogram normal 387 Arthrogram normal 388 Arthroscopy 389 Arthroscopy abnormal 390 Arthroscopy normal 391 < | 364 | Biopsy chest wall normal |
| 367 Biopsy ligament normal 368 Biopsy muscle 369 Biopsy muscle abnormal 370 Biopsy muscle normal 371 Biopsy send tissue 372 Biopsy tendon 373 Biopsy tendon abnormal 374 Biopsy tendon normal 375 Intervertebral disc biopsy 376 Synovial biopsy 377 Synovial biopsy abnormal 378 Synovial fluid cell count 379 Synovial fluid crystal 380 Synovial fluid red blood cells 381 Synovial fluid red blood cells 382 Synovial fluid white blood cells positive 383 Synovial fluid white blood cells positive 384 Synovial fluid white blood cells positive 385 Arthrogram 386 Arthrogram normal 387 Arthrogram normal 388 Arthroscopy 389 Arthroscopy abnormal 390 Arthroscopy abnormal 391 Bone density increased | 365 | Biopsy ligament |
| 368 Biopsy muscle 369 Biopsy muscle abnormal 370 Biopsy muscle normal 371 Biopsy soft tissue 372 Biopsy tendon 373 Biopsy tendon abnormal 374 Biopsy tendon normal 375 Intervertebral disc biopsy 376 Synovial biopsy 377 Synovial biopsy abnormal 378 Synovial fluid cell count 379 Synovial fluid crystal present 381 Synovial fluid red blood cells 382 Synovial fluid red blood cells positive 383 Synovial fluid white blood cells 384 Synovial fluid white blood cells positive 385 Arthrogram 386 Arthrogram abnormal 387 Arthrogram normal 388 Arthroscopy 389 Arthroscopy abnormal 390 Arthroscopy normal 391 Bone densitometry 392 Bone density increased | 366 | Biopsy ligament abnormal |
| 369 Biopsy muscle abnormal 370 Biopsy muscle normal 371 Biopsy soft tissue 372 Biopsy tendon 373 Biopsy tendon abnormal 374 Biopsy tendon normal 375 Intervertebral disc biopsy 376 Synovial biopsy 377 Synovial biopsy abnormal 378 Synovial fluid cell count 379 Synovial fluid crystal 380 Synovial fluid crystal present 381 Synovial fluid red blood cells 382 Synovial fluid red blood cells positive 383 Synovial fluid white blood cells 384 Synovial fluid white blood cells positive 385 Arthrogram 386 Arthrogram abnormal 387 Arthrogram normal 388 Arthroscopy 389 Arthroscopy abnormal 390 Arthroscopy normal 391 Bone densitometry 392 Bone density increased | 367 | Biopsy ligament normal |
| Biopsy muscle normal | 368 | Biopsy muscle |
| Biopsy soft tissue Biopsy tendon Biopsy tendon abnormal Biopsy tendon abnormal Biopsy tendon normal Bynovial biopsy Bynovial biopsy Bynovial fluid cell count Bynovial fluid crystal Biopsy tendon normal Biopsy tendon normal Bynovial fluid cystal present Bynovial fluid crystal present Bynovial fluid red blood cells Bynovial fluid red blood cells positive Bynovial fluid white blood cells | 369 | Biopsy muscle abnormal |
| Biopsy tendon Biopsy tendon abnormal Biopsy tendon normal Biopsy tendon abnormal Biopsy tendon normal Biopsy tendon abnormal Biopsy tendon normal Biopsy tendon abnormal Biopsy tendon normal Biopsy tendon abnormal Biopsy tendon normal Biopsy tendon normal Biopsy tendon abnormal Biopsy tendon abno | 370 | Biopsy muscle normal |
| Biopsy tendon abnormal Biopsy tendon normal Biopsy | 371 | Biopsy soft tissue |
| Biopsy tendon normal Biopsy abnormal Biopsy abnormal Biopsy abnormal Biopsy tendon normal Biopsy abnormal Biopsy tendon normal Biopsy abnormal Biopsy abn | 372 | Biopsy tendon |
| 375 Intervertebral disc biopsy 376 Synovial biopsy 377 Synovial biopsy abnormal 378 Synovial fluid cell count 379 Synovial fluid crystal 380 Synovial fluid crystal present 381 Synovial fluid red blood cells 382 Synovial fluid red blood cells 383 Synovial fluid white blood cells 384 Synovial fluid white blood cells 385 Arthrogram 386 Arthrogram normal 387 Arthrogram normal 388 Arthroscopy 389 Arthroscopy abnormal 390 Arthroscopy normal 391 Bone density increased | 373 | Biopsy tendon abnormal |
| Synovial biopsy Synovial biopsy abnormal Synovial fluid cell count Synovial fluid crystal Synovial fluid crystal Synovial fluid crystal present Synovial fluid red blood cells Synovial fluid red blood cells Synovial fluid white blood cells Synovial fluid white blood cells Synovial fluid white blood cells Arthrogram Arthrogram Arthrogram abnormal Arthrogram normal Arthroscopy Arthroscopy Synovial fluid white blood cells positive Synovial fluid white blood cells positive Arthrogram abnormal Bone densitometry Synovial fluid white blood cells positive | 374 | Biopsy tendon normal |
| 377Synovial biopsy abnormal378Synovial fluid cell count379Synovial fluid crystal380Synovial fluid crystal present381Synovial fluid red blood cells382Synovial fluid red blood cells positive383Synovial fluid white blood cells384Synovial fluid white blood cells positive385Arthrogram386Arthrogram abnormal387Arthrogram normal388Arthroscopy389Arthroscopy abnormal390Arthroscopy normal391Bone densitometry392Bone density increased | 375 | Intervertebral disc biopsy |
| Synovial fluid cell count Synovial fluid crystal Synovial fluid crystal present Synovial fluid red blood cells Synovial fluid red blood cells Synovial fluid red blood cells positive Synovial fluid white blood cells Synovial fluid white blood cells Synovial fluid white blood cells Arthrogram Arthrogram Arthrogram abnormal Arthrogram normal Arthroscopy Arthroscopy Synovial fluid white blood cells positive Synovial fluid white blood cells positive Arthrogram Synovial fluid white blood cells positive Arthrogram Synovial fluid white blood cells positive Arthrogram Synovial fluid red blood cells | 376 | Synovial biopsy |
| 379Synovial fluid crystal380Synovial fluid crystal present381Synovial fluid red blood cells382Synovial fluid red blood cells positive383Synovial fluid white blood cells384Synovial fluid white blood cells positive385Arthrogram386Arthrogram abnormal387Arthrogram normal388Arthroscopy389Arthroscopy abnormal390Arthroscopy normal391Bone densitometry392Bone density increased | 377 | Synovial biopsy abnormal |
| 380Synovial fluid crystal present381Synovial fluid red blood cells382Synovial fluid red blood cells positive383Synovial fluid white blood cells384Synovial fluid white blood cells positive385Arthrogram386Arthrogram abnormal387Arthrogram normal388Arthroscopy389Arthroscopy abnormal390Arthroscopy normal391Bone densitometry392Bone density increased | 378 | Synovial fluid cell count |
| Synovial fluid red blood cells Synovial fluid red blood cells positive Synovial fluid white blood cells Synovial fluid white blood cells Synovial fluid white blood cells positive Arthrogram Arthrogram abnormal Arthrogram normal Arthroscopy Arthroscopy Arthroscopy abnormal Arthroscopy normal Bone density increased | 379 | Synovial fluid crystal |
| Synovial fluid red blood cells positive Synovial fluid white blood cells Synovial fluid white blood cells positive Arthrogram Arthrogram abnormal Arthrogram normal Arthroscopy Arthroscopy Arthroscopy abnormal Arthroscopy normal Bone densitometry Bone density increased | 380 | Synovial fluid crystal present |
| Synovial fluid white blood cells Synovial fluid white blood cells positive Arthrogram Arthrogram abnormal Arthrogram normal Arthroscopy Arthroscopy Arthroscopy abnormal Arthroscopy normal Bone densitometry Bone density increased | 381 | Synovial fluid red blood cells |
| Synovial fluid white blood cells positive Arthrogram Arthrogram abnormal Arthrogram normal Arthroscopy Arthroscopy abnormal Arthroscopy normal Bone densitometry Bone density increased | 382 | Synovial fluid red blood cells positive |
| Arthrogram Arthrogram abnormal Arthrogram normal Arthroscopy Arthroscopy abnormal Arthroscopy normal Bone densitometry Bone density increased | 383 | Synovial fluid white blood cells |
| 386 Arthrogram abnormal 387 Arthrogram normal 388 Arthroscopy 389 Arthroscopy abnormal 390 Arthroscopy normal 391 Bone densitometry 392 Bone density increased | 384 | Synovial fluid white blood cells positive |
| Arthrogram normal Arthroscopy Arthroscopy abnormal Arthroscopy normal Bone densitometry Bone density increased | 385 | Arthrogram |
| Arthroscopy 389 Arthroscopy abnormal 390 Arthroscopy normal 391 Bone densitometry 392 Bone density increased | 386 | Arthrogram abnormal |
| Arthroscopy abnormal Arthroscopy normal Bone densitometry Bone density increased | 387 | Arthrogram normal |
| 390 Arthroscopy normal 391 Bone densitometry 392 Bone density increased | 388 | Arthroscopy |
| 391 Bone density increased Bone density increased | 389 | Arthroscopy abnormal |
| Bone density increased | 390 | Arthroscopy normal |
| | 391 | Bone densitometry |
| 393 Bone scan | 392 | Bone density increased |
| | 393 | Bone scan |

| | Selected Preferred Terms |
|-----|--------------------------------|
| 394 | Bone scan normal |
| 395 | Discogram |
| 396 | Discogram abnormal |
| 397 | Discogram normal |
| 398 | Face and mouth X-ray |
| 399 | Face and mouth X-ray normal |
| 400 | Skeletal survey |
| 401 | Skeletal survey abnormal |
| 402 | Skeletal survey normal |
| 403 | Skull X-ray |
| 404 | Skull X-ray abnormal |
| 405 | Skull X-ray normal |
| 406 | Spinal X-ray |
| 407 | Spinal X-ray abnormal |
| 408 | Spinal X-ray normal |
| 409 | Ultrasound joint |
| 410 | X-ray limb |
| 411 | X-ray limb normal |
| 412 | X-ray of pelvis and hip |
| 413 | X-ray of pelvis and hip normal |
| 414 | Acute phosphate nephropathy |
| 415 | Hyperphosphataemia |
| 416 | Hyperphosphaturia |
| 417 | Hypophosphataemia |
| 418 | Phosphorus metabolism disorder |
| 419 | Pseudohyperphosphataemia |
| 420 | Dislocation of vertebra |
| 421 | Intervertebral disc injury |
| 422 | Ankle arthroplasty |
| 423 | Ankle operation |
| 424 | Arthrectomy |
| 425 | Arthrolysis |
| 426 | Arthroscopic surgery |

| | Selected Preferred Terms |
|-----|------------------------------------|
| 427 | Arthrotomy |
| 428 | Baker's cyst excision |
| 429 | Bone groove deepening |
| 430 | Bunion operation |
| 431 | Capsulorrhaphy |
| 432 | Delayed spinal fusion |
| 433 | Elbow operation |
| 434 | Incomplete spinal fusion |
| 435 | Knee arthroplasty |
| 436 | Knee operation |
| 437 | Ligament operation |
| 438 | Maxillonasal dysplasia |
| 439 | Meniscus operation |
| 440 | Meniscus removal |
| 441 | Patella replacement |
| 442 | Patellectomy |
| 443 | Radiolucency around implant |
| 444 | Radiotherapy to joint |
| 445 | Removal of foreign body from joint |
| 446 | Rheumatoid nodule removal |
| 447 | Rotator cuff repair |
| 448 | Shoulder arthroplasty |
| 449 | Shoulder operation |
| 450 | Synovectomy |
| 451 | Synoviorthesis |
| 452 | Temporomandibular joint surgery |
| 453 | Tophus removal operation |

## **Appendix 4.** Potential Uveitis

The selected PTs of potential uveitis from SOC of Eye Disorders are listed as follows:

| | Selected Preferred Terms |
|----|--------------------------------------|
| 1 | Homonymous diplopia |
| 2 | Keratic precipitates |
| 3 | Retinal thickening |
| 4 | Vitreous haze |
| 5 | Acute zonal occult outer retinopathy |
| 6 | Anterior chamber cell |
| 7 | Anterior chamber fibrin |
| 8 | Anterior chamber flare |
| 9 | Anterior chamber inflammation |
| 10 | Aqueous fibrin |
| 11 | Autoimmune retinopathy |
| 12 | Autoimmune uveitis |
| 13 | Behcet's syndrome |
| 14 | Birdshot chorioretinopathy |
| 15 | Blau syndrome |
| 16 | Blindness |
| 17 | Blindness transient |
| 18 | Blindness unilateral |
| 19 | Chemical iritis |
| 20 | Chorioretinitis |
| 21 | Chorioretinopathy |
| 22 | Choroiditis |
| 23 | Ciliary hyperaemia |
| 24 | Cogan's syndrome |
| 25 | Cyclitic membrane |
| 26 | Cyclitis |
| 27 | Cystoid macular oedema |
| 28 | Cytomegalovirus chorioretinitis |
| 29 | Eales' disease |
| 30 | Endophthalmitis |

| | Selected Preferred Terms |
|----|--------------------------------|
| 31 | Exudative retinopathy |
| 32 | Eye inflammation |
| 33 | Fuchs' syndrome |
| 34 | Glaucomatocyclitic crises |
| 35 | Нуроруоп |
| 36 | Hypotony of eye |
| 37 | IRVAN syndrome |
| 38 | Infectious iridocyclitis |
| 39 | Iridocyclitis |
| 40 | Iritis |
| 41 | Koeppe nodules |
| 42 | Macular oedema |
| 43 | Necrotising retinitis |
| 44 | Non-infectious endophthalmitis |
| 45 | Noninfective chorioretinitis |
| 46 | Noninfective retinitis |
| 47 | Ocular lymphoma |
| 48 | Ocular sarcoidosis |
| 49 | Ocular toxicity |
| 50 | Ocular vasculitis |
| 51 | Optic discs blurred |
| 52 | Panophthalmitis |
| 53 | Photophobia |
| 54 | Photopsia |
| 55 | Retinal exudates |
| 56 | Retinal oedema |
| 57 | Retinal perivascular sheathing |
| 58 | Retinal pigment epitheliopathy |
| 59 | Retinal toxicity |
| 60 | Retinal vasculitis |
| 61 | Retinitis |
| 62 | Subretinal fluid |
| 63 | Sudden visual loss |

| | Selected Preferred Terms |
|----|---------------------------------------------------|
| 64 | Susac's syndrome |
| 65 | Sympathetic ophthalmia |
| 66 | Traumatic iritis |
| 67 | Tubulointerstitial nephritis and uveitis syndrome |
| 68 | Uveitic glaucoma |
| 69 | Uveitis |
| 70 | Uveitis-glaucoma-hyphaema syndrome |
| 71 | Vision blurred |
| 72 | Visual acuity reduced |
| 73 | Visual acuity reduced transiently |
| 74 | Visual field defect |
| 75 | Visual impairment |
| 76 | Vitreal cells |
| 77 | Vitreous fibrin |
| 78 | Vitreous floaters |
| 79 | Vitreous opacities |
| 80 | Vitritis |
| 81 | Vogt-Koyanagi-Harada syndrome |

## **Appendix 5.** Potential Cardiovascular or Cerebrovascular Events

| | Selected Preferred Terms |
|----|----------------------------------|
| 1 | Amaurosis fugax |
| 2 | Basal ganglia infarction |
| 3 | Basal ganglia stroke |
| 4 | Basilar artery occlusion |
| 5 | Basilar artery stenosis |
| 6 | Basilar artery thrombosis |
| 7 | Brachiocephalic arteriosclerosis |
| 8 | Brachiocephalic artery occlusion |
| 9 | Brachiocephalic artery stenosis |
| 10 | Brain hypoxia |
| 11 | Brain stem embolism |
| 12 | Brain stem infarction |
| 13 | Brain stem ischaemia |
| 14 | Brain stem stroke |
| 15 | Brain stem thrombosis |
| 16 | Capsular warning syndrome |
| 17 | Carotid angioplasty |
| 18 | Carotid arterial embolus |
| 19 | Carotid arteriosclerosis |
| 20 | Carotid artery bypass |
| 21 | Carotid artery calcification |
| 22 | Carotid artery disease |
| 23 | Carotid artery insufficiency |
| 24 | Carotid artery occlusion |
| 25 | Carotid artery restenosis |
| 26 | Carotid artery stenosis |
| 27 | Carotid artery stent insertion |
| 28 | Carotid artery stent removal |
| 29 | Carotid artery thrombosis |
| 30 | Carotid endarterectomy |
| 31 | Carotid revascularisation |
| 32 | Cerebellar artery occlusion |

| | Selected Preferred Terms |
|----|-----------------------------------------|
| 33 | Cerebellar artery thrombosis |
| 34 | Cerebellar embolism |
| 35 | Cerebellar infarction |
| 36 | Cerebellar ischaemia |
| 37 | Cerebral arteriosclerosis |
| 38 | Cerebral artery embolism |
| 39 | Cerebral artery occlusion |
| 40 | Cerebral artery restenosis |
| 41 | Cerebral artery stenosis |
| 42 | Cerebral artery thrombosis |
| 43 | Cerebral gas embolism |
| 44 | Cerebral infarction |
| 45 | Cerebral infarction foetal |
| 46 | Cerebral ischaemia |
| 47 | Cerebral microembolism |
| 48 | Cerebral revascularisation |
| 49 | Cerebral septic infarct |
| 50 | Cerebral small vessel ischaemic disease |
| 51 | Cerebral thrombosis |
| 52 | Cerebral vascular occlusion |
| 53 | Cerebral vasoconstriction |
| 54 | Cerebral venous thrombosis |
| 55 | Cerebrovascular accident |
| 56 | Cerebrovascular disorder |
| 57 | Cerebrovascular insufficiency |
| 58 | Cerebrovascular stenosis |
| 59 | Delayed ischaemic neurological deficit |
| 60 | Embolic cerebral infarction |
| 61 | Embolic stroke |
| 62 | Hypoxic-ischaemic encephalopathy |
| 63 | Inner ear infarction |
| 64 | Ischaemic cerebral infarction |
| 65 | Ischaemic stroke |

| 66 Lacunar infarction 67 Lacunar stroke 68 Lateral medullary syndrome 69 Migrainous infarction 70 Millard-Gubler syndrome 71 Moyamoya disease 72 Perinatal stroke 73 Post cardiac arrest syndrome 74 Post procedural stroke 75 Precerebral artery syndrome 76 Precerebral artery occlusion 77 Reversible cerebral vasoconstriction syndrome 78 Reversible ischaemic neurological deficit 79 Spinal artery thrombosis 80 Spinal artery thrombosis 81 Stroke in evolution 82 Subclavian steal syndrome 83 Thalamic infarction 84 Thrombotic stroke 85 Thrombotic cerebral infarction 84 Thrombotic stroke 86 Transient ischaemic attack 87 Vascular stent restenosis 90 Vascular stent restenosis 90 Vascular stent restenosis < | | Selected Preferred Terms |
|---|---|---|
| 68 Lateral medullary syndrome 69 Migrainous infarction 70 Millard-Gubler syndrome 71 Moyamoya disease 72 Perinatal stroke 73 Post cardiae arrest syndrome 74 Post procedural stroke 75 Precerebral arteriosclerosis 76 Precerebral artery occlusion 77 Reversible cerebral vasoconstriction syndrome 78 Reversible ischaemic neurological deficit 79 Spinal artery thrombosis 80 Spinal artery thrombosis 81 Stroke in evolution 82 Subclavian steal syndrome 83 Thalamic infarction 84 Thrombotic cerebral infarction 85 Transient ischaemic attack 86 Transient ischaemic attack 87 Vascular stent occlusion 88 Vascular stent restenosis 90 Vascular stent restenosis 91 Vertebral artery occlusion 92 Vertebral artery stenosis 93 Vertebral artery thrombosis 94 Vertebrobasilar insufficiency 95 Angina pectoris 96 Angina unstable 97 Anginal equivalent | 66 | Lacunar infarction |
| 69 Migrainous infarction 70 Millard-Gubler syndrome 71 Moyamoya disease 72 Perinatal stroke 73 Post cardiac arrest syndrome 74 Post procedural stroke 75 Precerebral artery occlusion 76 Precerebral artery occlusion 77 Reversible cerebral vasoconstriction syndrome 78 Reversible ischaemic neurological deficit 79 Spinal artery embolism 80 Spinal artery thrombosis 81 Stroke in evolution 82 Subclavian steal syndrome 83 Thalamic infarction 84 Thrombotic cerebral infarction 85 Thrombotic stroke 86 Transient ischaemic attack 87 Vascular stent occlusion 88 Vascular stent occlusion 89 Vascular stent stenosis 90 Vascular stent stenosis 91 Vertebral artery occlusion 92 Vertebral artery stenosis 93 Vertebral artery thrombosis <td>67</td> <td>Lacunar stroke</td> | 67 | Lacunar stroke |
| Millard-Gubler syndrome Moyamoya disease Perinatal stroke Perinatal stroke Post cardiac arrest syndrome Post procedural stroke Precerebral arteriosclerosis Precerebral artery occlusion Reversible cerebral vasoconstriction syndrome Reversible ischaemic neurological deficit Pspanial artery embolism Spinal artery embolism Spinal artery thrombosis Stroke in evolution Subclavian steal syndrome Subclavian steal syndrome Thalamic infarction Thrombotic cerebral infarction Thrombotic stroke Transient ischaemic attack Transient ischaemic attack Vascular encephalopathy Vascular stent occlusion Vascular stent restenosis Vertebral artery occlusion Vertebral artery stenosis Vertebral artery thrombosis Angina pectoris Angina pectoris Anginal equivalent | 68 | Lateral medullary syndrome |
| 71 Moyamoya disease 72 Perinatal stroke 73 Post cardiac arrest syndrome 74 Post procedural stroke 75 Precerebral arteriosclerosis 76 Precerebral artery occlusion 77 Reversible cerebral vasoconstriction syndrome 78 Reversible ischaemic neurological deficit 79 Spinal artery embolism 80 Spinal artery thrombosis 81 Stroke in evolution 82 Subclavian steal syndrome 83 Thalamic infarction 84 Thrombotic cerebral infarction 85 Thrombotic stroke 86 Transient ischaemic attack 87 Vascular encephalopathy 88 Vascular stent occlusion 89 Vascular stent restenosis 90 Vascular stent stenosis 91 Vertebral artery occlusion 92 Vertebral artery stenosis 93 Vertebral artery thrombosis 94 Vertebrobasilar insufficiency 95 Angina pectoris 96 Anginal equivalent | 69 | Migrainous infarction |
| Perinatal stroke Post cardiac arrest syndrome Post procedural stroke Post procedural stroke Precerebral arteriosclerosis Precerebral artery occlusion Reversible cerebral vasoconstriction syndrome Reversible ischaemic neurological deficit Psyndrome Reversible ischaemic neurological deficit Psyndrome Spinal artery embolism Spinal artery thrombosis Stroke in evolution Subclavian steal syndrome Thalamic infarction Thrombotic cerebral infarction Thrombotic cerebral infarction Thrombotic stroke Transient ischaemic attack Transient ischaemic attack Vascular encephalopathy Vascular stent occlusion Vascular stent stenosis Varcular artery occlusion Varcular artery occlusion Varcular artery stenosis Varcular artery stenosis Agina pectoris Angina pectoris Angina pectoris | 70 | Millard-Gubler syndrome |
| Post cardiac arrest syndrome Post procedural stroke Precerebral arteriosclerosis Precerebral artery occlusion Reversible cerebral vasoconstriction syndrome Reversible ischaemic neurological deficit Pspinal artery embolism Spinal artery embolism Spinal artery thrombosis Stroke in evolution Patholic cerebral infarction Thrombotic cerebral infarction Thrombotic erebral infarction Thrombotic stroke Transient ischaemic attack Vascular encephalopathy Vascular stent occlusion Vascular stent restenosis Vascular stent stenosis Vertebral artery occlusion Vertebral artery stenosis Vertebral artery thrombosis Angina pectoris Angina unstable | 71 | Moyamoya disease |
| Post procedural stroke Precerebral arteriosclerosis Precerebral artery occlusion Precerebral artery occlusion Reversible cerebral vasoconstriction syndrome Reversible ischaemic neurological deficit Pspinal artery embolism Spinal artery embolism Spinal artery thrombosis Stroke in evolution Subclavian steal syndrome Subclavian steal syndrome Thrombotic cerebral infarction Thrombotic stroke Transient ischaemic attack Vascular encephalopathy Vascular stent occlusion Vascular stent stenosis Vascular stent stenosis Vertebral artery occlusion Vertebral artery stenosis Vertebral artery thrombosis Vertebral artery thrombosis Vertebrobasilar insufficiency Anginal pectoris Anginal equivalent | 72 | Perinatal stroke |
| 75 Precerebral arteriosclerosis 76 Precerebral artery occlusion 77 Reversible cerebral vasoconstriction syndrome 78 Reversible ischaemic neurological deficit 79 Spinal artery embolism 80 Spinal artery trombosis 81 Stroke in evolution 82 Subclavian steal syndrome 83 Thalamic infarction 84 Thrombotic cerebral infarction 85 Thrombotic stroke 86 Transient ischaemic attack 87 Vascular encephalopathy 88 Vascular stent occlusion 89 Vascular stent restenosis 90 Vascular stent stenosis 91 Vertebral artery occlusion 92 Vertebral artery stenosis 93 Vertebral artery thrombosis 94 Vertebrobasilar insufficiency 95 Angina pectoris 96 Anginal equivalent | 73 | Post cardiac arrest syndrome |
| 76Precerebral artery occlusion77Reversible cerebral vasoconstriction syndrome78Reversible ischaemic neurological deficit79Spinal artery embolism80Spinal artery thrombosis81Stroke in evolution82Subclavian steal syndrome83Thalamic infarction84Thrombotic cerebral infarction85Transient ischaemic attack87Vascular encephalopathy88Vascular stent occlusion89Vascular stent restenosis90Vascular stent tersenosis91Vertebral artery occlusion92Vertebral artery thrombosis93Vertebral artery thrombosis94Vertebrobasilar insufficiency95Angina pectoris96Angina unstable97Anginal equivalent | 74 | Post procedural stroke |
| Reversible cerebral vasoconstriction syndrome Reversible ischaemic neurological deficit Reversible cerebral ischaemic Reversible ischaemic neurological deficit Reversible cerebral ischaemic Reversible ischaemic neurological deficit Reversible cerebral ischaemic Reversible ischaemic neurological deficit Reversible cerebral vasoconstriction Reversible ischaemic neurological deficit Reversible cerebral vasoconstriction Reversible ischaemic neurological deficit Reversible cerebral vasoconstriction Reversible ischaemic neurological deficit Reversible cerebral vasoconstriction Reversible schaemic neurological deficit Reversible cerebral vasoconstriction Reversible schaemic neurological deficit Reversible cerebral vasoconstriction Reversible schaemic neurological deficit Reversible cerebral vasoconstriction Reversible schaemic neurological deficit Reversible cerebral vasoconstriction Reversible cerebral artery thrombosis Parallel vasoconstriction Reversible cerebral vasoconstri | 75 | Precerebral arteriosclerosis |
| Reversible ischaemic neurological deficit Spinal artery embolism Spinal artery thrombosis Stroke in evolution Stroke in evolution Subclavian steal syndrome Thalamic infarction Thrombotic cerebral infarction Thrombotic stroke Thrombotic stroke Transient ischaemic attack Vascular encephalopathy Vascular stent occlusion Vascular stent restenosis Vascular stent restenosis Vertebral artery occlusion Vertebral artery stenosis Vertebral artery thrombosis Vertebral artery thrombosis Angina pectoris Angina lequivalent | 76 | Precerebral artery occlusion |
| Spinal artery embolism Spinal artery thrombosis Spinal artery thrombosis Stroke in evolution Stroke in evolution Subclavian steal syndrome Thalamic infarction Thrombotic cerebral infarction Thrombotic stroke Thrombotic stroke Transient ischaemic attack Vascular encephalopathy Subclavian stent occlusion Vascular stent occlusion Vascular stent restenosis Vascular stent stenosis Vertebral artery occlusion Vertebral artery stenosis Vertebral artery thrombosis Vertebral artery thrombosis Angina pectoris Angina unstable Anginal equivalent | 77 | Reversible cerebral vasoconstriction syndrome |
| Spinal artery thrombosis Stroke in evolution Stroke in evolution Subclavian steal syndrome Subclavian steat infarction Subclavian steation Subclavian | 78 | Reversible ischaemic neurological deficit |
| Stroke in evolution Subclavian steal syndrome Thalamic infarction Thrombotic cerebral infarction Thrombotic stroke Transient ischaemic attack Vascular encephalopathy Vascular stent occlusion Vascular stent restenosis Vascular stent stenosis Vertebral artery occlusion Vertebral artery stenosis Vertebral artery thrombosis Vertebral artery thrombosis Angina pectoris Angina unstable Anginal equivalent | 79 | Spinal artery embolism |
| Subclavian steal syndrome Thalamic infarction Thrombotic cerebral infarction Thrombotic stroke Thrombotic stroke Transient ischaemic attack Vascular encephalopathy Vascular stent occlusion Vascular stent restenosis Vascular stent stenosis Vertebral artery occlusion Vertebral artery stenosis Vertebral artery thrombosis Vertebral artery thrombosis Angina pectoris Angina unstable Anginal equivalent | 80 | Spinal artery thrombosis |
| Thalamic infarction Thrombotic cerebral infarction Thrombotic stroke Transient ischaemic attack Transient ischaemic attack Vascular encephalopathy Vascular stent occlusion Vascular stent restenosis Vascular stent stenosis Vertebral artery occlusion Vertebral artery stenosis Vertebral artery thrombosis Vertebral artery thrombosis Angina pectoris Angina unstable Anginal equivalent | 81 | Stroke in evolution |
| Thrombotic cerebral infarction Thrombotic stroke Transient ischaemic attack Vascular encephalopathy Vascular stent occlusion Vascular stent restenosis Vertebral artery occlusion Vertebral artery stenosis Vertebral artery thrombosis Vertebral artery thrombosis Angina pectoris Anginal equivalent | 82 | Subclavian steal syndrome |
| Thrombotic stroke Transient ischaemic attack Vascular encephalopathy Vascular stent occlusion Vascular stent restenosis Vascular stent stenosis Vascular stent stenosis Vertebral artery occlusion Vertebral artery stenosis Vertebral artery thrombosis Vertebral artery thrombosis Angina pectoris Angina unstable Anginal equivalent | 83 | Thalamic infarction |
| Transient ischaemic attack Vascular encephalopathy Vascular stent occlusion Vascular stent restenosis Vascular stent stenosis Vascular stent stenosis Vertebral artery occlusion Vertebral artery stenosis Vertebral artery thrombosis Vertebral artery thrombosis Angina pectoris Anginal equivalent | 84 | Thrombotic cerebral infarction |
| Vascular encephalopathy Vascular stent occlusion Vascular stent restenosis Vascular stent stenosis Vertebral artery occlusion Vertebral artery stenosis Vertebral artery thrombosis Vertebral artery thrombosis Angina pectoris Angina unstable Anginal equivalent | 85 | Thrombotic stroke |
| Vascular stent occlusion Vascular stent restenosis Vascular stent stenosis Vertebral artery occlusion Vertebral artery stenosis Vertebral artery thrombosis Vertebral artery thrombosis Angina pectoris Angina unstable Anginal equivalent | 86 | Transient ischaemic attack |
| Vascular stent restenosis Vascular stent stenosis Vertebral artery occlusion Vertebral artery stenosis Vertebral artery thrombosis Vertebrobasilar insufficiency Angina pectoris Angina unstable Anginal equivalent | 87 | Vascular encephalopathy |
| 90Vascular stent stenosis91Vertebral artery occlusion92Vertebral artery stenosis93Vertebral artery thrombosis94Vertebrobasilar insufficiency95Angina pectoris96Angina unstable97Anginal equivalent | 88 | Vascular stent occlusion |
| 91Vertebral artery occlusion92Vertebral artery stenosis93Vertebral artery thrombosis94Vertebrobasilar insufficiency95Angina pectoris96Angina unstable97Anginal equivalent | 89 | Vascular stent restenosis |
| 92 Vertebral artery stenosis 93 Vertebral artery thrombosis 94 Vertebrobasilar insufficiency 95 Angina pectoris 96 Angina unstable 97 Anginal equivalent | 90 | Vascular stent stenosis |
| 93 Vertebral artery thrombosis 94 Vertebrobasilar insufficiency 95 Angina pectoris 96 Angina unstable 97 Anginal equivalent | 91 | Vertebral artery occlusion |
| 94 Vertebrobasilar insufficiency 95 Angina pectoris 96 Angina unstable 97 Anginal equivalent | 92 | Vertebral artery stenosis |
| 95 Angina pectoris 96 Angina unstable 97 Anginal equivalent | 93 | Vertebral artery thrombosis |
| 96 Angina unstable 97 Anginal equivalent | 94 | Vertebrobasilar insufficiency |
| 97 Anginal equivalent | 95 | Angina pectoris |
| | 96 | Angina unstable |
| 98 Arteriosclerosis coronary artery | 97 | Anginal equivalent |
| | 98 | Arteriosclerosis coronary artery |

| | Selected Preferred Terms |
|-----|------------------------------------------------|
| 99 | Arteriospasm coronary |
| 100 | Coronary angioplasty |
| 101 | Coronary arterial stent insertion |
| 102 | Coronary artery bypass |
| 103 | Coronary artery disease |
| 104 | Coronary artery dissection |
| 105 | Coronary artery insufficiency |
| 106 | Coronary artery restenosis |
| 107 | Coronary artery stenosis |
| 108 | Coronary brachytherapy |
| 109 | Coronary bypass stenosis |
| 110 | Coronary endarterectomy |
| 111 | Coronary no-reflow phenomenon |
| 112 | Coronary ostial stenosis |
| 113 | Coronary revascularisation |
| 114 | Coronary vascular graft stenosis |
| 115 | Dissecting coronary artery aneurysm |
| 116 | ECG signs of myocardial ischaemia |
| 117 | External counterpulsation |
| 118 | Haemorrhage coronary artery |
| 119 | Ischaemic cardiomyopathy |
| 120 | Ischaemic mitral regurgitation |
| 121 | Microvascular coronary artery disease |
| 122 | Myocardial ischaemia |
| 123 | Percutaneous coronary intervention |
| 124 | Prinzmetal angina |
| 125 | Stress cardiomyopathy |
| 126 | Subclavian coronary steal syndrome |
| 127 | Subendocardial ischaemia |
| 128 | Arteriogram coronary abnormal |
| 129 | Cardiac stress test abnormal |
| 130 | Cardiopulmonary exercise test abnormal |
| 131 | Computerised tomogram coronary artery abnormal |

| | Selected Preferred Terms |
|-----|-------------------------------------------|
| 132 | Electrocardiogram ST segment depression |
| 133 | Electrocardiogram ST-T segment abnormal |
| 134 | Electrocardiogram ST-T segment depression |
| 135 | Electrocardiogram T wave abnormal |
| 136 | Electrocardiogram T wave inversion |
| 137 | Exercise electrocardiogram abnormal |
| 138 | Exercise test abnormal |
| 139 | Post angioplasty restenosis |
| 140 | Stress echocardiogram abnormal |
| 141 | Vascular stent restenosis |
| 142 | Vascular stent stenosis |
| 143 | Acute coronary syndrome |
| 144 | Acute myocardial infarction |
| 145 | Angina unstable |
| 146 | Blood creatine phosphokinase MB abnormal |
| 147 | Blood creatine phosphokinase MB increased |
| 148 | Coronary artery embolism |
| 149 | Coronary artery occlusion |
| 150 | Coronary artery reocclusion |
| 151 | Coronary artery thrombosis |
| 152 | Coronary bypass thrombosis |
| 153 | Coronary vascular graft occlusion |
| 154 | Kounis syndrome |
| 155 | Myocardial infarction |
| 156 | Myocardial necrosis |
| 157 | Myocardial reperfusion injury |
| 158 | Myocardial stunning |
| 159 | Papillary muscle infarction |
| 160 | Post procedural myocardial infarction |
| 161 | Postinfarction angina |
| 162 | Silent myocardial infarction |
| 163 | Troponin I increased |
| 164 | Troponin increased |

| | Selected Preferred Terms |
|-----|------------------------------------------|
| 165 | Troponin T increased |
| 166 | Blood creatine phosphokinase abnormal |
| 167 | Blood creatine phosphokinase increased |
| 168 | Cardiac ventricular scarring |
| 169 | ECG electrically inactive area |
| 170 | ECG signs of myocardial infarction |
| 171 | Electrocardiogram Q wave abnormal |
| 172 | Electrocardiogram ST segment abnormal |
| 173 | Electrocardiogram ST segment elevation |
| 174 | Electrocardiogram ST-T segment elevation |
| 175 | Infarction |
| 176 | Myocardial necrosis marker increased |
| 177 | Scan myocardial perfusion abnormal |
| 178 | Vascular graft occlusion |
| 179 | Vascular stent occlusion |
| 180 | Vascular stent thrombosis |